

Study Code D6930C00001(PT007001)

NCT # NCT03364608 Date 13 MARCH 2018

A Randomized, Double-blind, Single dose, Placebo-controlled, 5-Period, 5-Treatment, Crossover, Multi-center, Dose-ranging Study to Compare PT007 to Placebo MDI and Open-Label Proventil® HFA in Adult and Adolescent Subjects With Mild to Moderate Asthma

Protocol No. D6930C00001 (PT007001) Last Revision Date: 13 Mar 2018


### STATISTICAL ANALYSIS PLAN

| Trial Sponsor: | AstraZeneca |
|---|---|
| Study Number: | D6930C00001 (PT007001) |
| Study Phase: | II |
| Product Name: | Albuterol Sulfate Pressurized Inhalation Suspension (AS MDI); PT007 |
| PIND Number: | 136213 |
| Indication: | Asthma |
| Dosage Form/Strength | <ul> <li>AS MDI as</li> <li>2 actuations of 45 μg per actuation (90 μg)</li> <li>2 actuations of 90 μg per actuation (180 μg)</li> </ul> |

**Protocol Title:** A Randomized, Double-blind, Single dose, Placebo-controlled, 5-Period, 5-Treatment, Crossover, Multi-center, Dose-ranging Study to Compare PT007 to Placebo MDI and Open-Label Proventil<sup>®</sup> HFA in Adult and Adolescent Subjects With Mild to Moderate Asthma

**Date of Issue:** 13 Mar 2018

Version 1.0



Statistical Analysis Plan Protocol No. D6930C00001 (PT007001) Last Revision Date: 13 Mar 2018


### Signed Agreement on Statistical Analysis Plan

### **FINAL SIGN-OFF SIGNATURES**

| Study<br>Biostatistician: |
|---------------------------------|
| Peer Review<br>Biostatistician: |
| Approved by: |
| Approved by: |
| Approved by: |



Statistical Analysis Plan Protocol No. D6930C00001 (PT007001) Last Revision Date: 13 Mar 2018


### Signed Agreement on Statistical Analysis Plan

### FINAL SIGN-OFF SIGNATURES

| Study<br>Biostatistician: |
|---------------------------------|
| Peer Review<br>Biostatistician: |
| Approved by: |
| Approved by: |
| Approved by: |

Protocol No. D6930C00001 (PT007001) Last Revision Date: 13 Mar 2018


### **TABLE OF CONTENTS**

| LIST | OF | TABLES | 5 |
|---|---|---|---|
| LIST | OF | FIGURES | 5 |
| LIST | OF | ABBREVIATIONS AND DEFINITIONS OF TERMS | 6 |
| 1. | | RODUCTION | |
| 2. | | DY OBJECTIVES | |
| ۷. | | | |
| | 2.1 | PRIMARY OBJECTIVE | |
| | 2.2 | SECONDARY OBJECTIVE | |
| | 2.3 | SAFETY OBJECTIVE | |
| 3. | STU | DY ENDPOINTS | 8 |
| | 3.1 | EFFICACY ASSESSMENTS | |
| | 3.2 | PRIMARY EFFICACY ENDPOINT | |
| | 3.3 | SECONDARY EFFICACY ENDPOINTS | |
| | 3.4 | OTHER EFFICACY ENDPOINTS | |
| | 3.5 | SAFETY ENDPOINTS | 9 |
| 4. | STU | DY DESIGN | 9 |
| | 4.1 | STUDY DESIGN AND PLAN | 9 |
| | 4.2 | RANDOMIZATION | |
| | 4.3 | HYPOTHESIS TESTING | |
| | 4.4 | INTERIM ANALYSIS | 17 |
| | 4.5 | SAMPLE SIZE | 17 |
| 5. | DAT | A AND ANALYTICAL QUALITY ASSURANCE | 18 |
| 6. | | LYSIS SETS | |
| | 6.1 | Intent-to-Treat (ITT) Analysis Set | |
| | 6.2 | MODIFIED ITT (MITT) ANALYSIS SET | |
| | 6.3 | SAFETY ANALYSIS SET | |
| | 6.4 | Not-randomized Analysis Set | |
| | 6.5 | ANALYSIS SETS FOR ANALYSES | |
| 7. | | TISTICAL ANALYSIS | |
| 7. | SIA | | |
| | | 7.1.1 General Data Handling Rules and Definitions | |
| | | 7.1.2 Data Exclusion and Missing Data Imputation | |
| | 7.2 | SUBJECT DISPOSITION | |
| | 7.3 | DEMOGRAPHY | |
| | | <ul> <li>7.3.1 Asthma History, Screening/Baseline Spirometry, and Reversibility</li> <li>7.3.2 Medical and Surgical History at Screening, Pregnancy Testing at Screening and</li> </ul> | 21 |
| | | 7.3.2 Medical and Surgical History at Screening, Pregnancy Testing at Screening and Baseline | |
| | | 7.3.3 Prior, Concomitant, and Post-Treatment Medications/Treatments | 22 |
| | | 1.5.5 1 1101, Concommuni, and 1 051-110auntent Medications/110auntents | |
| | | 7.3.4 Extent of Exposure to Study Drug | 22 |
| | 74 | 7.3.4 Extent of Exposure to Study Drug | 22 |
| | 7.4 | EFFICACY ANALYSES | 22<br>22<br>23 |
| | 7.4 | EFFICACY ANALYSES | 22<br>22<br>23 |
| | 7.4 | EFFICACY ANALYSES | 22<br>23<br>23 |



**Statistical Analysis Plan** Protocol No. D6930C00001 (PT007001)

Last Revision Date: 13 Mar 2018

| Page | 4 | of | 48) | ١ |
|------|---|----|-----|---|

| | 7 | .4.5 | Secondary Efficacy | 26 |
|-----|--------|---------|-----------------------------------------|----|
| | 7 | .4.6 | Other Efficacy | 26 |
| | 7 | .4.7 | Data Validation and Transformation | 27 |
| | 7.5 S. | | NALYSES | |
| | 7 | .5.1 | Adverse Events | 28 |
| | 7 | .5.2 | Clinical Laboratory Data | 30 |
| | 7 | .5.3 | Vital Signs | 32 |
| | 7 | .5.4 | Electrocardiogram (ECG) | 33 |
| | 7 | .5.5 | Physical Examination | 33 |
| 8. | CHANG | GES FR | OM METHODS PLANNED IN THE PROTOCOL | 33 |
| 9. | STATIS | STICAL | SOFTWARE | 33 |
| 10. | REFER | RENCES | S | 34 |
| API | PENDIX | 1 DATA | HANDLING RULES | 35 |
| API | PENDIX | 2 ANAI | YSIS DATASET SPECIFICATIONS | 42 |
| API | PENDIX | 3 SAS C | CODE FOR STATISTICAL ANALYSES | 43 |
| API | PENDIX | 4 MOC | KUP TABLES, LISTINGS, AND GRAPHS (TLGS) | 48 |



**Statistical Analysis Plan** Protocol No. D6930C00001 (PT007001)

Last Revision Date: 13 Mar 2018

### 

### List of Tables

| | 2100 01 1 100200 | |
|---|---|---|
| Table 1 | Schedule of Events | 12 |
| Table 2 | Timed Assessments at Visits 2, 3, 4, and 5 | 14 |
| | Timed Assessments at Visit 6 | |
| Table 4 | Analysis Study Time Windows for Spirometry Assessments | 24 |
| | Lab Parameters | |
| Table 6 | Potentially Clinically Significant Criteria for Systolic and Diastolic Blood Pressure Parameters and Heart Rate | 32 |
| | List of Figures | |
| Figure 1 | Study Flow Diagram: | 11 |





Protocol No. D6930C00001 (PT007001)

Last Revision Date: 13 Mar 2018


### LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE Adverse event

ALT Alanine aminotransferase

AS Albuterol Sulfate

AST Aspartate aminotransferase

ATC Anatomical Therapeutic Chemical

ATS American Thoracic Society

AUC $_{0-6}$  Area under the curve from time 0 to 6 hours AUC $_{0-4}$  Area under the curve from time 0 to 4 hours

β-hCG β-human chorionic gonadotropin

BID Bis in die, twice daily
BMI Body mass index

BMP Basic metabolic panel
BPM Beats per minute
BUN Blood urea nitrogen

CKD-EPI Chronic Kidney Disease Epidemiology Collaboration

CI Confidence interval

CTCAE Common Terminology Criteria for Adverse Events

DBP Diastolic blood pressure
DMP Data Management Plan

CRF Case report form

DMP Data management plan ECG Electrocardiogram

eCRF Electronic case report form

eDiary Electronic diary

eGFR Estimated glomerular filtration rate ERS European Respiratory Society

FEF<sub>25-75</sub> Forced expiratory flow from 25% to 75% of FVC

FEV<sub>1</sub> Forced expiratory volume in 1 second

FVC Forced vital capacity

GGT Gamma-glutamyl transpeptidase

H<sub>0</sub> Null hypothesis

H<sub>1</sub> Alternative hypothesis HFA Hydrofluoroalkane

HR Heart rate

ICS Inhaled corticosteroid ITT Intention-to-treat

IWRS Interactive web response system



Protocol No. D6930C00001 (PT007001)

Last Revision Date: 13 Mar 2018


LABA Long-acting β2-agonist

Mean corpuscular hemoglobin **MCH** 

Mean corpuscular hemoglobin concentration MCHC

MCV Mean corpuscular volume MDI Metered dose inhaler

Medical Dictionary for Regulatory Activities MedDRA

Modified intent-to-treat mITT

OTC Over-the-counter

**PDV** Premature discontinuation visit PCS Potentially clinically significant

PEFR Peak expiratory flow rate PFT Pulmonary function test

PR Time from electrocardiogram P wave to the end of the R wave

corresponding to electrical systole

QA Quality assurance QC Quality control

Time from electrocardiogram Q wave to the end of the T wave QΤ

corresponding to electrical systole

QTcF QT corrected using Fridericia's formula [QT/(RR1/3)]

Time from electrocardiogram R wave to the next R wave corresponding to RR

electrical systole

SAE Serious adverse event Short-acting β-agonist SABA

SAL Salmeterol

SAP Statistical analysis plan

sPDP Statistical protocol deviation plan SAS Statistical Analysis System SBP Systolic blood pressure SD Standard deviation

SI International System of Units (Système International d'Unités)

SOC System organ class TC Telephone call

TEAE Treatment emergent adverse event

TP Treatment period ULN Upper limit of normal

**United States** US/USA

World Health Organization Drug Dictionary Enhanced WHO DDE

WHO HD World Health Organization Herbal Dictionary



Protocol No. D6930C00001 (PT007001)

Last Revision Date: 13 Mar 2018 

### 1. INTRODUCTION

AstraZeneca is developing a broad range of metered dose inhaler (MDI)-based inhalation aerosols using its porous particle technology platform, including Albuterol Sulfate Pressurized Inhalation Suspension (AS) MDI.

This Statistical Analysis Plan (SAP) outlines the statistical methods for the display, summary, and analysis of data collected within the scope of Clinical Trial Protocol D6930C00001 (PT007001), Version 2.0 (Amendment 1), dated January 12, 2018.

All references to doses of AS MDI and Proventil<sup>®</sup> HFA (hereafter referred to as Proventil) refer to the albuterol base (i.e., 90 µg albuterol base, which equals 108 µg albuterol sulfate).

### 2. STUDY OBJECTIVES

### 2.1 Primary Objective

• To confirm the dose of albuterol delivered from AS MDI that is comparable to Proventil

### 2.2 Secondary Objective

• To assess the dose response of AS MDI versus Placebo for AS MDI (hereafter referred to as Placebo MDI)

### 2.3 Safety Objective

• To evaluate the safety and tolerability of AS MDI relative to Placebo MDI and Proventil

### 3. STUDY ENDPOINTS

### 3.1 Efficacy Assessments

This is a 5-period, 5-treatment Williams design (Williams 1949). Each Treatment Period will be 1 day, with a Washout Period of 3 to 7 days between Treatment Periods. The day of treatment in each Treatment Period is Day 1. Baseline forced expiratory volume in 1 second (FEV<sub>1</sub>) will be calculated using the mean of available pre-dose values on the first day of each Treatment Period (as defined in Section 7.4.3.1).

### 3.2 Primary Efficacy Endpoint

• Change from baseline in  $FEV_1$  area under the curve from 0 to 6 hours (AUC<sub>0-6</sub>)



Protocol No. D6930C00001 (PT007001)

Last Revision Date: 13 Mar 2018 

### 3.3 Secondary Efficacy Endpoints

- Change from baseline in FEV<sub>1</sub> AUC from 0 to 4 hours (AUC<sub>0-4</sub>)
- Peak change from baseline in FEV<sub>1</sub>

### 3.4 Other Efficacy Endpoints

- Change from baseline in FEV<sub>1</sub> at each post-dose timepoint
- Time to peak FEV<sub>1</sub>
- Percentage of subjects achieving 12% improvement in FEV<sub>1</sub> from baseline within 30 minutes of dose
- Percentage of subjects achieving 15% improvement in FEV<sub>1</sub> from baseline within 30 minutes of dose
- Time to onset of response
- Duration of response

### 3.5 Safety Endpoints

The safety endpoints include:

- Adverse Events (AEs)/serious adverse events (SAEs)
- Vital signs
- Clinical laboratory parameters
- Electrocardiograms (ECGs)

### 4. STUDY DESIGN

### 4.1 Study Design and Plan

This is a randomized, double-blind, single-dose, placebo-controlled, 5-period, 5-treatment, crossover, multi-center study to assess the bronchodilatory effect and safety of 2 dose levels of AS MDI (90  $\mu$ g and 180  $\mu$ g) compared with Placebo MDI and open-label Proventil (90  $\mu$ g and 180  $\mu$ g) in adult and adolescent subjects with mild to moderate asthma.

This study will be conducted at 10 sites in the US, contributing approximately 7 subjects per site. Across these sites, it is planned that approximately 70 subjects with mild to moderate asthma will be randomized to provide approximately 64 subjects to complete the study.

The sequence of visits is displayed in the Study Flow Diagram (Figure 1).

For more details on the study plan please refer to Protocol Section 4.



Protocol No. D6930C00001 (PT007001)

Last Revision Date: 13 Mar 2018 

Randomization criteria for the study are listed in Section 3.3.1 of Protocol D6930C0001.

Inclusion criteria for the study are listed in Section 3.1 of Protocol D6930C00001. Subjects eligible for enrollment in the study must meet all of the inclusion criteria. To be eligible, must be at least 12 years of age and no older than 65 years with stable physician-diagnosed asthma for 6 months. Subjects must be on either a SABA as needed as their only asthma therapy or a low to medium ICS dose (either alone or in combination with a LABA) for at least 30 days, as a consistent regimen before screening. Also, subjects must have a prebronchodilator FEV<sub>1</sub> between  $\geq$ 40 and <90% of predicted normal value after withholding SABA for  $\geq$ 6 hours (and/or Visit 1a and/or Visit 1b, as applicable). Additionally, confirmed FEV<sub>1</sub> reversibility to Ventolin, defined as Post-Ventolin increase in FEV<sub>1</sub> of  $\geq$ 15% at either Visit 1, Visit 1a, or Visit 1b. Exclusion criteria for the study are listed in Section 3.2 of Protocol D6930C00001. Subjects meeting any of the exclusion criteria are to be excluded from the study. Reasons for exclusion from the study include: chronic obstructive pulmonary disease or other significant lung disease, receipt of oral corticosteroid use (any dose) within 6 weeks of their Visit 1 of the study, and hospitalization for asthma within 6 months of Visit 1.

Detailed schedules for pre- and post-dose procedures to be performed at each study visit are provided in Section 4 of the protocol. A time—and-events schedule is provided below in Table 1.

Visit procedures at each treatment visit (Visits 2, 3, 4, and 5) are provided in Table 2 and at Visit 6 in Table 3.

Protocol No. PT007001 Last Revision Date: 13 Mar 2018 

Figure 1 Study Flow Diagram:



\*Subjects on ICS or ICS/LABA prior to Visit 1 will be run-in on Pulmicort Flexhaler 180 or 360 µg BID for a minimum of 14 days.

Abbreviations: BID = twice a day, V=visit, R=randomization, Rx=treatment.



Last Revision Date: 13 Mar 2018 Protocol No. PT007001


# Schedule of Events Table 1

| | Screenin | Screening Period <sup>a</sup> | | | Treatme | Treatment Phase <sup>b</sup> | | | Follow-up |
|---|---|---|---|---|---|---|---|---|---|
| | Visit 1 | Visit 1a/b | Visit 2 | | | | | | TC |
| Treatment Day <sup>a</sup> | Dav -28 to Dav -1 | to Dav -1 | Rand.<br>(TP 1)<br>Dav 1 | Visit 3<br>(TP 2) | Visit 4 (TP 3) | Visit 5<br>(TP 4) | Visit 6<br>(TP 5) | PDV (if<br>Applicable) <sup>c</sup> | 3 to / days<br>after final<br>dose |
| Procedures | • | • | • | | | | | | |
| Informed consent (and assent, as appropriate) | × | | | | | | | | |
| Eligibility Criteria | × | | | | | | | | |
| Verify randomization criteria | | | X | | | | | | |
| Verify continued eligibility | | × | | × | × | × | × | | |
| MDI demonstration/training | X | | X | X | X | X | X | | |
| Ventolin reversibility test | X | X | | | | | | | |
| Medical/surgical history | × | | | | | | | | |
| Demographics | X | | | | | | | | |
| Concomitant medications <sup>e</sup> | X | X | X | X | X | X | X | $_{ m q}{ m X}$ | |
| Spirometry | × | × | X | × | X | X | × | | |
| | | | | X | X | X | X | | |
| Physical Examination | X | | | | | | X | X | |
| Vital Signs | × | | X | X | X | X | X | X | |
| 12-lead ECG | X | | | | | | X | X | |
| Pregnancy test <sup>g</sup> | X | | X | | | | | | |
| Clinical laboratory testing | X | | | | | | X | X | |
| Adjust asthma medications per protocol <sup>h</sup> | X | X | | | | | X | X | |
| Randomization | | | X | | | | | | |
| Randomized study drug administered | | | X | X | X | X | X | | |
| AEs | X | X | X | X | X | X | X | X | X |
| Telenhone contact | | | | | | | | | × |

Abbreviations: AE=adverse event; β-hCG= β-human chorionic gonadotropin; ECG=electrocardiogram; FEV<sub>1</sub>=forced expiratory volume in 1 second; ICS=inhaled corticosteroid; LABA= long-acting β2-agonist; MDI=metered dose inhaler; PDV=Premature Discontinuation Visit; Rand.=randomization; SABA= short-acting β-agonist; TC=telephone call; TP=Treatment Period.

Note: When data collection timepoints are concurrent, variables will be collected in the following order: vital signs, ECG, clinical laboratory assessments, and spirometry.

Screening Period will be 3 to 28 days for subjects on SABA only before study entry, and 14 to 28 days for subjects on ICS or ICS/LABA before study entry.




- Subjects to return to clinic within 3 to 7 days following Visits 2, 3, 4, and 5.
- Subjects who prematurely withdraw from the study will undergo a Premature Discontinuation Visit (see Protocol Section 4.2.5).
- For subjects who received their regularly inhaled asthma medications and/or SABA on the morning of the visit, spirometry and reversibility will be measured at Visit 1a, which will occur within 10 days of Visit 1. For subjects who do not meet reversibility criteria at Visit 1a, Visit 1b will be scheduled for a second reversibility test, to occur within 7 days. Subjects who do not meet reversibility criteria after the second attempt will be screen failed.
- At all visits beyond Visit 1, note time of the last dose of asthma medications. The visit must be rescheduled if the last dose of Ventolin was <6 hours before the visit.
- <sup>1</sup> Includes evaluation of heig and weight at Visit 1.
- A serum pregnancy test (\(\beta\)-hCG) will be performed at Visit 1; urine \(\beta\)-hCG test will be performed before randomization at Visit 2 (for women of child-bearing potential only).
- At Visit 1, prohibited asthma medications are to be stopped and asthma medications changed as specified in Section Protocol 7.2.2. At the end of Visit 6 (or upon premature discontinuation or screen failure, if applicable), subjects will return to pre-study or other appropriate maintenance asthma medications.

Statistical Analysis Plan Protocol No. PT007001 Last Revision Date: 13 Mar 2018 

Timed Assessments at Visits 2, 3, 4, and 5 Table 2

| | Pre-Dose (minutes) | Jose<br>ites) | | | | | Post-Dose (minutes) | (minutes | <b>~</b> | | | | Before<br>leaving<br>clinic |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 09- | -30 | 2 | 15 | 30 | 45 | 09 | 120 | 180 | 240 | 300 | 360 | |
| Vital signs | X | | | | | | | | | | | | X |
| Spirometry | X | X | X | X | X | X | X | X | X | X | X | X | |
| AEs | X | X | X | X | X | X | X | X | X | X | X | X | X |

Abbreviations: AE=adverse event.

Statistical Analysis Plan Protocol No. PT007001 Last Revision Date: 13 Mar 2018 

# Timed Assessments at Visit 6 Table 3

| | Pre-Dose<br>(minutes) | Pre-Dose (minutes) | | | | <u> </u> | Post-Dose (minutes) | (minutes | <u> </u> | | | | Before<br>leaving<br>clinic |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 09- | -30 | w | 15 | 30 | 45 | 09 | 120 | 180 | 240 | 300 | 360 | |
| Vital signs | × | | | | | | | | | | | | × |
| 12-lead ECG <sup>b</sup> | | | | | | | | | | | | | × |
| Spirometry | × | × | × | × | × | × | × | × | × | × | × | X | |
| Physical examination | | | | | | | | | | | | | X |
| Clinical laboratory testing | | | | | | | | | | | | | X |
| AEs | X | X | X | X | X | X | X | X | X | X | X | X | X |

Abbreviations: AE=adverse event; ECG=electrocardiogram.



Last Revision Date: 13 Mar 2018 

### 4.2 Randomization

Subjects will be randomly assigned to 1 of 10 treatment sequences based on a Williams design (Williams 1949) using an interactive web response system (IWRS). Each sequence will comprise all 5 of the treatments included in this study in a randomized order.

| Sequence | Period 1 | Period 2 | Period 3 | Period 4 | Period 5 |
|----------|----------|----------|----------|----------|----------|
| 1 | A | В | Е | С | D |
| 2 | В | С | A | D | Е |
| 3 | С | D | В | Е | A |
| 4 | D | Е | С | A | В |
| 5 | Е | A | D | В | С |
| 6 | D | С | Е | В | A |
| 7 | Е | D | A | С | В |
| 8 | A | Е | В | D | С |
| 9 | В | A | С | E | D |
| 10 | С | В | D | A | Е |

Note: A=Placebo; B=AS MDI 90 μg; C=AS MDI 180 μg; D= Proventil 90 μg; E= Proventil 180 μg.

Randomization will be centralized and stratified by pre-study background therapy consisting of either inhaled corticosteroid (ICS) or non-ICS (subjects not previously treated with ICS).

### 4.3 Hypothesis Testing

Hypothesis testing will be performed within the context of a linear mixed model analysis, including all treatments. For the primary efficacy comparisons for change from baseline in  $FEV_1$   $AUC_{0-6}$  for the overall population, the primary endpoint, the null hypothesis for each pairwise comparison is that the mean test treatment effect is equal to that of Placebo MDI; the alternative hypothesis is then that the test treatment effect and that of Placebo MDI are not equal. However, while the hypotheses are written for inequality testing, demonstration of superiority relative to placebo is the objective. P-values will be reported as two-sided.

The primary null  $(H_0)$  and alternative  $(H_1)$  hypotheses with  $\mu$  representing the mean are:

- $H_0$ :  $\mu_{Proventil\ 180\ \mu g} = \mu_{placebo}$ 
  - $H_1$ :  $\mu_{Proventil\ 180\ \mu g} \neq \mu_{placebo}$
- $H_0$ :  $\mu_{AS\ MDI\ 180\ \mu g} = \mu_{placebo}$ 
  - $H_1$ :  $\mu_{AS\ MDI\ 180\ \mu g} \neq \mu_{placebo}$



Protocol No. PT007001

Last Revision Date: 13 Mar 2018 

•  $H_0$ :  $\mu_{Proventil 90 \mu g} = \mu_{placebo}$  $H_1$ :  $\mu_{Proventil 90 \mu g} \neq \mu_{placebo}$ 

•  $H_0$ :  $\mu_{AS\ MDI\ 90\ \mu g} = \mu_{placebo}$  $H_1$ :  $\mu_{AS\ MDI\ 90\ \mu g} \neq \mu_{placebo}$ 

The Type I error rate will be controlled at the 5% level (two-sided) across the superiority comparisons of the primary endpoint,  $FEV_1$  AUC<sub>0-6</sub>. In general, the superiority of Proventil relative to Placebo MDI will be tested first using a dose-ordered approach. If Proventil 180  $\mu g$  is superior to Placebo MDI, AS MDI 180  $\mu g$  will be compared to Placebo MDI. If AS MDI 180  $\mu g$  is superior to Placebo MDI, the superiority of Proventil 90- $\mu g$  relative to Placebo MDI will be tested. If Proventil 90  $\mu g$  is superior to placebo, then AS MDI 90  $\mu g$  will be compared to Placebo MDI.



Comparisons among the dose levels within a product will also be conducted for exploratory purposes. Estimated treatment differences and 95% CIs will be provided.

### 4.4 Interim Analysis

No interim analyses are planned for this trial.

### 4.5 Sample Size

Power calculations were based on the properties of the primary endpoint, the change from baseline in FEV<sub>1</sub> AUC<sub>0-6</sub>. Randomization of 70 subjects in order to achieve at least 64 subjects completing the study will provide >95% overall probability to demonstrate superiority of each treatment relative to Placebo MDI assuming a minimum detectable difference (active–Placebo MDI) of 100 mL, within-subject standard deviation of 115 mL, and two-sided 5% level test. The estimate of the within-subject standard deviation was obtained from a 5-treatment, 5-period doseranging study to evaluate albuterol dry powder inhaler and HFA in subjects ages 12 and older with persistent asthma (NCT01058863).






### 5. DATA AND ANALYTICAL QUALITY ASSURANCE

| The overall quality assurance procedures for the study data, statistical programming and analyses |
|---|
| are described in Standard Operating Procedures (SOPs) |
| ). Detailed data management procedures are documented in the study Data |
| Management Plan, Data Validation Check Specifications, and Integrated Safety Data Review Plan. |
| Detailed statistical and programming quality control and quality assurance procedures are |
| documented in the Statistical Analysis and Programming QC/QA Plan. |
| Transfer of PFT data from the central PFT laboratory to Everest will |
| be defined in the DMP (Data Management Plan), and data handling rules |
| related to this data are included in Appendix 1 of this SAP. The quality of all PFTs obtained at |
| each timepoint will be graded independently at iCardiac Technologies by qualified personnel. |
| Quality grading assessments will be based on ATS/ERS criteria and will be included in data |
| transfers. |

### 6. ANALYSIS SETS

The following analysis sets are defined in this study.

### 6.1 Intent-to-Treat (ITT) Analysis Set

The Intent-To-Treat (ITT) analysis set is defined as all subjects who are randomized to treatment and receive at least 1 dose of the study drug. Subjects will be analyzed in each period according to the treatment they were assigned to per the randomization scheme (Note that a subject who used study drug but took less than 1 full dose will qualify for this analysis set).

### 6.2 Modified ITT (mITT) Analysis Set

A Modified ITT (mITT) analysis set is a subset of the ITT analysis set including subjects who received treatment and have post-treatment efficacy data from at least 2 Treatment Periods. Data judged to be impacted by major protocol deviations will be determined prior to unblinding and excluded per the statistical protocol deviation plan (sPDP). Statistical tabulations and analyses will be by randomized treatment, but data obtained after subjects receive an incorrect treatment will be excluded from the affected periods.

Any evaluability criteria with a potential impact on efficacy results will be defined in an sPDP. The evaluability criteria will be programmatically identified in a blinded fashion aided by a review of data listings prior to database lock. Major protocol deviations (protocol violations), therefore, can result in exclusion of all data from a particular subject from the analysis population or require exclusion of data from a specific timepoint or treatment period and/or subsequent timepoints or subsequent treatment periods for an endpoint(s). Protocol deviations for exclusion of data from the mITT Analysis Set will be agreed by the study team and documented in the blinded data review meeting minutes prior to database lock.




### 6.3 Safety Analysis Set

The Safety analysis set is defined as all subjects who are randomized to treatment and receive at least 1 dose of the study drug. Subjects will be analyzed according to treatment received rather than per the randomization scheme.

### 6.4 Not-randomized Analysis Set

The Not Randomized analysis set is defined as subjects who did not receive a randomization number and therefore did not receive a dose of study drug (eg, subjects who were screen failures or stopped participation before being randomized).

### 6.5 Analysis Sets for Analyses

Analyses will be performed as follows:

Demographics and baseline characteristics will be summarized for the ITT, mITT, Safety, and Not-randomized analysis sets. Extent of exposure will be listed for the Safety analysis set. The Safety analysis set will be used to summarize safety.

Efficacy analyses will be performed for the mITT analysis set. As a sensitivity analysis, the primary endpoint, change from baseline in FEV<sub>1</sub> AUC<sub>0-6</sub>, will also be analyzed using the ITT analysis set.

### 7. STATISTICAL ANALYSIS

### 7.1.1 General Data Handling Rules and Definitions

All data collected on case report forms will be provided in listings, except data collected only for confirmation of study entry criteria and for study administrative purposes. If any randomized subject is found to not have valid documented informed consent, that subject's data will be excluded from the report, except as necessary to document the error.

Except where specified all continuous variables will be summarized with descriptive statistics (the number of non-missing values, mean, standard deviation, median, minimum and maximum) and all categorical variables will be summarized with frequency counts and percentages, by treatment.

Missing data will be maintained as missing in the analysis datasets, unless specified otherwise. For variables where missing data are imputed, another analysis dataset will contain a variable with the imputed value. Thus, the original variable value will be maintained as missing in 1 of the analysis datasets.

All efficacy and safety parameters will be summarized by treatment (unless specified otherwise). Summary statistics for safety will be provided for the Safety Analysis Set, unless otherwise specified.





Last Revision Date: 13 Mar 2018


### 7.1.2 Data Exclusion and Missing Data Imputation

Pre-dose spirometry values will use the average of the non-missing -60 minute and -30 minute values. A detailed description of the baseline value calculation is in Section 7.4.3.1.

For the mITT analyses, FEV<sub>1</sub> AUC<sub>0-6</sub>, FEV<sub>1</sub> AUC<sub>0-4</sub>, and peak FEV<sub>1</sub> will be calculated if there is at least 1 non-missing data point during the first 2 hours post-dose.

Unless otherwise specified, all lung function assessments analyzed that have at least 1 effort that meets ATS/ERS criteria for acceptability will be considered acceptable and contribute to the post-dose assessments. If the PFT assessments at a specific timepoint were deemed to be of unacceptable quality, i.e., none of the efforts met ATS/ERS criteria for acceptability, the PFT assessments obtained at the timepoint will not be included in any efficacy analysis and will be considered missing (Miller et al. 2005). Thus, all observed data will be included in the ITT Analysis Set analysis, with the exception of data at a timepoint which had unacceptable quality based on ATS/ERS criteria.

### 7.2 Subject Disposition

A disposition table for all screened subjects will be provided (*Table 1.1.1 and Listing 1.2*). This tabulation will include the number of subjects in each randomized treatment who received study drug, who were withdrawn prematurely, and who completed each treatment. The number of subjects who completed the study will also be provided. The number and percentage of screened subjects who were included in the ITT, mITT, Safety and Not Randomized Analysis Sets will also be tabulated (*Table 1.1.1*).

A summary of reasons subjects were not randomized, as reported for inclusion/exclusion criteria violated, will be provided for all subjects not randomized (*Table 1.1.2*). A listing of reasons subjects were not randomized will be provided (*Listing 1.4*). Subjects discontinued from study drug will be withdrawn from the study. Reasons for Premature discontinuation will be summarized for the ITT Analysis Set by randomized treatment (*Table 1.2.1*). The number and percentage of subjects in the mITT and Safety Analysis Sets withdrawn for each reason for withdrawal will be tabulated by treatment actually received (*Tables 1.2.2 and 1.2.3*).

The number and percentage of randomized subjects who were in each of the analysis sets will be tabulated for each treatment - i.e. for the set of subjects who were randomized to receive the treatment (*Table 1.3*).

The reason for exclusion from the mITT Analysis Set will be tabulated by study drug for all ITT subjects (*Table 1.4*). The reasons for exclusion from the ITT and mITT Analysis Sets of a subject or of partial data for a subject will be listed for all randomized subjects, in addition to listing reasons for any subjects to have been excluded from the Safety Analysis Set (*Table 1.1.3*). A listing of subjects who did not comply with the use of rescue medication and xanthine-containing products (protocol deviations requiring removal of data from the mITT Analysis Set analysis) just prior to spirometry will be provided in *Listing 6.1*. Use of Ventolin HFA (hereafter referred to as Ventolin) at pre-dose or during the post-dose assessments on each specific test day (yes/no), will




be provided in *Listing 6.4*. In addition, the eligibility information (inclusion/exclusion criteria with any waivers granted), of all subjects who are randomized will be listed (*Listing 2*). Subject visits where the stability criteria were not met will be listed (*Listing 6.2*).

If there are any subjects who took study drug other than what was randomized during the study, both the treatment assigned at randomization and actual treatment(s) received during the Treatment Period will be listed (*Listing 1.3*). All data listings will show the treatment actually received.

### 7.3 Demography

The demographic variables are age, gender, race, ethnicity, smoking status (current [a disallowed category], non-smoker, or former smoker), number of years smoked (for former smokers), average number of cigarettes smoked per day (for former smokers), number of pack years smoked (for former smokers), and prior asthma treatment regimen (SABA prn use only, ICS, ICS/LABA). The physical characteristics variables are weight, height, and BMI (body mass index). The data handling rules for age, BMI, and number of pack years smoked are described in Appendix 1.

Subject demographics and smoking status/history will be summarized for the mITT, ITT, and Safety Analysis Sets and for Non-Randomized subjects (*Tables 1.5.1 through 1.5.4, respectively, and Listing 1.2*) for all subjects.

### 7.3.1 Asthma History, Screening/Baseline Spirometry, and Reversibility

The number of months since the date of the diagnosis of asthma as shown on the Screening Visit 1 eCRF, and determined relative to the first dose of study drug in the study (Appendix 1) will be summarized for the mITT and Safety Analysis Sets (Tables 1.6.1 through 1.6.2 respectively, and Listing 4.1). The screening and baseline spirometry variables FEV<sub>1</sub>, FEF<sub>25-75</sub>, and FVC will be summarized separately for Visit 1 and Visit 2 (Tables 1.7.1 and 1.7.2, respectively, for the mITT and ITT Analysis Sets, and Listing 6.4). For this purpose, Visit 1 will be Visit 1, 1a, or 1b, whichever visit had the highest FEV<sub>1</sub> result post-dose.

Per Protocol Section 4.1, reversibility to Ventolin (SABA) will be evaluated at Visits 1, 1a (if needed), or 1b (if needed) and defined as:

The comparison of the best FEV<sub>1</sub> effort obtained at 30 minutes pre-bronchodilator to the best FEV<sub>1</sub> effort obtained at 30 minutes post-bronchodilator following administration of Ventolin. A subject is considered reversible to Ventolin if the improvement in FEV<sub>1</sub> at 30 minutes post-Ventolin is ≥15%.

See Appendix 1 for data handling rules and the formula for determination of reversibility variables.

Reversibility to Ventolin at Screening will be summarized for the mITT and ITT Analysis Sets and listed (*Tables 1.8.1 and 1.8.2, respectively, and Listing 3*). Also included will be a summary of the change in FEV<sub>1</sub> from pre-bronchodilator to post-bronchodilator.



Last Revision Date: 13 Mar 2018 

## 7.3.2 Medical and Surgical History at Screening, Pregnancy Testing at Screening and Baseline

Medical history at Screening will be coded using the version of the Medical Dictionary for Regulatory Activities (MedDRA) that is current at the time of data base lock.

Medical and Surgical History at Screening will be summarized by actual treatment for the Safety Analysis Set and listed for all randomized subjects (*Table 1.9 and Listing 4.2*).

Pregnancy Testing Results from Screening and Baseline will be listed (Listing 4.3).

### 7.3.3 Prior, Concomitant, and Post-Treatment Medications/Treatments

All prescription and over-the-counter (OTC) medications, as well as any herbal or vitamin supplements, taken by the subject within 30 days of Visit 1 will be recorded on the Prior and Concomitant Medications eCRF page. All concomitant medications taken during the study will be recorded on the Prior and Concomitant Medications eCRF page.

**Coding:** Verbatim medication/treatment terms coded by will be assigned a preferred term and an ATC (anatomic therapeutic chemical class) term using the latest version of the World Health Organization Drug Dictionary Enhanced and World Health Organization Herbal Dictionary (WHO DDE and WHO HD) available (Version: Q3; 2017 or later).

**Multiple ATC Assignments:** If there are multiple ATC codes assigned to the same concomitant medication, the "primary" one based on an AstraZeneca medical evaluation will be used.

Additional details for the definition of **Prior medication/treatment**, Concomitant medication/treatment, and Post-Treatment medication/treatment are described in Appendix 1.

Concomitant asthma and non-asthma related medications/treatments will be summarized by preferred term and actual treatment received for the Safety Analysis Set separately during the Treatment and Washout Periods (*Tables 1.11.1a, 1.11.1.b, 1.11.2a, and 1.11.2b*). Prior, concomitant, and post-treatment medications will be displayed in separate listings for Asthma and Other medications (*Listings 4.4 and 4.5, respectively*).

Reported prior medication for asthma and other indications will be tabulated for all subjects (*Tables 1.10.1 and 1.10.2*) and listed separately (*Listings 4.4 and 4.5, respectively*).

Ventolin or Pulmicort dispensing will be listed (*Listing 5.1.2*).

### 7.3.4 Extent of Exposure to Study Drug

A listing of treatment dosing information will be provided in Listings 5.1.1 and 5.2. Any comments related to study drug or any other study comments will be listed (Listing 9.3).

Last Revision Date: 13 Mar 2018


### 7.4 Efficacy Analyses

Reasons for missed visits (asthma-related or not) for each subject will be listed (*Listing 6.3*). Spirometry measurements will be listed (*Listing 6.4*).

### 7.4.1 Primary Efficacy

### 7.4.2 Study Day

Study day is defined relative to the date of the first study drug administration. Within-period study day, or day of assessment/event, is defined relative to the date of study drug within the period. Additional definitions are provided in Appendix 1. Handling of unscheduled visits for efficacy endpoints is discussed in Section 7.4.3.3.

### 7.4.3 Time Points and Time Intervals for Efficacy Endpoints

The definitions of several terms related to time points and time intervals for efficacy endpoints are given in this section.

### 7.4.3.1 Baselines for Analysis

Since pre-dose values are known to be variable and an isolated timepoint may not accurately reflect the true baseline, the following baseline will be used for the statistical analyses of study assessments unless otherwise specified: the mean of available pre-dose values on the first day of each treatment cycle, i.e., the mean of pre-dose values at Visits 2, 3, 4, 5, and 6, where the mean of the 60- and 30-minute pre-dose value for each visit is obtained and then the visit means are averaged.

### 7.4.3.2 Change from Baseline

Change from baseline denotes the value at a timepoint minus the value at baseline, where baseline was defined in the previous subsection.

### 7.4.3.3 Handling of Unscheduled Visits:

Data from unscheduled visits will not be used for efficacy analyses, but will be listed (Listing 6.4).

### 7.4.3.4 Time Windows for Spirometry Assessments

All available data with the actual timepoints (versus nominal timepoints) will be used for AUC calculations, determination of peak change from baseline in  $FEV_1$ , re sponders analyses, onset of response, and offset of response. Time windows will apply only to the change from baseline in  $FEV_1$  by-timepoint analysis.



Last Revision Date: 13 Mar 2018 

### 7.4.4 Primary Efficacy Analysis

The primary objective of this study is to confirm the dose of albuterol delivered from AS MDI that is comparable to Proventil.

The  $FEV_1$   $AUC_{0-6}$  is the area under the curve for the change from baseline in  $FEV_1$  calculated using the trapezoidal rule. All observed data will be utilized with the trapezoidal rule to calculate



Protocol No. PT007001

Last Revision Date: 13 Mar 2018


AUC. For the purpose of AUC calculations, the value of the spirometry parameter at time 0 will be the change from baseline in pre-bronchodilator  $FEV_1$  at the visit. To aid in interpretation, all AUC values will be normalized by dividing the AUC by the time from the first to the last non-missing value (typically 6 hours). If AUC is based on just one 1 assessment (i.e., a change from baseline value), that change from baseline value will be the value of the AUC (the trapezoidal rule and normalization will not apply as the area is 0 and the time interval is 0).

The FEV<sub>1</sub> AUC<sub>0-6</sub> will be analyzed using a linear mixed model with a random subject effect. The fixed effects in the model will include treatment, treatment sequence, baseline FEV<sub>1</sub>, and period. An ICS use subgroup analysis will be based on a linear mixed model with covariates of treatment, treatment sequence, baseline FEV<sub>1</sub>, period, ICS Use subgroup (ICS use at Screening and Did not use ICS at Screening), and treatment-by-subgroup interaction.

The least squares (LS) mean and the standard error of this mean with the corresponding two-sided 95% confidence interval will be provided for each treatment based on the overall study population and then separately within each of the 2 ICS subgroups. The estimated treatment differences and 95% CIs will be provided for all treatment comparisons based on the overall study population, and then separately within each of the 2 ICS Use subgroups.

Superiority comparisons of AS MDI relative to Placebo MDI and Proventil versus Placebo MDI will be conducted first using a dose-ordered approach. A two-sided alpha level of 0.05 will be employed. Estimated treatment differences and 95% confidence intervals (CIs) will be provided for the superiority comparisons. As described in detail in Section 4.3, the superiority of Proventil relative to Placebo MDI will be tested first using this dose-ordered approach. If Proventil 180 µg is superior to Placebo MDI, AS MDI 180 µg will be compared to Placebo MDI. If AS MDI 180 µg is superior to Placebo MDI, the superiority of the Proventil 90-µg dose relative to Placebo MDI will be tested. If Proventil 90 µg is superior to placebo, then AS MDI 90 µg will be compared to Placebo MDI.



Comparisons among the dose levels within a product and comparisons within the ICS Use subgroups will be conducted for exploratory purposes. Estimated treatment differences and 95% CIs will be provided.

The primary analysis will be conducted using the mITT Analysis Set. Supportive analyses for the primary endpoint will be performed using the ITT Analysis Set. Assumptions underlying the primary analysis will be evaluated and additional analyses may be performed (see Section 7.4.7).




Summary statistics and the results of statistical testing for the primary endpoint will be provided in *Table 2.1.1* by treatment overall and for each subgroup for the mITT Analysis Set and in *Table 2.1.2* for the ITT Analysis Set.

### 7.4.5 Secondary Efficacy

The secondary endpoints will be analyzed using a similar approach as that of the primary endpoint. Linear mixed models will be fit with a random subject effect. The fixed effects in the model will include baseline FEV<sub>1</sub>, treatment, treatment sequence, and period.

The FEV<sub>1</sub> AUC<sub>0-4</sub> will be calculated in a similar manner as FEV<sub>1</sub> AUC<sub>0-6</sub>; however, the trapezoidal rule will only be implemented through the 4-hour nominal timepoint. The AUC values will be normalized accordingly.

The peak change from baseline in FEV<sub>1</sub> will be calculated using the largest FEV<sub>1</sub> value measured during the 6 hours post-dosing.

Secondary efficacy endpoints will be analyzed using the mITT Analysis Set. Tables and figures will be as follows:

- Change from baseline in FEV<sub>1</sub> AUC<sub>0-4</sub>: Table 2.2.1 for the mITT Analysis Set.
- Peak change from baseline in FEV<sub>1</sub>: Table 2.2.2 for the mITT Analysis Set.

### 7.4.6 Other Efficacy

Change from baseline in  $FEV_1$  at each post-dose timepoint will be presented graphically by treatment and will be analyzed using a linear mixed model with a random subject effect. The fixed effects will include treatment, time point, treatment-by-time point interaction, treatment sequence, baseline  $FEV_1$ , and period. The covariance within subject-periods will be unstructured over the time points. Note that the sample sizes (N) at 180- and 300-minutes post-dose will be smaller than the remaining timepoints due to adjustment to the spirometry assessment schedule outlined in Version 2 of the protocol (See Section 8).

The median values for time to peak FEV<sub>1</sub> will be reported by treatment. The median differences and corresponding Hodges-Lehmann 95% CIs will be presented for pairwise comparisons among the treatments.

The percentages of subjects achieving a 12% and 15% improvement from baseline within 30 minutes post dose will be tabulated by treatment. Responders will be defined as subjects achieving  $\geq$ 15% (or  $\geq$ 12%) improvement in FEV<sub>1</sub> within 30 minutes after dosing. The odds of being a responder will also be estimated using a generalized mixed effects model with fixed effects of treatment and period, and a random subject effect.

The time to onset of response for each individual subject will be defined as the first timepoint for which an increase from baseline FEV<sub>1</sub> of at least 15% (or 12%) is observed within the first 30 minutes post dose. The median time to onset of response will be reported by treatment. The

## AstraZeneca

Statistical Analysis Plan Protocol No. PT007001

Last Revision Date: 13 Mar 2018


median differences and corresponding Hodges-Lehmann 95% CIs will be presented for pairwise comparisons among the treatments (Han L, Paper ST-154). Only subjects who achieved the 15% (or 12%) improvement within the first 30 minutes post dose will be included in this analysis.

The duration of response for each subject will be defined as the time from onset of at least a 15% (or 12%) increase in FEV<sub>1</sub> to the offset of the 15% (or 12%) increase in FEV<sub>1</sub> relative to baseline. If offset of response was not achieved during the assessment period, the last available time of assessment will be used as the offset. If a subject had a 2<sup>nd</sup> onset of response subsequent to achievement of offset, their data for that period will be excluded from the duration of response analysis. Descriptive statistics including the N, arithmetic mean, standard deviation, median, minimum, and maximum for duration of response will be reported by treatment. The duration of response will be analyzed using a linear mixed effects model similar to that of the primary endpoint or a distribution-free method (Hodges-Lehmann) as appropriate to the data. As an additional sensitivity analysis to assess potential bias imposed by the limited spirometry sampling scheme of protocol Version 1.0, the duration of response analysis will be repeated excluding those subjects who are missing the 180- and 300-minute post timepoints.

The other efficacy endpoints will be analyzed using the mITT Analysis Set. Tables and figures will be as follows.

- Change from Baseline in FEV<sub>1</sub> at each post-dose timepoint: *Table 2.3.1 and Figures 2.3.1.1* and 2.3.1.2 for the mITT Analysis Set.
- Time to peak FEV<sub>1</sub>: Table 2.3.2 for the mITT Analysis Set.
- Percentage of subjects achieving 12% improvement in FEV<sub>1</sub> from baseline within 30 minutes of dose: *Table 2.3.3 for the mITT Analysis Set*.
- Percentage of subjects achieving 15% improvement in FEV<sub>1</sub> from baseline within 30 minutes of dose: *Table 2.3.3 for the mITT Analysis Set*.
- Time to onset of response: Table 2.3.4 and Table 2.3.5 for the 12% Improvement in  $FEV_1$  and the 15% Improvement in  $FEV_1$ , respectively, for the mITT Analysis Set.
- Duration of response: Tables 2.3.6, 2.3.7, 2.3.8, and 2.3.9 for the 12% Improvement in FEV<sub>1</sub>, 12% Improvement in FEV<sub>1</sub> in subjects who have assessments at the 180- and 300-minute post-dose timepoints, 15% Improvement in FEV<sub>1</sub>, and 15% Improvement in FEV<sub>1</sub>, in subjects who have assessments at the 180- and 300-minute post-dose timepoints, respectively, for the mITT Analysis Set.

### 7.4.7 Data Validation and Transformation

In general, the distribution of spirometry measures is well approximated by a normal distribution. Under some circumstances, however (eg, during an exacerbation unrelated to treatment), extreme and atypical values can arise. Such values have high influence on estimation of variance parameters and on standard errors of fixed effect estimates. The distribution of scaled marginal residuals, and influence statistics will be examined to identify such cases. In the event that a single or small number of such outlying values are found to exist and found to be highly influential, the




effects may be ameliorated by either transformation or removal of the outlier. Transformations to be considered may include the logarithmic transformation or normal rank transformations. Where outliers are removed, sensitivity analyses including those values will be reported.

The assumption of normality in the primary, secondary, and other efficacy endpoints, Change from Baseline in FEV<sub>1</sub> AUC<sub>0-6</sub>, Change from Baseline in FEV<sub>1</sub> AUC<sub>0-4</sub>, Peak change from baseline in FEV<sub>1</sub>, and duration of response will be checked by visually inspecting the distribution of the scaled (decorrelated) residuals. Also, model fit and the assumption of homogeneity of variance among treatments will be verified by inspection of scatter plots of predicted vs. residuals, residuals vs. treatment, and by box plots of residuals for treatment. Plots for scaled (marginal) residuals will be prepared using option=VCIRY on the model statement and the ODS graphics option. If the assumption of homogeneity does not hold (sample variances appear heterogeneous), then the final model will be fit with an UN or CSH covariance structure. (Appendix 3).

Changes in spirometry measures from baseline, and from timepoint to timepoint will be examined graphically before database lock, and before unblinding, as part of data quality management.

### 7.5 Safety Analyses

All safety analyses are based on Safety Analysis Set. Hypothesis testing will not be performed for any safety analyses. No formal statistical analysis of safety data is planned. Safety data will be summarized by treatment and listed.

### 7.5.1 Adverse Events

Adverse events will be collected and coded using the latest version (20.1 or later) of the MedDRA available. A glossary of MedDRA preferred terms used for AEs reported in the study along with the associated Investigator's verbatim will be provided in Listing 7.2. The version of MedDRA current at the time of database lock will be used for the final analysis of data.

Adverse events occurring from the time the subject signs informed consent until the subject is randomized will be summarized as medical history and not as an AE unless the event meets the definition of an SAE as defined in Protocol Section 6.2.

An adverse event is considered treatment-emergent if the date of onset is on or after the date of first dose of study drug in the study. An AE would be considered attributable to a treatment (corresponding to a treatment period or washout or final follow-up period) if the onset of the AE was during a treatment period (or washout period or final follow-up period). Should there not be sufficient information to determine during which period that an AE started, the AE will be counted as having occurred in all treatment periods (and washout periods or final follow-up period) prior to the end date of the AE if this is reported as long as the subject received study drug during those treatment periods. If both start and end date of an AE are unavailable, the AE will be counted in all treatment periods prior to the date of last contact on the End of Treatment eCRF (including the treatment taken on the day of the last contact) as long as the subject received study drug during those treatment periods. Any AE with onset after the last treatment in the study will be attributed to this last treatment. Adverse events after the Follow-up Telephone Call scheduled 3-7 days after

### Statistical Analysis Plan Protocol No. PT007001



Last Revision Date: 13 Mar 2018


Visit 6 or a discontinuation visit will not be considered treatment-emergent, but will be listed in adverse event data listings.

# Counting Rules for Adverse Events with Onset in a Treatment Period or Washout Period (or Follow-up Period):

- 1. A subject with more than 1 different AE in a particular system organ class (SOC) will be counted only once in the total of subjects experiencing AEs in that particular SOC.
- 2. A subject having experienced the same event (AE preferred term) more than once will be counted only once in the number of subjects with that event.

**Events with Irregular Start Dates**: All adverse events will be included in the tabulations regardless of the completeness of the onset dates.

Missing/incomplete (partial) AE start and end dates will not be imputed for data listings.

Both the treatment and the washout periods include treatment with Pulmicort Flexhaler if subjects were previously on an ICS prior to the start of the study. Additionally, the washout periods included treatment with Ventolin. AEs reported as starting during a Washout Period or the final follow-up period will be excluded from the main analyses of AEs. As a supportive analysis, AEs will be assigned to the last randomized treatment received including those occurring during the Washout Period (*Table 3.2.2 for AEs and Table 3.6.2 for SAEs*).

All adverse events, whether treatment-emergent or not, will be included in the listings. Reported adverse events by system organ class, preferred term, treatment, center, subject, and onset day will be provided (*Listing 7.1*). Reported adverse events by treatment, center, subject, and onset date will also be provided (*Listing 7.3*).

The listing of adverse events will provide the severity, maximum severity, relationship to study drug, action taken and outcome for each adverse event. Any SAEs reported will be listed (*Table 3.7.1 for the treatment period analysis not including the washout and follow-up period and Table 3.7.2 for the analysis including all AEs including those with onset during the washout or follow-up period after the treatment period)*. Suspect drug assessment data associated with an SAE (collected on the Suspect Drug Assessment CRF) will be listed by SAE (*Listing 4.6*). Adverse events leading to discontinuation of study drug will be listed (*Table 3.5*). A listing of any reported deaths during the study will be provided (*Table 3.10*); the study drug taken most recently prior to the death and the number of days since the dose of this study drug at the time of the death will be included in the listing.

An overview summary table will be prepared. The table will provide the incidences of subjects, for all subjects and for each treatment, with the following: at least 1 treatment-emergent adverse event, at least 1 treatment-emergent related adverse event, at least 1 treatment-emergent serious adverse event, at least 1 treatment-emergent serious related adverse event, at least 1 treatment-emergent adverse event leading to study drug discontinuation and premature study withdrawal, and




a report of death (Table 3.1.1, washout TEAEs excluded). As a supportive analysis, AEs will be assigned to the last randomized treatment received including those occurring during the washout period or the final follow-up period (Table 3.1.2).

The incidence of an adverse event (AE) for a treatment will be defined as the number and percent of subjects experiencing an event attributable to that treatment. For each group, the following will be prepared for each treatment and for overall, for each primary system organ class, and for each preferred term within a system organ class:

- 1. The incidence of all treatment-emergent adverse events (*Table 3.2.1*)
- 2. The incidence of non-serious treatment-emergent adverse events occurring in  $\geq 5\%$  of subjects in a treatment (Table 3.2.4)
- 3. The incidence of all treatment-related treatment-emergent adverse events (*Table 3.3*)
- 4. The incidence of treatment-emergent adverse events leading to study drug discontinuation (*Table 3.4*)
- 5. The incidence of treatment-emergent serious adverse events (*Table 3.6.1*)
- 6. The incidence of treatment-emergent serious related adverse events (Table 3.8)
- 7. The incidence of all treatment-emergent adverse events by highest severity (Tables 3.9.1-3.9.5). There will be a separate table for each treatment.
- 8. The incidence of treatment-emergent adverse events occurring in at least 2% of subjects in any treatment (*Table 3.2.3*, sorted by descending frequency of events in a preferred term).

### 7.5.2 **Clinical Laboratory Data**

Clinical safety laboratory tests will be collected at Visit 1, Visit 6 (post-dose) and during a Premature Discontinuation Visit, if applicable. Laboratory tests will be analyzed by a central laboratory according to standardized, validated assays. The following clinical laboratory parameters that will be assessed are noted in Table 5.

Table 5 Lab Parameters

| Hematology | |
|---|---|
| Hemoglobin | Mean corpuscular hemoglobin (MCH) |
| Hematocrit | Mean corpuscular hemoglobin concentration (MCHC) |
| White Blood Cell count with differential | Mean corpuscular volume (MCV) |
| Red Blood Cell count | |
| Platelet Count | |
| Clinical Blood Chemistry | |
| Liver Enzyme and Other Function Tests | Other Clinical Blood Chemistry |
| Alanine aminotransferase (ALT) | Albumin |
| Aspartate aminotransferase (AST) | Blood urea nitrogen (BUN) <sup>a</sup> |
| Alkaline phosphatase | Calcium <sup>a</sup> |



### Statistical Analysis Plan Protocol No. PT007001

Last Revision Date: 13 Mar 2018


Bilirubin, total

Chloride

Cholesterol

Bicarbonate

Creatinine

Glucose

Magnesium

Potassium

Phosphate

Protein, total

Sodium

Triglycerides

Urea

### Other Tests:

Pregnancy test (women of child-bearing potential only): serum (human chorionic gonadotropin [hCG]) at Visit 1, and urine HCG before randomization at Visit 2, as detailed in Table 1

Creatinine clearance will be estimated by the central laboratory at Screening only using eGFR (estimated glomerular filtration rate) using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) published formula.

Clinically Significant Laboratory Abnormalities as identified by the investigator after the start of study drug will be recorded as an Adverse Event and tabulated as an AE in the AE analysis. Abnormalities occurring prior to the start of treatment will be noted in medical history and presented in a data listing. Per protocol, the criteria for a "clinically significant" laboratory abnormality are:

- a. A laboratory abnormality that leads to study drug dose suspension or discontinuation
- b. A laboratory abnormality that results in any therapeutic intervention (i.e., concomitant medication or therapy)
- c. Any other laboratory abnormality judged by the Investigator to be of any particular clinical concern (eg., significant fall in hemoglobin not requiring transfusion)

For laboratory abnormalities that do not meet the above criteria but are outside of the normal reference range, the investigator should indicate whether the value is clinically significant or not clinically significant for the subject.

All laboratory data will be stored in the database with the units in which they are originally reported. Laboratory data in subject data listings will be presented in the International System of Units (SI units; Système International d'Unités) where available. Laboratory data not reported in SI units will be converted to SI units before further processing or data analysis. Individual clinical laboratory variables for hematology and clinical chemistry, including creatinine clearance (eGFR), will be provided in listings (Listing 8.1 for central laboratory hematology, Listing 8.2 for central

<sup>&</sup>lt;sup>a</sup> Parameters included in the Basic Metabolic Panel (BMP).


laboratory blood chemistry and kidney function, and Listing 9.3 for pregnancy test results after the start of treatment). Comments for central laboratory testing will be listed (Listing 8.3). For listings, laboratory values will be flagged as Low or High based on the reference ranges provided by the central laboratory, Covance. These flags along with the reference ranges will be provided in the laboratory data listings.

### 7.5.3 Vital Signs

A Clinically Significant Abnormality in vital signs identified by the investigator will be recorded as an Adverse Event if it occurs after the start of treatment. These adverse events will be included in the AE summaries; abnormalities prior to the start of treatment will be noted in medical history and listed.

Potentially clinically significant changes in systolic blood pressure (SBP), diastolic blood pressure (DBP), and Heart Rate will be defined based on the following criteria provided by AstraZeneca:

Table 6 Potentially Clinically Significant Criteria for Systolic and Diastolic Blood Pressure Parameters and Heart Rate

| Parameter (mmHg) | Post-Baseline Criteria |
|-------------------|------------------------------------------------------|
| SBP, increase | ≥180 and increase from baseline ≥20 |
| SBP, decrease | ≤90 and decrease from baseline ≥20 |
| DBP, increase | $\geq$ 105 and increase from baseline $\geq$ 15 |
| DBP, decrease | $\leq$ 50 and decrease from baseline $\geq$ 15 |
| Tachycardia Event | $\geq$ 110 bpm and increase $\geq$ 15% from baseline |
| Bradycardia Event | $\leq$ 50 bpm and decrease $\geq$ 15% from baseline |

Vital signs, height, weight, BMI, SBP, DBP, and Heart Rate will be listed (Listing 9.1).

Baseline is defined as the last pre-dose measurement taken prior to dosing on Day 1 of a treatment period.

Change from baseline for a timepoint of a Treatment Period is defined as the vital sign value for the timepoint minus the baseline value.

For summaries by timepoint, the latest vital sign value (in the case of multiple values) for a scheduled post-baseline timepoint on a scheduled visit for a Treatment Period will be employed.

Descriptive statistics (mean, median, standard deviation, and range) for change from baseline will be tabulated by vital sign parameter and treatment for each scheduled assessment time.






Summary statistics (n, mean, median, standard deviation, minimum and maximum) of scheduled pre-dose and post-dose values as well as changes from baseline for each vital sign parameter will be tabulated by treatment (*Table 3.11.1*). Values will not be allocated across Treatment Periods.

### 7.5.4 Electrocardiogram (ECG)

A Clinically Significant Abnormality for a 12-Lead ECG measurement identified by the investigator as a clinically significant abnormality will be recorded as an Adverse Event if it occurred after the start of study drug. These adverse events will be included in the AE summaries.

The ECG parameters that will be assessed include heart rate (HR), RR interval, PR interval, QRS axis, QRS interval, QT interval, and QTcF (Fridericia's Formula) interval. The QTcF (Fridericia Corrected QT) is defined as [QT/(RR<sup>1/3</sup>)].

All 12-Lead ECG measurements for the Safety Analysis Set will be listed (*Listing 9.2*).

### 7.5.5 Physical Examination

Any physical examination abnormality reported after the start of treatment for a subject is to be reported as an adverse event and included in the AE summaries.

### 8. CHANGES FROM METHODS PLANNED IN THE PROTOCOL



. All subjects will be included in the efficacy analyses irrespective of their spirometry sampling scheme.

The protocol specified that the baseline for vital signs analyses would be the average of the vital sign values taken prior to dosing on the day of randomization. Since multiple values were not scheduled to be collected at randomization and since each treatment visit had vital signs measurements taken prior to dosing (under the condition that restricted asthma medications were not to be taken within 6 hours of test day assessments), the baseline for vital signs has been updated as follows: Baseline is defined as the last pre-dose measurement taken prior to dosing on Day 1 of a treatment period.

### 9. STATISTICAL SOFTWARE

Data processing, statistical screening, descriptive reporting, and analysis of the efficacy and safety data will be performed using SAS (Version 9.4 or higher).




### 10. REFERENCES

Miller et al 2005. Miller MR, Hankinson J, Brusasco V, et al. Standardisation of spirometry. Eur Respir J 2005;26(2):319-338.

Han L, Calculating the point estimate and confidence interval of Hodges-Lehmann's median using SAS® software. Southeast SAS® Users Group (SESUG) 2008; Paper ST-154.



### **APPENDIX 1 DATA HANDLING RULES**

Programming of the tables, listings and figures will be performed using SAS Version 9.4 or a more recent version. The following table presents algorithms (not stated elsewhere) to be used in SAS to calculate the derived variables, including rules for handling missing data or partial dates, or irregular/unexpected data issues.

| Category | Description | Data Handling Rules |
|---|---|---|
| Pulmonary<br>Function<br>Testing Data | data transferred | <ul> <li>Only data of rank =1 (best effort) will be transferred; data transferred will be grade 1 = acceptable, grade 2 = borderline, or grade = 3 (unacceptable). Only data of grade = 1 or grade = 2 will be included in baseline or on-treatment spirometry calculations.</li> <li>All data transferred from</li></ul> |
| Age (years) | Age (years) | Age = integer part of ((Visit 1 date – Birth date + 1)/365.25) |
| Smoking<br>History | Number of pack years smoked | Number of pack years smoked = (number of cigarettes per day/20) x number of years smoked. It is zero if the number of years smoked is zero or if the subject is a non-smoker. |
| BMI | Body Mass Index | $BMI = (weight(kg))/(height(cm)/100)^2$ |
| Asthma History | Months Since Diagnosis | Months Since Diagnosis = (Date of First Dose of Study Drug in the study – Date Asthma First Diagnosed)/30.475. |
| | Missing Date Asthma First<br>Diagnosed | Day of Diagnosis will be imputed for all subjects as the 1st of the month. |
| | Missing month of Date<br>Asthma First Diagnosed | Missing month of Diagnosis will be imputed as June, or the month in which 1st will be the latest before informed consent date, whichever is earliest. |
| Medical<br>History | Medical History Begin<br>Date of Condition | Missing month of Condition will be imputed as June, or the month in which 1 <sup>st</sup> will be the latest before informed consent date, whichever is earliest. Begin date of Condition will be imputed for all subjects as the 1 <sup>st</sup> of the month. |




| Category | Description | Data Handling Rules |
|---|---|---|
| | Medical History End Date of Condition | Other than for 'Ongoing' conditions, missing month of End Date of Condition will be imputed as June, or the month in which 1 <sup>st</sup> will be the latest before informed consent date, whichever is earliest. End date of Condition will be imputed for all subjects as the 1 <sup>st</sup> of the month. |
| Surgical<br>History | Surgical History Date of<br>Surgery | Missing month of Surgery will be imputed as June, or the month in which 1 <sup>st</sup> will be the latest before informed consent date, whichever is earliest. Begin date of Surgery will be imputed for all subjects as the 1 <sup>st</sup> of the month. |
| Screening<br>Reversibility | Screening Percent Reversibility | The screening percent reversibility to Ventolin is $100 \text{ x}$ [post-Ventolin FEV <sub>1</sub> – pre-Ventolin FEV <sub>1</sub> )]/ [pre-Ventolin FEV <sub>1</sub> ]. For this definition, "post-Ventolin FEV <sub>1</sub> " and "pre-Ventolin FEV <sub>1</sub> " are the best effort values obtained after the dose of Ventolin and before the dose of Ventolin, respectively. |
| First and Last<br>Treatment<br>Dates | Date/time of first dose of<br>the first study drug taken<br>in the study and the<br>date/time of the last dose<br>of the last study drug taken<br>in the study. | The date and time (24 hr. clock) of the dose of study drug will be taken from the Study Drug Administration eCRF. The time of the last dose of study drug will be the last time of dosing from the dataset. |
| Last Visit Date | Date of Last Visit | Date of last Visit according to the Visit eCRF. |
| Last Study Participation Date (STDM variable, RFPENDTC) | Last Study Participation Date (STDM variable, RFPENDTC) | Last study participation date is defined as last known date of contact which would be the later of the following dates: last visit date, date of the last dose, date of last contact if lost-to-follow-up, date of telephone follow-up, or death date. |
| Study Day<br>Definitions | Study Day for<br>assessment/event which<br>occurs on or after the date<br>of a study drug | Study Day = Date of assessment/event – date of the dose of study drug + 1. |
| | Within-Period Study Day<br>for an on-treatment<br>assessment/event study | Within-Period Study Day = Date of assessment/event – date of dose of study drug within the respective Treatment Period + 1. |



| ic. 15 Wiai 2010 |
|------------------|

| Category | Description | Data Handling Rules |
|---|---|---|
| | drug | |
| | Study Day for<br>assessments/events on<br>days prior to the dose of<br>the first study drug in the<br>study | Study Day = date of assessment/event - dose date of treatment in the study. |
| | Study Day Post-<br>Treatment of Assessment<br>or event which occurs after<br>a study drug | Study Day = 'P' concatenated with the number of days post-treatment that the assessment or event occurred which is defined as Date of assessment/event – date of dose of study drug in the last period (i.e. most recent treatment). |
| | Study Day of<br>Randomization | Study Day of Randomization = date of randomization – date of the first dose of study drug in the study if date of randomization is before date of first dose of study drug. Study Day is 1 if the day of first study drug in the study is on the day of randomization. |
| | First Dose Date | <b>First Dose Date</b> in the study is defined as the date of the first dose of study drug in the study. |
| | Last Dose Date | Last Dose Date in the study is defined as the date of the last dose of study drug in the study (defined as the last date of dosing from the Study Drug Administration eCRF). |
| | Last Study Day | For subjects who did not receive study drug in the study (e.g., Non-Randomized Subjects), Last Study Day is defined as (the later of the last visit date or the date of last contact for subjects lost-to-follow-up from the End of Treatment eCRF) – Date of Screening Visit + 1. |
| | | For subjects who received study drug in the study, Last Study Day is defined as (the later of the last visit date or the date of last contact for subjects lost-to-follow-up from the End of Treatment eCRF) – first dose date in the study + 1. |




| Category | Description | Data Handling Rules |
|---|---|---|
| | Days Since Last Dose for event (e.g., Death) | Days Since Last Dose is defined as date of event – date of last dose of study drug. |
| | Treatment Day | Treatment Day 1 is the study day of the dose of a study drug. |
| Treatment<br>Period | Treatment Period | A treatment period for a treatment is the date of the dose of the treatment (Treatment Day 1 of a treatment) |
| Duration of<br>Event | The duration of any event (not including duration of asthma) | The duration of any event is defined as (stop date – start date + 1). |
| Duration of<br>Asthma | Duration of asthma (months) | The duration of asthma = (first dose date of study drug – date asthma first diagnosed)/30.475, where the day of asthma diagnosed is assumed to be the 1 <sup>st</sup> of the month. |
| Multiple | Vital Signs assessments | All data will be listed in data listings. |
| Assessments for<br>the Same Visit | | The last non-missing assessment of multiple valid assessments within a pre-dose or post-dose study time window will be used for summaries |
| Spirometry<br>Assessments | Spirometry assessments | The last of multiple valid assessments within a post-baseline study time window will be used for summaries and statistical testing, except for AUC parameters, where all post-baseline assessments in the study time window will be used. |
| Tine to onset of response | Time to onset of response | Time to Onset of Response (minutes) = (time of first achievement of a $\geq$ 15% (or 12%) increase in FEV <sub>1</sub> from baseline, within 30 minutes of dose – treatment administration time). |
| Time to offset of response | Time to offset of response | Time to Offset of Response: For responders only: (time of first assessment after achievement of response for which the increase from baseline in FEV <sub>1</sub> is < 15% (or 12%) – treatment administration time). If offset of FEV1 < 15% (or 12%) is not achieved and the last available |




Last Revision Date: 13 Mar 2018

c. Either the medication/treatment start date or end date or both are before Visit 1.

medication/treatment taken on or after Visit 1 and on or before the date prior to the last dose of study drug for the subject. A medication/treatment will be identified as

a. Medication/treatment start date is after

b. The end date is after Visit 1 to the date

Visit 1 to the date prior to the last dose of

prior to the last dose of study drug for the

2. Concomitant medication/treatment is any

concomitant if:

study drug, or

subject, or

| Category | Description | Data Handling Rules |
|---|---|---|
| | | assessment is $\geq 15\%$ (or 12%), the time to offset will be defined as (the time of the last available assessment – treatment administration time |
| Duration of response | Duration of response | Duration of Response = time of offset of<br>Response – time of onset of Response |
| Special Lab<br>Value Handling | Lab values with a prefix such as: '>', '<', '+' and 'Less than' etc | <ul> <li>'&gt;': use the available original value +0.001 in the analyses.</li> <li>'&lt;': use the available original value -0.001 in the analyses.</li> <li>'+': use the available original value without the prefix in the analyses.</li> <li>'&gt;=': use the available original value in the analyses.</li> <li>'&lt;=': use the available original value in the analyses.</li> </ul> |
| Prior, Concomitant, and Post- treatment Medication/ Treatment | Prior, concomitant, and post-treatment medication/treatment | <ol> <li>Prior medication/treatment is any medication/treatment taken prior to Visit 1, even if this medication continued after Visit 1. A medication/treatment will be considered prior if: <ol> <li>The start and end date of the medication/treatment are missing, or</li> <li>The start date is missing and the end date is on or after Visit 1, or</li> </ol> </li> </ol> |

### Confidential and Proprietary




| | <ul> <li>c. 'Ongoing' is checked.</li> <li>3. A medication with an onset date on or after the last dose of study drug for the subject will not be considered concomitant, but will be considered a Post-Treatment medication/treatment.</li> <li>4. Any medication/treatment which cannot be identified as Prior, Concomitant, or Post-</li> </ul> |
|---|---|
| | identified as Prior, Concomitant, or Post- |
| | Treatment will be considered as being in each of the categories that are possible from the available information. |
| Missing severity | For the AE summary by severity, an AE with missing severity will be deemed as Severe. Imputed values will not be listed in data listings. |
| Missing relationship to study drug | For AE summary by relationship, an AE with a missing relationship to study drug (yes/no) will be deemed as Related. Imputed values will not be listed in data listings. |
| Treatment-emergent adverse event | An adverse event is considered treatment-<br>emergent if the date of onset is on or after the<br>date of first dose of study drug. The study site<br>will enter a new onset date when there is an<br>increase in severity or intensity for a pre-existing<br>event after the start of a study drug. |
| | <ul> <li>If the AE start date is partial/missing, then the AE is considered as treatment emergent.</li> <li>If both AE start month and day are missing and AE start year is the same or after the first dose year, then the AE is considered as treatment emergent.</li> <li>If AE start day is missing and AE start year and month are the same or after the first dose year and month, then the AE is considered as treatment emergent.</li> <li>Missing/incomplete (partial) AE start and end</li> </ul> |
| Γ | Aissing relationship to tudy drug Treatment-emergent |



Statistical Analysis Plan Protocol No. PT007001

Last Revision Date: 13 Mar 2018


| Category | Description | Data Handling Rules |
|---|---|---|
| | | dates will not be imputed for data listings. |
| Exposure (days) | Exposure (days)<br>(Treatment Duration) | Exposure is defined as the number of days at which doses were administered. |
| Hard Coding | Hard coding for data analysis | Hard Coding is not allowed during data analysis unless it is agreed to in writing by AstraZeneca. |



Statistical Analysis Plan Protocol No. PT007001

Last Revision Date: 13 Mar 2018


### **APPENDIX 2 ANALYSIS DATASET SPECIFICATIONS**

Analysis datasets will be built to gain efficiency and ensure consistency in data analyses and presentation for this trial. The specifications for each analysis data set will be prepared separately and will not be a part of this SAP.




Last Revision Date: 13 Mar 2018

### APPENDIX 3 SAS CODE FOR STATISTICAL ANALYSES

| Test | Template SAS Code for Modeling (SAS Version 9.4) |
|---|---|
| Linear Mixed Model analysis for a continuous efficacy endpoint, change from baseline in AUC <sub>0-6</sub> , change from baseline in AUC <sub>0-4</sub> , or Peak Change from Baseline in FEV <sub>1</sub> . Use this code for the analysis of the primary and secondary endpoints. | PROC MIXED PLOTS (ALL) METHOD=REML; CLASS SUBJECT PERIOD TRT SEQUENCE; MODEL Y = BASE PERIOD TRT SEQUENCE / DDFM=KENWARDROGER SOLUTION VCIRY OUTP=OUT; RANDOM SUBJECT; LSMEANS TRT / PDIFF CL ALPHA=0.05 CORR COV; ODS OUTPUT LSMEANS=MEANS; ODS OUTPUT DIFFS=DIFF; RUN; Where BASE is the baseline value of the endpoint and TRT is the treatment. THE PLOTS (ALL) OPTION FOR PROC MIXED WILL BE USED TO GET PLOTS TO PERFORM MODEL DIAGNOSTICS (for normality and heterogeneity of variance). Scaled residuals will be used. Influence statistics will be requested. If the assumption of homogeneity does not hold (sample variances appear heterogeneous), the following will replace the Random subject and ODS statements above. REPEATED TRT / TYPE=UN (or CSH) SUBJECT=SUBJECT; LSMEANS TRT / PDIFF CL ALPHA=0.05 CORR COV; ODS OUTPUT LSMEANS=MEANS; ODS OUTPUT DIFFS=DIFF; |
| Linear mixed effects model for a continuous efficacy | PROC MIXED PLOTS (ALL) METHOD=REML; CLASS SUBJECT PERIOD TRT SEQUENCE; MODEL Y = BASE PERIOD TRT TIMEPOINT TRT*TIMEPOINT SEQUENCE |
| endpoint | / DDFM=KENWARDROGER SOLUTION VCIRY |
| involving | OUTP=OUT; |
| multiple<br>measures per<br>period. Use this | RANDOM SUBJECT;<br>REPEATED TIMEPOINT / TYPE=UN SUBJECT=SUBJECT;<br>LSMEANS TRT*TIMEPOINT / PDIFF CL ALPHA=0.05 |



Last Revision Date: 13 Mar 2018 

| code for the | CORR COV; |
|---|---|
| Other Efficacy | ODS OUTPUT LSMEANS=MEANS; |
| parameter | ODS OUTPUT DIFFS=DIFF; |
| Change from | RUN; |
| Baseline in FEV <sub>1</sub> | |
| at each post-dose | Where BASE is the baseline value of the endpoint and TRT is the |
| timepoint at 5, | treatment. |
| 15, 30, 45, 60, | |
| 120, 180, 240, | One model includes all time points. |
| 300, and 360 | |
| Minutes Post | |
| Dose. | |
| Generalized | PROC GLIMMIX METHOD=QUAD; |
| mixed effects | CLASS TRT(REF=FIRST) PERIOD SUBJECT; |
| model for an | MODEL Y=TRT PERIOD / DIST=BIN LINK=LOGIT; |
| other efficacy | RANDOM INT / SUBJECT=SUBJECT; |
| categorical | LSMEANS TRT / DIFF OR; |
| endpoint, | RUN; |
| percentages of | WI TRATE I |
| subjects | Where TRT is the treatment. |
| achieving a 12% and 15% | |
| improvement | |
| from baseline | |
| within 30 | |
| minutes post | |
| dose. | |
| Non-parametric | |
| descriptive | The following macro can be used to calculate the point estimate and |
| statistics and | confidence interval of the Hodges-Lehmann's median for paired data |
| CI's of the | (Han L, Paper ST-154): |
| treatment differences for | %macro HL_paired(dsn=, trt1=, trt2=, alpha=); |
| Time to Peak | *** STEP 1: Calculate the differences between each pair of treatments |
| FEV <sub>1</sub> , Time to | for each subject and record the sample size as a macro variable for later |
| onset of | use. Note that the macro only calculates differences for 2 treatments so |
| response, and | repeat this macro as needed. |
| Duration of | DATA ONE; SET &DSN |
| response (as | CALL SYMPUT('SIZE',TRIM(LEFT(_N_))); |
| appropriate) | DIFF=&TRT1-&TRT2 |
| | RUN; |




Last Revision Date: 13 Mar 2018

\*\*\* STEP 2: Use ARRAY to form all possible ordered pairs of differences and average values;

PROC TRANSPOSE DATA=ONE OUT=TWO(DROP=\_NAME\_); VAR DIFF;

RUN;

DATA THREE; SET TWO;

ARRAY X{&SIZE} COL1-COL&SIZE;

DO I=1 TO &SIZE;

DO J= I TO &SIZE;

 $STAT = (X{I}+X{J})/2;$ 

OUTPUT;

END;

END;

\*\*\* STEP 3: Calculate the point estimate of the Hodges-Lehmann median difference;

PROC SORT DATA=THREE;

BY STAT;

RUN;

PROC MEANS MEDIAN NOPRINT;

VAR STAT;

OUTPUT OUT=EST(DROP= FREQ TYPE )

MEDIAN=ESTIMATE;

RUN;

\*\*\* STEP 4: Calculate the confidence interval of the Hodges-Lehmann median difference;

DATA FOUR;

LOWORD=1+INT(&SIZE\*(&SIZE+1)/4 + PROBIT(&ALPHA/2)

\*SORT(&SIZE\*(&SIZE+1)\*(2\*&SIZE+1)/24));

UPPORD= CEIL(&SIZE\*(&SIZE+1)/4 + PROBIT(1-&ALPHA/2)

\*SQRT(&SIZE\*(&SIZE+1)\*(2\*&SIZE+1)/24));

RUN;

DATA FIVE; SET THREE END=LAST;

IF N = 1 THEN SET FOUR;

RETAIN LOWER UPPER;

IF N =LOWORD THEN LOWER=STAT;

IF N = UPPORD THEN UPPER=STAT;

IF LAST THEN OUTPUT;

KEEP LOWER UPPER;

RUN;



Last Revision Date: 13 Mar 2018

| (1 age | e 46 of 48) |
|--------|-------------|

| DATA HL_EST; MERGE EST FIVE; RUN; %MEND HL_PAIRED; Linear mixed effects model for CLASS SUBJECT PERIOD TRT SEQUENCE; |
|---|
| %MEND HL_PAIRED; Linear mixed PROC MIXED PLOTS (ALL) METHOD=REML; effects model for CLASS SUBJECT PERIOD TRT SEQUENCE; |
| Linear mixed PROC MIXED PLOTS (ALL) METHOD=REML; effects model for CLASS SUBJECT PERIOD TRT SEQUENCE; |
| effects model for CLASS SUBJECT PERIOD TRT SEQUENCE; |
| , |
| 1 4' C MODEL W DAGE DEDIOD TRIT GEOLIENGE |
| duration of MODEL Y = BASE PERIOD TRT SEQUENCE |
| response / DDFM=KENWARDROGER SOLUTION VCIRY |
| parameters when OUTP=OUT; |
| a parametric RANDOM SUBJECT; |
| analysis is LSMEANS TRT / PDIFF CL ALPHA=0.05; |
| appropriate ODS OUTPUT LSMEANS=MEANS CORR COV; |
| (Hodges- ODS OUTPUT DIFFS=DIFF; |
| Lehmann code RUN; |
| below when a |
| non-parametric Where BASE is the baseline value of the endpoint and TRT is the |
| analysis is treatment. |
| appropriate) |
| Descriptive PROC FREQ; |
| statistics for TABLES Y / OUT=FREQCOUNT SPARSE; |
| Percentage of BY TRT; |
| subjects RUN; |
| achieving 12% |
| improvement in Where TRT is the treatment. |
| FEV <sub>1</sub> from |
| baseline within 30 minutes of |
| dose and |
| Percentage of |
| subjects |
| achieving 15% |
| improvement in |
| FEV <sub>1</sub> from |
| baseline within 30 minutes of |
| dose |
| Linear Mixed PROC MIXED PLOTS (ALL) METHOD=REML; Maddal analysis CLASS SUBJECT REPLOD TRT SEQUENCE: |
| Model analysis CLASS SUBJECT PERIOD TRT SEQUENCE;<br>for a continuous MODEL Y = BASE PERIOD TRT SEQUENCE |
| efficacy SUBGROUP TRT*SUBGROUP |
| endpoint, change / DDFM=KENWARDROGER VCIRY SOLUTION OUTP=OUT |





Last Revision Date: 13 Mar 2018


| from baseline in | RANDOM SUBJECT; |
|---|---|
| AUC <sub>0-6</sub> , change | LSMEANS TRT SUBGROUP / PDIFF CL ALPHA=0.05 |
| from baseline in | CORR COV; |
| AUC <sub>0-4</sub> , or Peak | ODS OUTPUT LSMEANS=MEANS; |
| Change from | ODS OUTPUT DIFFS=DIFF; |
| Baseline in | RUN; |
| FEV <sub>1</sub> . Use this | |
| code for the | Where BASE is the baseline value of the endpoint, TRT is the |
| subgroup | treatment, and SUBGROUP is 1=ICS Use at Screening and 2=No ICS |
| analysis of the | Use at Screening |
| primary and | |
| secondary | THE PLOTS (ALL) OPTION FOR PROC MIXED WILL BE USED |
| endpoints. | TO GET PLOTS TO PERFORM MODEL DIAGNOSTICS (for |
| | normality and heterogeneity of variance). Scaled residuals will be used. |



Last Revision Date: 13 Mar 2018 

### APPENDIX 4 MOCKUP TABLES, LISTINGS, AND GRAPHS (TLGS)

Mockup tables, listings, and graphs are presented in a separate document.

## APPENDIX 4 SPECIFICATION OF END-OF-TEXT STANDARD OUTPUT TABLES, LISTINGS, AND FIGURES (TLFs)

**Protocol Title:** A Randomized, Double-blind, Single dose, Placebo-controlled, 5-Period, 5-Treatment, Crossover, Multi-center, Dose-ranging Study to Compare PT007 to Placebo MDI and Open-Label Proventil® HFA in Adult and Adolescent Subjects With Mild to Moderate Asthma

### PT007001

| Trial Sponsor: | AstraZeneca AB |
|---|---|
| Study Number: | D6930C00001 (PT007001) |
| Study Phase: | П |
| <b>Product Name:</b> | Albuterol Sulfate Pressurized Inhalation Suspension (AS MDI); PT007 |
| PIND Number: | 136213 |
| Indication: | Asthma |
| Dosage Form/Strength | <ul> <li>AS MDI as</li> <li>2 actuations of 45 μg per actuation (90 μg)</li> <li>2 actuations of 90 μg per actuation (180 μg)</li> </ul> |

**Date of Issue:** 13 Mar 2018

Version 1.0

### **General Instructions for End-of-Text TFLs**

Following are the specifications for end of text standard Tables, listings, and Figures (TFLs).

### Header

The following header should appear at the very top of each page of a Table, a listing, or a Figure (TLF):

Protocol PT007001

Albuterol Sulfate Pressurized Inhalation Suspension

### Footer

The following footer should appear at the bottom of each page of a TLF generated in SAS:

Report generated by program:/sasdir/PGNAME.sas Version YYYY-mm-dd hh:mm (Page n of N)

where: PGNAME = SAS program name. Version will be replaced by "Draft" or "Final". Page number will be right-justified.

### <u>Title</u>

At least two (2) lines should be reserved for the whole title. The first line of the title is for the TLF number (i.e., title index #) and the actual title (title); a longer title may continue onto subsequent lines. The analysis analysis set descriptor (Analysis Set) will be specified on the line following the title line(s). All titles should be centered, as shown in the following example:

Table 1.5.3 Demographics Analysis Set: Safety Analysis Set

### Footnotes

- In general, a footnote serves as a brief explanation/clarification/definition/concept of a flag symbol or a character, an abbreviation, a terminology, etc., that appears in or related directly to the displayed content of a TLF. Detailed/technical elaboration of, for example, a mathematical/statistical formula, a statistical term/test, or an algorithm for deriving a parameter value, should be addressed in the text of the statistical analysis plan (SAP).
- All footnotes should follow immediately after a horizontal solid line. There should be one and only one space between the
  last footnote and the footer.
- Each line of a complete footnote should end with a period. When a footnote needs more than 1 line, one (1) period is needed.
- Large data listings will have footnotes on the first page only.

Row Labels/Column Labels: The mockups will reflect the preferred style of capitalization.

### Page Layout

- All output should be in landscape orientation. A margin of 1.5, 1, 1, and 1 inch should be on the top, right, left, and bottom, respectively.
- All efforts should be made to present all Treatment groups in one page.
- When 3 or more Treatment groups are designed for a study and if it is not possible to fit all of them in one page, the 4<sup>th</sup> and 5<sup>th</sup> treatment groups should be displayed on the 2nd page, etc. The Study Biostatistician will pre-determine the order for the display of the treatment groups.

### Page Format

- There should be a solid line at the top of the Tables and listings just below the title.
- There should be a solid line just below the column headings that runs completely across the width of the Tables and listings.
- There should be a solid line at the bottom of the Tables and listings just above the footnote(s) on every page.

### **Font**

- The default font to be used in the actual study Tables/listings should be Courier New 8 point which is approximately equivalent to the accepTable font size of Times New Roman 9-10 in accordance with the FDA's guidance on Electronic Common Technical Document Specification.
- The use of Courier New 7 point is optional for some Tables/listings and will be determined at the study level by the Study Biostatistician and Study Programmer. However, it is recommended that this option be used primarily for data listings.

### Descriptive Statistics

By default, descriptive statistics in this template covers: n, Mean, Median, Standard Deviation (SD), Minimum (Min), and Maximum (Max). Unless otherwise specified in the actual Table shells, the mean, standard deviation, standard error of the mean, and median should be displayed to one more decimal place than the original data. The standard error of the mean will be displayed with at least 2 significant digits for efficacy Tables.

### Rounding for Percentage

Unless specified in the actual Table shells for a study, all percentages will be rounded to 1 decimal place in all TLFs. Percentage signs will not be included in the body of the Table (i.e., 99.9 will be displayed, not 99.9%), but may be included in row or column headings.

Unless specified in the actual Table shells for a study, p-values will be presented with 4 decimal places.

### Alignment of Decimals

• It is recommended that all the decimal places be aligned in summary Tables, as shown in the following example:

| | Decimal Align |
|------------------|---------------|
| n | xxx |
| Mean | XX.XX |
| SD | XX.XX |
| Median | XX.XX |
| Minimum, Maximum | XX.X. XX.X |

• When numbers with decimal points are included in brackets (e.g., percentages), have the brackets aligned to the right and then padded to allow for all possible percentages and then the left brackets will also be aligned. For example:

| | Brackets Align | |
|--------|----------------|--------|
| (99.9) | | (xx.x) |
| (99) | | ( x x) |

- It is recommended that all column entries in a summary Tables and listings are aligned to the center.
- Columns for text fields are all left justified. Columns with whole numbers are all right justified.
- For graphs, the lines are distinguishable and that the symbols for each line are appropriate. Legend is consistent across output for Treatment names and abbreviations.

### Use of N Versus n

- N = total number of subjects in the defined analysis set.
- n = total number of subjects in the specific category.
- If N is specified in the column heading then any reference to the number of subjects in the body should be small n, as shown in the following example:


| | Treatment<br>Group A | Treatment<br>Group B | Total |
|---|---|---|---|
| Demographic Parameter | (N=XXX) | (N=XXX) | (N=XXX) |
| Age (years) | | | |
| n | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X |
| SD | X.X | X.X | X.X |
| Median | XX.X | XX.X | XX.X |
| Minimum, Maximum | XX, XX | XX, XX | XX, XX |

### A Note for Subject Data Listings

- Observed Dates/AE Severity/Relationship to investigational product are used in subject data listings.
- Observed values or raw assessment scores are used in data listings along with their derived values used in analyses, e.g., raw
  assessment scores and derived total scores.

### **Table of Contents**

| Table 1.1.1 | Subject Disposition | |
|---|---|---|
| | Analysis Set: All Screened Subjects | |
| Table 1.1.2 | Reasons for Subjects Not Randomized | |
| Table 1.1.3 | Exclusions From ITT, mITT, and Safety Analysis Sets | |
| Table 1.2.1 | Reason for Premature Treatment Discontinuation | |
| Table 1.2.2 | Reason for Premature Treatment Discontinuation | • |
| Table 1.2.3 | Reason for Premature Treatment Discontinuation | |
| Table 1.3 | Analysis Sets by Treatment | |
| Table 1.4 | Reason for Exclusion From the mITT Analysis Set | |
| Table 1.5.1 | Demographics and Baseline Characteristics | |
| Table 1.5.2 | Demographics and Baseline Characteristics | |
| Table 1.5.3 | Demographics and Baseline Characteristics | |
| Table 1.5.4 | Demographics and Baseline Characteristics | |
| Table 1.6.1 | Duration of Asthma | |
| Table 1.6.2 | Duration of Asthma | |
| Table 1.7.1 | Screening Pre- and Post-Bronchodilator and Baseline Spirometry Parameters<br>Analysis Set: mITT Analysis Set | |
| Table 1.7.2 | Screening Pre- and Post-Bronchodilator and Baseline Spirometry Parameters<br>Analysis Set: ITT Analysis Set | |
| Table 1.8.1 | Reversibility to Ventolin HFA at Screening | |
| Table 1.8.2 | Reversibility to Ventolin HFA at Screening | |
| Table 1.9 | Medical/Surgical History<br>Analysis Set: Safety Analysis Set | • |

| Table 1.10.1 | Prior Medications – Asthma-Related | 26 |
|---|---|---|
| Table 1.10.2 | Prior Medications-Other than Asthma-Related | 26 |
| Table 1.11.1 | Concomitant Medications During Treatment Period – Asthma-Related<br>Analysis Set: Safety Analysis Set | 27 |
| Table 1.11.1 | Concomitant Medications During Washout Period – Asthma-Related | 27 |
| Table 1.11.2 | a Concomitant MedicationsDuring Treatment Period-Non-Asthma Related<br>Analysis Set: Safety Analysis Set | 27 |
| Table 1.11.2 | Concomitant Medications During Washout Period-Non-Asthma Related<br>Analysis Set: Safety Analysis Set | 27 |
| 2. EFFICACY | SUMMARY TABLES AND FIGURES | 28 |
| PRIMARY EFFIC | CACY ENDPOINT | 28 |
| Table 2.1.1 | Change from Baseline in $FEV_1$ $AUC_{0-6}$ (L) Overall and by ICS Use Subgroups Analysis Set: mITT Analysis Set | 29 |
| Table 2.1.2 | Change from Baseline in FEV $_1$ AUC $_{0-6}$ (L) Overall and by ICS Use Subgroups Analysis Set: ITT Analysis Set | 31 |
| SECONDARY EF | FFICACY ENDPOINTS | 31 |
| Table 2.2.1 | Change from Baseline in $FEV_1$ $AUC_{0-4}$ $(L)$ | 31 |
| Table 2.2.2 | Peak Change from Baseline in $FEV_1$ (L) | 31 |
| OTHER EFFICAC | CY ENDPOINTS | 32 |
| Table 2.3.1 | Change from Baseline in $FEV_1$ (L) by Timepoint | 32 |
| Figure 2.3.1. | Change from Baseline in FEV $_1$ (L) $\pm$ SE Over Time | 34 |
| Figure 2.3.1. | Treatment Differences From Placebo*: Change from Baseline in FEV <sub>1</sub> (L) ± 95% CI Over Time | 35 |
| Table 2.3.2 | Time to Peak FEV <sub>1</sub> | 36 |
| Table 2.3.3 | Percentage of Subjects Achieving a 12% or 15% Improvement in FEV <sub>1</sub> from Baseline Within 30 Minutes Post-Dose | 37 |
| Table 2.3.4 | Time to Onset of 12% Improvement in $FEV_1$ | 38 |
| Table 2.3.5 | Time to Onset of 15% Improvement in ${\rm FEV}_1$ | 38 |
| Table 2.3.6 | Duration of 12% Improvement in FEV <sub>1</sub> | 39 |

| Table 2.3 | Duration of 12% Improvement in FEV <sub>1</sub> : Subjects who Have Assessments at the 180- and 300-Minute Post-Dose Timepoints | 40 |
|---|---|---|
| Table 2.3 | Duration of 15% Improvement in FEV <sub>1</sub> | 41 |
| Table 2.3 | Duration of 15% Improvement in FEV <sub>1</sub> : Subjects who Have Assessments at the 180- and 300-Minute Post-Dose Timepoints | 41 |
| 3. SAFETY | | 42 |
| ADVERSE EV | VTS | 42 |
| Table 3.1 | Overall Summary of Treatment-Emergent Adverse Events | 42 |
| Table 3.1 | Overall Summary of Treatment-Emergent Adverse Events Including Adverse Events on a Treatment Day or During the Washout or Follow-up Periods | 43 |
| Table 3.2 | Treatment-Emergent Adverse Events by MedDRA Primary System Organ Class and Preferred Term | 44 |
| Table 3.2 | Treatment-Emergent Adverse Events by MedDRA Primary System Organ Class and Preferred Term Including Events Occurring During the Washout or Follow-up Periods: Sensitivity Analysis | 44 |
| Table 3.2 | Treatment-Emergent Adverse Events Occurring in >=2% of Subjects in a Treatment by Descending Frequency Analysis Set: Safety Analysis Set | 44 |
| Table 3.2 | Non-serious Treatment-Emergent Adverse Events Occurring in >=5% of Subjects in a Treatment by MedDRA Primary System Organ Class and Preferred Term Analysis Set: Safety Analysis Set | 45 |
| Table 3.3 | Treatment-Related Treatment-Emergent Adverse Events by MedDRA Primary System Organ Class and Preferred Term | 46 |
| Table 3.4 | Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by MedDRA Primary System Organ Class and Preferred Term | 46 |
| Table 3.5 | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment | 47 |
| Table 3.6 | Serious Adverse Events by MedDRA Primary System Organ Class and Preferred Term | 48 |
| Table 3.6 | Serious Adverse Events by MedDRA Primary System Organ Class and Preferred Term Including Events Occurring During the Washout and Follow-up Period: Sensitivity Analysis | 48 |

| | Table 3.7.1 | Listing of Serious Adverse Events (SAEs) | 49 |
|---|---|---|---|
| | Table 3.7.2 | Listing of SAE-Specific Report Information | 50 |
| | Table 3.8 | Treatment Related Serious Adverse Events by MedDRA Primary System Organ Class and Preferred Term Analysis Set: Safety Analysis Set | 52 |
| | Table 3.9.1 | TEAEs by Primary System Organ Class, Preferred Term, and Highest Severity – Placebo | 53 |
| | Table 3.9.2 | TEAEs by Primary System Organ Class, Preferred Term, and Highest Severity – AS MDI 90 µg<br>Analysis Set: Safety Analysis Set | 53 |
| | Table 3.9.3 | TEAEs by Primary System Organ Class, Preferred Term, and Highest Severity – AS MDI 180 μg<br>Analysis Set: Safety Analysis Set | 53 |
| | Table 3.9.4 | TEAEs by Primary System Organ Class, Preferred Term, and Highest Severity – Proventil 90 µg Analysis Set: Safety Analysis Set | 53 |
| | Table 3.9.5 | TEAEs by Primary System Organ Class, Preferred Term, and Highest Severity – Proventil 180 μg | 53 |
| | Table 3.10 | Listing of Deaths Analysis Set: All Subjects Screened | 54 |
| VIT | AL SIGNS | | 55 |
| | Table 3.11.1 | Vital Sign Parameters<br>Analysis Set: Safety Analysis Set | |
| 4. | SUBJECT DATA | LISTINGS | 56 |
| 4.1 | SUBJECT DISCO | ONTINUATIONS/COMPLETIONS | 56 |
| | Listing 1.1 | Study Centers | 56 |
| | Listing 1.2 | Subject Disposition and Demographic Data<br>Analysis Set: All Subjects Screened | 57 |
| | Listing 1.3 | Randomized Treatment, Actual Treatment, and Duration of Treatment | 59 |
| | Listing 1.4 | Reasons Subjects Were Not Randomized | 61 |
| 4.2 | PROTOCOL DE | VIATIONS | 62 |
| | Listing 2 | Violation of Inclusion/Exclusion Criteria | 62 |
| 4.3 | SCREENING LU | NG FUNCTION AND REVERSIBILITY | 63 |
| | Listing 3 | Screening Lung Function and Ventolin HFA Reversibility | 63 |

| 4.4 | BASELINE CHA | ARACTERISTICS | 64 |
|---|---|---|---|
| | Listing 4.1 | Asthma Diagnosis | 64 |
| | Listing 4.2 | Medical and Surgical HistoryAnalysis Set: All Subjects Randomized | 65 |
| | Listing 4.3 | Screening Reproductive Status and Pregnancy Test Results | 66 |
| | Listing 4.4 | Prior, Concomitant, and Post-Treatment Asthma Medications | 67 |
| | Listing 4.5 | Prior, Concomitant, and Post-Treatment Non-Asthma-Related Medications<br>Analysis Set: All Subjects Randomized | 67 |
| | Listing 4.6 | Suspect Drug Assessment for SAEs<br>Analysis Set: All Subjects Randomized | 68 |
| 4.5 | DOSING | | 69 |
| | Listing 5.1.1 | Study Drug Administration | 69 |
| | Listing 5.1.2 | Ventolin HFA and Pulmicort Flexhaler Dispensing | 70 |
| | Listing 5.2 | Exposure to Study Treatment | 71 |
| 4.6 | INDIVIDUAL E | FFICACY DATA | 72 |
| 4.6.1 | Efficacy | | 72 |
| | Listing 6.1 | Subjects Who Failed Restrictions Prior to Spirometry Assessment | |
| | Listing 6.2 | Failure of Stability Criteria | 73 |
| | Listing 6.3 | Reason for Missed Visit | 74 |
| | Listing 6.4 | Spirometry Measurements | 75 |
| | Listing 6.5 | Spirometry Derived Endpoints | 76 |
| 4.7 | ADVERSE EVE | NT LISTINGS | 78 |
| | Listing 7.1 | Adverse Events by Primary System Organ Class, Preferred Term, Treatment, Country, Center, Subject ID, and Onset Day | 78 |
| | Listing 7.2<br>Listing 7.3 | Glossary of Adverse Event Preferred Terms vs. Investigator's Verbatim | 80<br>81 |
| 4.8 | LABORATORY | VALUES | 82 |
| | Listing 8.1 | Laboratory Test Results (Hematology Panel) | |

### 

| | Listing 8.2 | Laboratory Test Results (Chemistry Panel and Kidney Function) | 82 |
|---|---|---|---|
| | Listing 8.3 | Laboratory Test Comments | 83 |
| 4.9 | OTHER CLINICA | AL OBSERVATIONS AND MEASUREMENTS | 84 |
| | Listing 9.1 | Vital Signs, Weight, and Height<br>Analysis Set: All Subjects Randomized | 84 |
| | Listing 9.2 | 12-Lead Electrocardiogram (ECG) | 86 |
| | Listing 9.3 | Comments | 87 |

# 1. Subject Disposition, Demographic, Baseline, and Other Summary Tables

Table 1.1.1 Subject Disposition Analysis Set: All Screened Subjects

| | All Subjects |
|---|---|
| | (N=XXX) |
| | n (%) |
| Not Treated | xx (xx.x) |
| Treated | xx (xx.x) |
| Treated with AS MDI 90 µg | xx (xx.x) |
| Treated with AS MDI 180 µg | xx (xx.x) |
| Treated with Proventil 90 µg | XX (XX.X) |
| Treated with Proventil 180 µg | XX (XX.X) |
| Treated with Placebo | xx (xx.x) |
| Length of Subject Participation in the Study | |
| 5 Treatment Periods | xx (xx.x) |
| 4 Treatment Periods | xx (xx.x) |
| 3 Treatment Periods | xx (xx.x) |
| 2 Treatment Periods | XX (XX.X) |
| 1 Treatment Period only | XX (XX.X) |
| O Treatment Periods | xx (xx.x) |
| Completed Study | xx (xx,x) |
| Premature Discontinuation | xx (xx.x) |
| ITT Analysis Set [a] | xx (xx.x) |
| MITT Analysis Set [b] | xx (xx.x) |
| Safety Analysis Set [c] | XX (XX.X) |
| Not Randomized Analysis Set [d] | XX (XX.X) |
| [a] The Intent-To-Treat (ITT) Analysis Set was defined as all subjects who were randomized to treat | d to treatment and received at least 1 dose |
| OH HOO DHIDIN HOODHBOOKH CIPOTON ON ON THE SOOK SOOK ON THE SOOK HOO | |

of the study treatment. Subjects were analyzed in each period according to the treatment they were assigned to per the randomization scheme (Note that a subject who used a study treatment but took less than 1 full dose of treatment qualified for this analysis set). treatment efficacy data from at least 2 Treatment Periods. Data judged to be impacted by major protocol deviations was determined prior to unblinding and excluded per the statistical protocol deviation plan. Statistical tabulations and analyses were by randomized [b] The mITT Analysis Set was defined as a subset of the ITT analysis set including subjects who received treatment and had posttreatment, but data obtained after subjects received an incorrect treatment were excluded from the affected periods.

[d] The Not Randomized analysis set was defined as subjects who did not receive a randomization number and therefore did not receive a [c] The Safety Analysis Set was defined as all subjects who were randomized to treatment and received at least 1 dose of the study treatment. Subjects were analyzed according to treatment received rather than per the randomization scheme.

dose of study treatment (eg, subjects who were screen failures or stopped participation before being randomized).


Reasons for Subjects Not Randomized Analysis Set: All Subjects Not Randomized Table 1.1.2

| | All Subjects Not Randomized (N=xxx) |
|---|---|
| Reason Not Randomized | n (%) |
| Any Inclusion/Exclusion Criterion | xxx (xx.x) |
| Exclusion Criterion #x: xxxx xxxx xx xxxxx xxxxx | xxx (xx.x) |
| Exclusion Criterion #x: xxx xxxxxxxxxx xx xxxxx x | xxx (xx.x) |
| Inclusion Criterion #x: xx x xxx xxxx xxxx xxxxxxxxxx | xxx (xx.x) |
| Inclusion Criterion #x: xxxx xxxx xx xxxxx xxxxx xxxx | xxx (xx.x) |
| FANY Fallure of Kandolmzation Criteria | (xxx) (xx.x) |
| Cfiteria #X; XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX (XX.X) |
| Note: Reasons of Other are listed by subject in Listing 1 X | |

Notes to Programmer: Order by frequency within each category. Display all protocol-specified criteria shown on the End of Treatment/ CRF that have counts> 0.. Report generated by program: PT007001/sasdir/programs/statout/t010102.sas Version YYYY-MM-DD xx:xx From Section 3.3.1 of the Protocol, the Randomization Criteria are:

(Page n of N)

- 1. Subjects of childbearing potential must have a negative urine pregnancy test
- 2. Received no asthma medication other than Sponsor-provided Pulmicort Flexhaler
  - 180 µg or 360 µg BID as assigned and/or Sponsor-provided Ventolin from Visit I
- to Visit 2, except for allowable allergy medications defined in Table 8 of the Protocol.
  - 3. The last dose of Pulmicort Flexhaler (if applicable) was the previous night (ie,
    - morning dose of Pulmicort Flexhaler was not administered), and the last dose of
      - Sponsor-provided Ventolin was no later than 6 hours before the study visit (if Ventolin is needed in the morning, the visit must be rescheduled)
        - 4. Pre-bronchodilator  $FEV1 \ge 40\%$  percent predicted normal value
- 5. Has not used >8 actuations per day (ie, 4 doses of 2 actuations per day) of Sponsorprovided
  - Ventolin for rescue on more than any 3 days during the previous 7 days
- 6. No upper respiratory infection, lower respiratory infection, or asthma exacerbation during the Screening Period
  - 7. Demonstrate acceptable MDI administration technique
    - 8. Able to comply with all study procedures


Exclusions From ITT, mITT, and Safety Analysis Sets

Analysis Set: All Subjects Randomized

Table 1.1.3

| Subject | Treatment<br>Sequence | Analysis<br>Set<br>Excluded | Period<br>Excluded | Timepoints<br>Excluded | Variable(s)<br>Excluded | Reason for Exclusion |
|---|---|---|---|---|---|---|
| Study Ce | Study Center # / (Investigator): | estigator): | (**********) / ### | (xxxx) | | |
| ×××× | -/-/-/- | III | A11 | A11 | A11 | Subject did not receive treatment in at least 1 |
| | | MITT | A11 | A11 | A11 | Subject did not have post-treatment efficacy data from at least 2 Treatment Periods |
| | | Safety | A11 | A11 | A11 | and receive at least one dose of the study treatment in the study |
| | | TIIW | Period 1 | 300, 360<br>Minutes | All | Subject did not have post-treatment efficacy data from at least 2 Treatment Periods. |
| ×××× | A/B/E/C/D | Safety | All | All | All | Subject did not receive treatment in at least 1 treatment period. |
| ×××× | B/C/-/-/- | TTI | A11 | All | A11 | Subject did not receive treatment in at least 1 |
| | | TII | A11 | A11 | A11 | ureaument periou.<br>Subject did not have post-treatment efficacy data from |
| | | Safety | All | All | All | Did not receive at least one dose of the study treatment in the study. |
| ×××× | A/E/-/- | TII | A11 | All | All | Subject took incorrect study medication. |
| ××××× | B/A/C/E/- | TIIm | Period 4 | Al 1 | A11 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. Subjects may be included in a analysis set as a whole, but have period or timepoint data excluded.

Report generated by program: PT007001/sasdir/programs/statout/t010103.sas Version YYYY-MM-DD xx:xx

(Page n of N)

# Notes to Programmer:

Sort by Study Center, Investigator, and Subject within Study Center. List records per subject, analysis set excluded, period excluded, and timepoint excluded.

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


Reason for Premature Treatment Discontinuation Analysis Set: ITT Analysis Set Table 1.2.1

| | Placebo<br>(N=xxx) | AS MDI<br>90 µg<br>(N=xxx) | AS MDI<br>180 µg<br>(N=xxx) | Proventil<br>90 µg<br>(N=xxx) | Proventil<br>180 µg<br>(N=xxx) |
|---|---|---|---|---|---|
| | U (%) | n (%) | n (%) | n (%) | n (%) |
| Premature Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for Premature Treatment Discontinuation | | | | | |
| Administrative Reasons | xx (xx.x) | xx (xx.x) | (xx.x) | (xx.x) | xx (xx.x) |
| Adverse Event | xx (xx.x) | xx (xx.x) | (xx.x) | (xx.x) | xx (xx.x) |
| Lack of Efficacy | xx (xx.x) | xx (xx.x) | (xx.x) | (xx.x) | xx (xx.x) |
| Subject Discretion | (x.xx) xx | (x.xx) xx | (x.xx) xx | (x.xx) xx | (xxxx) xx |
| Withdrawal of Consent | | | | | |
| Asthma | xx $(xx.x)$ | (xx.x) | (xx.xx) | (x.x.) | xx (xx.x) |
| Other | (x.x.) | (xx.x) | (xx.xx) xx | (x.x) | xx (xx.x) |
| Investigator or Designee Considers it to be in the Best Interest of<br>the Subject | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject Lost-to-Follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Major Protocol Deviation | xx (xx.x) | xx (xx.x) | (x.xx) xx | (x.xx) xx | xx (xx.x) |
| Protocol-Specified Discontinuation Criteria | xx (xx.x) | xx (xx.x) | (xx.x) | (xxxx) xx | xx (xx.x) |
| FEV1 Stability Criteria Sec 5.1.4 | xx (xx.x) | xx (xx.x) | (xx.x) | (xxxx) xx | xx (xx.x) |
| Requirement of any Prohibited Medications Listed in Sec 7.7.3 | xx (xx.x) | xx (xx.x) | (xx.x) | (x.xx) xx | xx (xx.x) |
| Positive Pregnancy Test | (x.xx) xx | xx (xx.x) | (xx.x) | (xx.xx) | xx (xx.x) |
| Asthma Worsening Requiring Change in Asthma Treatment Sec 3.9 | xx (xx.x) | xx (xx.x) | (xx.x) | (xxxx) xx | xx (xx.x) |
| The Subject's Treatment Code Prematurely Broken by Investigator | xx $(xx.x)$ | (xx.x) | (xx.xx) | (x.x.) | xx (xx.x) |
| Other | (xx,x) | (xx,x) | (xx,x) | (xx,x) | (xx,x) |

Note: Reasons of Other are listed by subject in Listing 1.2.

Report generated by program: PT007001/sasdir/programs/statout/t010201.sas Version YYYY-MM-DD xx:xx

(Page n of N)

Notes to Programmer:Sort by descending frequency of major reason category using AS MDI column. Within a major reason category, sort by descending frequency of subcategory using AS MDI column.

Reason for Premature Treatment Discontinuation Table 1.2.2

Analysis Set: mITT Analysis Set

Footnotes: Subjects were included in summaries for a treatment if they received at least one dose of the treatment.

Table 1.2.3 Reason for Premature Treatment Discontinuation Analysis Set: Safety Analysis Set

Footnotes: Subjects were included in summaries for a treatment if they received at least one dose of the treatment.


Table 1.3 Analysis Sets by Treatment Analysis Set: All Subjects Randomized

| | Placebo<br>(N=xxx) | AS MDI<br>90 µg<br>(N=xxx) | AS MDI<br>180 µg<br>(N=xxx) | Proventil 90 Proventil 180 µg µg (N=xxx) (N=xxx) | Proventil 180<br>µg<br>(N=xxx) |
|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) |
| Intent-to-treat Analysis Set [a] | xx (xx.x) | (xx.x) | xx (xx.x) | (x.xx) | (x.xx) |
| mITT Analysis Set [b] | (x.xx) xx | (xx.x) | xx (xx.x) | (x.x) xx | (x.xx) xx |
| Safety Analysis Set [c] | xx (xx.x) | (x.xx) xx | (x.xx) xx | (x.x) xx | (x.x) xx |

treatment efficacy data from at least 2 Treatment Periods. Data judged to be impacted by major protocol deviations were determined Subjects were analyzed in each period according to the treatment they were assigned to per the randomization [b] The mITT Analysis Set was defined as a subset of the ITT analysis set including subjects who received treatment and had post-[a] The Intent-To-Treat (ITT) Analysis Set was defined as all subjects who were randomized to treatment and received at least 1 dose prior to unblinding and excluded per the statistical protocol deviation plan. Statistical tabulations and analyses were by randomized scheme (Note that a subject who used a study treatment but took less than 1 full dose of treatment qualified for this analysis set). [c] The Safety Analysis Set was defined as all subjects who were randomized to treatment and received at least 1 dose of the study treatment, but data obtained after subjects received an incorrect treatment was excluded from the affected periods. n=1 n = number of subjects in the category, N=# of subjects who were randomized to the treatment,  $\$=100 \times n/N$ . of the study treatment.

Report generated by program: PT007001/sasdir/programs/statout/t0103.sas Version YYYY-MM-DD xx:xx

treatment. Subjects were analyzed according to treatment received rather than per the randomization scheme.

 $\widehat{z}$ 

(Page n of


Table 1.4 Reason for Exclusion From the mITT Analysis Set
Analysis Set: ITT Analysis Set

| | | 7 | AS MDI | AS MDI | Pr | Proventil | Proventil |
|---|---|---|---|---|---|---|---|
| | Placebo | | 90 pg | 180 µg | | 90 pd | 180 µg |
| | (N=xxx) | <u> </u> | (N=xxx) | (N=XXX) | ٦ | N=xxx) | (N=xxx) |
| Reason for | n (%) | | (%) u | n (%) | | n (%) | n (%) |
| Exclusion of a Subject from mITT Analysis Set | (x.xx) | | (x.xx) xx | (x.xx) | | (x.xx) xx | (xx.x) |
| <reason 1=""></reason> | (x.xx) xx | | xx (xx.x) | (x.xx) xx | | xx (xx.x) | xx (xx.x) |
| <reason 2=""></reason> | (x.xx) xx | | xx (xx.x) | (x.xx) xx | | (x.xx) xx | xx (xx.x) |
| • | | | | | | | |
| Exclusion of a Treatment Period from mITT Analysis Set | (x.xx) | | xx (xx.x) | (x.xx) | | (xx.x) | xx (xx.x) |
| <reason 1=""></reason> | (xx.xx) | | xx (xx.x) | xx (xx.x) | XX (X | (xx.xx) | xx (xx.x) |
| <reason 2=""></reason> | (x.xx) xx | | xx (xx.x) | (x.xx) xx | | xx (xx.x) | xx (xx.x) |
| = | | | | | | | |

Subjects may have multiple reasons for exclusion; therefore, counts for individual reasons may not add up to the total number of subjects excluded from the analysis set.

Report generated by program: PT007001/sasdir/programs/statout/t0104.sas Version YYYY-MM-DD xx:xx N)

Note to the Programmer: Subjects are to be included in summaries and N= in the column header for a treatment if they attended a visit designated for a treatment in their treatment sequence. 

Demographics and Baseline Characteristics Analysis Set: mITT Analysis Set

Table 1.5.1

| Daramatar | All Subjects |
|---|---|
| - מדמוויי כי כי | ( ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, |
| Age (Years)[a] | |
| u. | XXX |
| Mean | XX.X |
| SD | XX.X |
| Median | XX.X |
| Minimum | XX |
| Maximum | ×× |
| Age Group, n (%) | |
| Age 12 to < 18 years | xxx (xx.x) |
| Age 18 to 65 years | XXX (XX.X) |
| Missing | x (xx.x) |
| Gender, n (%) | |
| Male | xxx (xx.x) |
| Female | XXX (XX.X) |
| Missing | x (xx.x) |
| Race, n (%) | |
| Black or African | (X, XX) XX |
| American | |
| White | XXX (XX.X) |
| Native Hawaiian or Other Pacific Islander | XX (XX.X) |
| American Indian or Alaska Native | XX (XX.X) |
| Asian | |
| Other | xx (xx.x) |
| Missing | xx (xx.x) |
| Ethnicity, n (%) | |
| Hispanic | XXX (XX.X) |
| Not Hispanic or Latino | XXX (XX.X) |
| Unknown | XXX (XX.X) |
| Not Reported | xx (xx.x) |
| Smoking Status, n (%) [b] | |
| Former Smoker | XXX (XX.X) |
| Non Smoker | xxx (xx.x) |
| Missing | xxx (xx.x) |

Number of Years Smoked


Albuterol Sulfate Pressurized Inhalation Suspension Protocol D6930C00001 (PT007001)

| | איסיליוי רוע |
|---------------------------------------------|--------------|
| Parameter | |
| ជ | XXX |
| Mean | XX.X |
| SD | XX.X |
| Median | XX.X |
| Minimum | XX.X |
| Maximum | x.xx |
| Average Number of Cigarettes Smoked Per Day | |
| | XXX |
| Mean | XX.X |
| SD | XX.X |
| Median | XX.X |
| Minimum | XX.X |
| Maximum | XX.XX |
| Number of Pack Years Smoked [c] | |
| u | XXX |
| Mean | XX.X |
| SD | XX.X |
| Median | XX.X |
| Minimum | XX.X |
| Maximum | xx.x |
| Prior Asthma Medication | |
| | ×·×× |
| | X.XX |
| ICS/LABA, n (%) | XX.X |
| Weight (kg) | |
| u | XXX |
| Mean | × · ×× |
| SD | XX.XX |
| Median | XX.X |
| Minimum | XX.X |
| Maximum | xx.x |
| Height (cm) | |
| n | XXX |
| Mean | XXX.X |
| SD | XXX.X |
| Median | XXX.X |
| Minimum | XXX.X |
| Maximum | xxx.x |
| BMI $(kg/m^2)$ | |
| u u | XXX |


| All Subjects | (N=XX) | XX.X | XX.X | XX.X | XX.X | xxx |
|--------------|-----------|------|------|--------|---------|---------|
| | Parameter | Mean | SD | Median | Minimum | Maximum |

- Age is age at Visit 1. The remaining characteristics were based on data from Screening visits prior to the start of the study. []
- Former Smoker was defined as those who have stopped smoking for at least 6 months prior to first [2]
  - Screening Visit and have no more than 10 pack years history of smoking. Number of pack years smoked = (number of cigarettes per day / 20) x number of years smoked. []

Report generated by program: PT007001/sasdir/programs/statout/t010501.sas Version YYYY-MM-DD xx:xx (Page n of N)

Notes to Programmer:

Sort race by decreasing frequecing. The race/ethnicities of Native Hawaiian or Other Pacific Islander OR American Indian or Alaska Native can be removed from this Table if Repeat titles, column headers, and footnotes on each page. Keep the summary for a parameter in the same page when breaking the Table into multiple pages. they do not exist in the database.

Calculate BMI using Height at Visit 1. BMI = weight  $(kg)/height (m)^2$ . Please delete Missing row when there are no missing values.

Table 1.5.2Demographics and Baseline CharacteristicsAnalysis Set: ITT Analysis Set

Table 1.5.3 Demographics and Baseline Characteristics Analysis Set: Safety Analysis Set

Note to Programmer: Remove Table 1.5.3 if Safety Analysis Set is the same as the ITT Analysis Set.

Table 1.5.4 Demographics and Baseline Characteristics

Analysis Set: All Subjects Not Randomized


Table 1.6.1 Duration of Asthma Analysis Set: mITT Analysis Set

| | (XXX=Z) |
|---------------------------------|---------|
| Duration of Asthma (months) [a] | |
| | XXX |
| Mean | XX.X |
| | XX.X |
| 25 <sup>th</sup> Percentile | XX.X |
| Median | XX.X |
| 75 <sup>th</sup> Percentile | XX.X |
| Minimum | XX.X |
| Maximum | x.xx |

Notes to Programmer: Duration of Asthma = (First Dose date of Study Treatment - Date Asthma First Diagnosed)/30.4375, where day of Asthma diagnosed is assumed to be the  $1^{st}$  of the month.

Report generated by program: PT007001/sasdir/programs/statout/t010601.sas Version YYYY-MM-DD xx:xx (Page n of N)

Table 1.6.2 Duration of Asthma Analysis Set: Safety Analysis Set


Table 1.7.1 Screening Pre- and Post-Bronchodilator and Baseline Spirometry Parameters
Analysis Set: mITT Analysis Set

| | All Subjects (N=xxx) |
|------------------------------------------|----------------------|
| 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
| Fev1 (8 predicted) | |
| Visit 1 [a] | |
| Pre-Ventolin HFA: | |
| n | XX |
| Mean | XX.XXX |
| SD | XX.XXX |
| 25 <sup>th</sup> Percentile | XX.XXX |
| Median | XX.XXX |
| 75 <sup>th</sup> Percentile | XX.XXX |
| Minimum | XX.XXX |
| Maximum | XX.XXX |
| Post-Ventolin HFA: | |
| | ×× |
| i W | 000 000 |
| Meall | VYY.VYV |
| Qss. | XX.XX |
| 25th Percentile | XX.XXX |
| Median | XX.XX |
| 75 <sup>th</sup> Percentile | XX.XX |
| Minimum | XX.XXX |
| Maximum | XX.XXX |
| () ( | |
| VISIC Z (FIE-GOSE)<br>Pre-Ventolin HFA: | |
| n | XX |
| Mean | XXX.XX |
| SD | XX.XXX |
| 25 <sup>th</sup> Percentile | XX.XXX |
| Median | XX.XXX |
| 75 <sup>th</sup> Percentile | XX.XXX |
| Minimum | XX.XXX |
| Maximum | XX.XXX |
| Dost-Ventolin HRA. | |
| | ×× |
| Mean | XXX.XX |
| SD | XX. |
| 25 <sup>th</sup> Percentile | XX.XX |
| Median | XXX.XX |


75<sup>th</sup> Percentile Minimum Maximum

Repeat the above for these parameters:

 $FEV_I(L)$ 

FVC (% predicted) FVC (L) FEF 25-75 (% predicted) FEF 25-75 (L/sec)

[a] Visit 1, for this purpose, was Visit 1, 1a, or 1b, whichever visit had the highest  ${\rm FEV_1}$  result post-dose.

Report generated by program: PT007001/sasdir/programs/statout/t010701.sas Version YYYY-MM-DD (Page n of N) xx:xx

Table 1.7.2 Screening Pre- and Post-Bronchodilator and Baseline Spirometry Parameters Analysis Set: ITT Analysis Set


Table 1.8.1 Reversibility to Ventolin HFA at Screening Analysis Set: mITT Analysis Set

| | All Subjects (N=xxx) |
|---|---|
| Post-Ventolin HFA FEV <sub>1</sub> - Pre-Ventolin HFA FEV <sub>1</sub> (mL) | |
| n | XX |
| Mean | xx.x |
| SD | XX.X |
| Median | XX.X |
| Minimum | XX.X |
| Maximum | x.xx |
| Reversibility (%) Post-Ventolin HFA for FEV1 [a] | |
| n | XX |
| Mean | XX.X |
| SD | XX.X |
| Median | XX.X |
| Minim | XX.X |
| Maximum | xx.x |
| Reversible [b], n (%) | XX (XX.X) |

If a subject was missing a Post- or Pre-Ventolin HFA FEV; value at Screening Visit 1, these values were replaced by the Pre- and Post-Ventolin HFA values from Screening Visit 1a. Similarly, if values were missing at Screening Visits 1 and 1a, the values were replaced by those from Screening Visit 1b.

- [a] Reversibility (%) is defined as 100 x (the change from pre-Ventolin HFA to post for FEV,)/pre-Ventolin HFA FEV1.
  - Reversible is defined as Improvement in FEV1 post-Ventolin HFA administration compared to pre-Ventolin HFA of >=15%. [9]

Report generated by program: PT007001/sasdir/programs/statout/t010801.sas Version YYYY-MM-DD xx:xx (Page n of N)

Table 1.8.2 Reversibility to Ventolin HFA at Screening Analysis Set: ITT Analysis Set


Table 1.9 Medical/Surgical History Analysis Set: Safety Analysis Set

| | All subjects (N=xxx) |
|--------------------------------------|----------------------|
| | n (%) |
| Subject Had Medical/Surgical History | |
| No | XXX (XX.X) |
| Yes | XXX (XX.X) |
| Cardiovascular | XXX (XX.X) |
| CNS/Neurological | XXX (XX.X) |
| Dermatologic | XXX (XX.X) |
| Drug Allergy | XXX (XX.X) |
| BENT | XXX (XX.X) |
| Endocrine/Metabolic | XXX (XX.X) |
| Gastrointestinal | XXX (XX.X) |
| Genitourinary | XXX (XX.X) |
| Hepatic | XXX (XX.X) |
| Hematologic | XXX (XX.X) |
| Immunological | XXX (XX.X) |
| Malignancy | XXX (XX.X) |
| Musculoskeletal | XXX (XX.X) |
| Psychiatric | XXX (XX.X) |
| Respiratory | XXX (XX.X) |
| Renal | XXX (XX.X) |
| Other | XXX (XX.X) |

Report generated by program: PT007001/sasdir/programs/statout/t0109.sas Version YYYY-MM-DD xx:xx (Page n of N)

Note to Programmer: Please sort by descending frequency of occurrence in All Subjects. Denominator should be N from the column header for a treatment.


).1 Prior Medications – Asthma-Related Analysis Set: Safety Analysis Set Table 1.10.1

| | All Subjects |
|---|---|
| | (N=XXX) |
| Preferred Term | n (%) |
| Any Prior Asthma Medication | xxx (xx.x) |
| Medication 1 | XXX (XX.X) |
| Medication 2 | xxx (xx.x) |
| Preferred term is according to WHODRUG Qxxxx. | |
| Report generated by program: PT007001/sasdir/programs/statout/t011001.sas Version YYYY-MM-DD xx:xx (Page n of N) | 011001.sas Version YYYY-MM-DD xx:xx |

Notes to Programmer: Sort Medications by descending frequency of use in All Subjects.

Prior Medications-Other than Asthma-Related Table 1.10.2 Prior Medication Analysis Set: Safety Analysis Set

Notes to Programmer: Sort Medications by descending frequency of use for All Subjects. Add a row for "Any Prior Other Medication".


Table 1.11.1a Concomitant Medications During Treatment Period – Asthma-Related Analysis Set: Safety Analysis Set

| | | AS MDI | AS MDI | Proventil 90 | Proventil 180 |
|---|---|---|---|---|---|
| | Placebo | 90 pd | 180 µg | hg | рц |
| | (N=XXX) | (N=xxx) | (N=XXX) | (N=XXX) | (N=XXX) |
| Preferred Term | (%) u | (%) u | (%) u | (%) u | (%) u |
| Any Concomitant Asthma Medication | (x.xx) xxx | (x.xx) xxx | (x.xx) xxx | xxx (xxxx) | (x.xx) xxx |
| Medication 1 | (x.xx) xxx | (x.xx) xxx | (xxx) xxx | (xxx) xxx | (x.xx) xxx |
| Medication 2 | (x.xx) xxx | (x.xx) xxx | xxx (xx.x) | xxx (xx.x) | (x.xx) xxx |
| Preferred term is according to WHODRUG Qxxxx.<br>All subjects were allowed only sponsor-provided Ventolin HFA and/or Pulmicort Flexhaler for relief of symptoms.<br>See Listing 6.4 for the use of Ventolin HFA as rescue medication. | JG Qxxxx.<br>>r-provided Ventc<br>lin HFA as rescue | lin HFA and/or Pul<br>medication. | lmicort Flexhaler | for relief of sympi | oms. |
| Report generated by program: PT007001/sasdir/programs/statout/t011101a.sas Version | 1/sasdir/programs | s/statout/t011101a. | | YYYY-MM-DD xx:xx | (Page n of |

Notes to Programmer: Sort Medications by descending frequency of use in All Subjects.

Table 1.11.1b Concomitant Medications During Washout Period – Asthma-Related Analysis Set: Safety Analysis Set

| Period just prior to the washout.<br>ler for relief of symptoms. | YYYY-MM-DD xx:xx (Page n of |
|---|---|
| Concomitant medications are tabulated by the treatment received during the Treatment Period just prior to the washout. Preferred term is according to WHODRUG Qxxxx. All subjects were allowed only sponsor-provided Ventolin HFA and/or Pulmicort Flexhaler for relief of symptoms. See Listing 6.4 for the use of Ventolin HFA as rescue medication. | <pre>teport generated by program: PT007001/sasdir/programs/statout/t011101b.sas Version YYYY-MM-DD xx:xx</pre> |
| Concomitant medications are tabula<br>Preferred term is according to WHAII subjects were allowed only spo<br>See Listing 6.4 for the use of Ver | Report generated N) |

Table 1.11.2.a Concomitant MedicationsDuring Treatment Period-Non-Asthma Related

Analysis Set: Safety Analysis Set

Notes to Programmer: Sort Medications by descending frequency of use in All Subjects. Add a row for "Any Concomitant Other Medication".

Table 1.11.2b Concomitant Medications During Washout Period-Non-Asthma Related Analysis Set: Safety Analysis Set

Notes to Programmer: Sort Medications by descending frequency of use in All Subjects. Add a row for "Any Concomitant Other Medication


# 2. Efficacy Summary Tables and Figures

## Primary Efficacy Endpoint


Table 2.1.1 Change from Baseline in FEV<sub>1</sub> AUC<sub>0-6</sub> (L) Overall and by ICS Use Subgroups Analysis Set: mITT Analysis Set

| | | Change From | | LS Mean Differences | s Between Treatments | |
|---|---|---|---|---|---|---|
| Treatment | Baseline ${\tt FEV}_1$ | AUC <sub>0-6</sub> | Placebo | AS MDI 90 µg | Proventil 180 µg | Proventil 90 µg |
| Combined ICS Use | e Groups [a] | | | | | |
| AS MDI 180 µg | | | | | | |
| N | ×× | XX | | | | |
| Mean | x.xx | x.xx | | | | |
| SD | x.xx | ×.xx | | | | |
| Median | x.xx | x.xx | | | | |
| | XXX-X-XXX | xxx-x-xxx | | | | |
| LS Mean (SE) | | X.XXX () | (X.XXX) | X.XXX (X.XXXX) | X.XXX (X.XXXX) | (X.XXX) |
| 95% CI | | ( ××××× ) | (XXXX, XXXX) | (XXXX, XXXX) | ( x.xxx, x.xxx) | ( x.xx, x.xxx) |
| | | X.XXX) | | | | |
| P-value | | | X.XXX | x.xxxx | x.xxxx | |
| AS MDI 90 µg | | | | | | |
| Z | XX | ×× | | | | |
| Mean | x.xxx | x.xx | | | | |
| SD | XXXX.X | X.XXX | | | | |
| Median | x.xxx | x.xxx | | | | |
| Min-Max | xxx-x-xxx | xxx-x-xxx | | | | |
| LS Mean (SE) | | x.xxx<br>(x.xxxx) | x.xxx (x.xxxx) | Not Applicable | x.xxx (x.xxxx) | x.xxx (x.xxxx) |
| 95% CI | | ( x.xxx, x x x x x x x x x x x x x x x x | ( x.xx, x.xxx) | | ( x.xx, x.xxx) | ( x.xx, x.xxx) |
| P-value | | 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 4 | ×××× × | | | ×××× × |
| Proventil 180 µg | Z, | | | | | |
| Z | ×× | ×× | | | | |
| Mean | X.XXX | X.XXX | | | | |
| SD | X.XXX | ×.xxx | | | | |
| Median | X.XXX | X.XX. | | | | |
| | X.XX-X.XXX | XXXX-XXXX | | | | |
| LS Mean (SE) | | x.xxx<br>(x.xxxx) | x.xxx (x.xxxx) | Shown Above | Not Applicable | x.xxx (x.xxxx) |
| 95% CI | | ( X.XX., | ( x.xx, x.xxx) | | | ( x.xx, x.xx) |
| 1 | | ×.xxx) | | | | |
| P-value | | | x.xxx | | | xxxxx x |
| Proventil 90 | | | | | | |
| ) | XX | | | | | |


| | | Change From | | LS Mean Difference | LS Mean Differences Between Treatments | |
|---|---|---|---|---|---|---|
| Treatment | Baseline $\mathtt{FEV}_1$ | Baseline<br>AUC <sub>0-6</sub> | Placebo | AS MDI 90 µg | Proventil 180 µg | Proventil 90 µg |
| Mean | x.xxx | | | | | 1 |
| SD | X.XXX | | | | | |
| Median | x.xxx | | | | | |
| Min-Max | XXXX-X-XXX | | | | | |
| LS Mean (SE) | | x.xxx | (X.XXXX) | Shown Above | Shown Above | Not Applicable |
| | | (X.XXXX) | | | | |
| 95% CI | | ( x.xx, | ( x.xx, x.xxx) | | | |
| | | x.xxx) | | | | |
| P-value | | | X.XXXX | | | |
| Placebo | | | | | | |
| Z | XX | | | | | |
| Mean | X.XXX | | | | | |
| SD | x.xxx | | | | | |
| Median | x.xx | | | | | |
| Min-Max | ×. x. x-x. x | | | | | |
| LS Mean (SE) | | x.xxx | Not Applicable | Shown Above | Shown Above | Shown Above |
| | | (x.xxxx) | | | | |
| 95% CI | | ( x.xxx, | | | | |
| | | (××××) | | | | |
| Repeat Above for: | г: | | | | | |
| Subgroup: ICS Use | se at Screening [b] | [q] | | | | |
| Repeat Above for:<br>Subgroup: Did Not | Repeat Above for:<br>Subgroup: Did Not Use ICS at Screening [b] | reening [b] | | | | |
| Treatment-by-Sul | Treatment-by-Subgroup Interaction P-value: 0.xxxx | on P-value: 0.xx | XX | | | |

A linear mixed effect model with a random subject effect for the correlation across periods and fixed effects for treatment, A linear mixed effect model with a random subject effect and fixed effects for treatment, treatment sequence, baseline FEV1, period, ICS Use subgroup, and treatment-by-subgroup interaction. The p-value is for the superiority comparison of AS MDI or Proventil to Placebo. The non-inferiority of AS MDI 180 µg to Proventil 180 µg or of AS MDI 90 µg to Proventil 90 µg is concluded when the lower CI limit for the difference between Baseline is defined as the mean of evaluable 60 and 30 minute pre-dose values across Visits 2, 3, 4, 5, and 6. LS Mean = least squares mean from the the linear mixed effects model treatment sequence, baseline  ${ t FEV}_1$ , and period. [a] Combined ICS Use Groups Model: ICS = Inhaled Corticosteroid [b] ICS Use Subgroups Model: treatments is >-100 mL.

Report generated by program: PT007001/sasdir/programs/statout/t020101.sas Version YYYY-MM-DD hh:mm

(Page n of N)


Table 2.1.2 Change from Baseline in  $FEV_1$   $AUC_{0-6}$  (L) Overall and by ICS Use Subgroups Analysis Set: ITT Analysis Set

## Secondary Efficacy Endpoints

Table 2.2.1 Change from Baseline in  $FEV_1$   $AUC_{0-4}$  (L) Analysis Set: mITT Analysis Set

Notes to Programmer: Follow the format of Table 2.1.1.

Table 2.2.2Peak Change from Baseline in FEV1 (L)Analysis Set: mITT Analysis Set

Notes to Programmer: Follow the format of Table 2.1.1.


## Other Efficacy Endpoints

Table 2.3.1 Change from Baseline in FEV<sub>1</sub> (L) by Timepoint Analysis Set: mITT Analysis Set

| | | 田<br>り<br>と<br>と<br>は<br>た<br>に<br>れ<br>り | | LS Mean Difference | LS Mean Differences Between Treatments | |
|---|---|---|---|---|---|---|
| Treatment | Baseline ${\tt FEV}_1$ | Baseline | Placebo | AS MDI 90 µg | Proventil 180 µg | Proventil 90 µg |
| 5 Minutes Post- | Post-Dose [a] | | | | | |
| AS MDI 180 µg | | | | | | |
| Z | ×× | ×× | | | | |
| Mean | x.xxx | X.XXX | | | | |
| SD | X.XXX | x.xx | | | | |
| Median | X.XXX | x.xx | | | | |
| | XXXX-XXXX | XXXX-X.XXX | | | | |
| LS Mean (SE) | | x.xxx | X.XXX (X.XXXX) | X.XXX (X.XXXX) | X.XXX (X.XXXX) | X.XXX (X.XXXX) |
| | | (XXXXX) | | | | |
| ₩<br>₩ | | , ××××, × | ( x.xx, x.xxx) | ( ××××, ××××) | ( | ( X.XX, X.XXX) |
| P-value | | | X.XXX | X.XXXX | X.XXXX | |
| AS MDI 90 µg | | | | | | |
| | ×× | ×× | | | | |
| Mean | XXXX X | X.XXX | | | | |
| SD | x.xxx | x.xxx | | | | |
| Median | X.XXX | X.XXX | | | | |
| Min-Max | XXX-X.XXX | XXXX-X.XXX | | | | |
| LS Mean (SE) | | ××××× × | x.xxx (x.xxxx) | Not Applicable | x.xxx (x.xxxx) | (X.XXXX) |
| 95% CI | | ( X X X X ) | ( X.XXX, X.XXX) | | ( x.xx, x.xx) | ( x.xx, x.xxx) |
| P-value | | ( | X.XXX | | | X.XXXX |
| Proventil 180 µg | <u>.</u> | | | | | |
| Z | XX | ×× | | | | |
| Mean | x.xx | x.xx | | | | |
| SD | X.xxx | X.XXX | | | | |
| Median | X.XXX | XXX.X | | | | |
| | xxx-x.xxx | XXXX-XXXX | | | | |
| LS Mean (SE) | | xxxx.x | x.xxx (x.xxxx) | Shwon Above | Not Applicable | x.xxx (x.xxxx) |
| | | (x.xxx) | | | | , |
| www. | | ( ×.××, × | ( X.XX, X.XXX) | | | ( X.XX, X.XX) |
| P-value | | | XXXXX X | | | XXXXX X |


Albuterol Sulfate Pressurized Inhalation Suspension Protocol D6930C00001 (PT007001)

| | | でかった 日本の開 | | 2 | TO LICALI DIFFERENCES DOCUMENTS | |
|---|---|---|---|---|---|---|
| Treatment | Baseline ${\tt FEV}_1$ | Baseline | Placebo | AS MDI 90 µg | Proventil 180 µg | Proventil 90 µg |
| Proventil 90 µg | | | | | | |
| Z | ×× | | | | | |
| Mean | ×.×× | | | | | |
| SD | X.XXX | | | | | |
| Median | X.XXX | | | | | |
| Min-Max | XXX-X-XXX | | | | | |
| LS Mean (SE) | | XXXXX<br>(******) | x.xxx (x.xxxx) | Shown Above | Shown Above | Not Applicable |
| 95% CI | | ( x.xxx, x x x x x x x x x x x x x x x x | ( x.xx, x.xxx) | | | |
| P-value | | | X.XXX | | | |
| Placebo | | | | | | |
| N | ×× | | | | | |
| Mean | x.xxx | | | | | |
| SD | X.XXX | | | | | |
| Median | X.XXX | | | | | |
| Min-Max | XXX-X-XXX | | | | | |
| LS Mean (SE) | | x.xxx<br>(x.xxxx) | Not Applicable | Shown Above | Shown Above | Shown Above |
| 95% CI | | ( x.xx, x x x x x x x x x x x x x x x x x | | | | |


Figure 2.3.1.1 Change from Baseline in  $FEV_1(L) \pm SE$  Over Time Analysis Set: mITT Analysis Set



Source: Table 2.3.1

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/f02030101.sas Version YYYY-MM-DD xx:xx

Replace the treatment labels with 'AS MĎI 180 μg', 'AS MĎI 90 μg', 'Proventil 180 μg', 'Proventil 90 μg', and 'Placebo'. Replace y-axis label with 'FEV<sub>I</sub> Change From Baseline'. Notes to Programmer: Replace Number of Weeks Post-Dose with Number of Minutes Post-Dose.


Treatment Differences From Placebo\*: Change from Baseline in FEV $_1$  (L)  $\pm$  95% CI Over Time Analysis Set: mITT Analysis Set Figure 2.3.1.2



\*Differences of active treatments vs. Plabebo.

Source: Table 2.3.1

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/f02030102.sas Version YYYY-MM-DD xx:xx

Replace the treatment labels with 'AS MDI 180 µg', 'AS MDI 90 µg', 'Proventil 180 µg', and 'Proventil 90 µg' Notes to Programmer: Replace Number of Weeks Post-Dose with Number of Minutes Post-Dose. Replace y-axis label with 'FEV<sub>1</sub> Change From Baseline'.


Table 2.3.2 Time to Peak FEV<sub>1</sub> Analysis Set: mITT Analysis Set

| | Placebo<br>(N=xxx) | AS MDI<br>90 µg<br>(N=xxx) | AS MDI<br>180 µg<br>(N=xxx) | Proventil<br>90 µg<br>(N=xxx) | Proventil<br>180 µg<br>(N=xxx) |
|---|---|---|---|---|---|
| Subjects with a Post-Dose $FEV_1$ , n(%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | (xx) |
| Time to Peak $\mathrm{FEV}_1$ (mins) Median (Min, Max) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) | x.x (x.x, x.x) |
| Median Difference (95% CI) | | | | | |
| Placebo (n=xxx) | Not Applicable | X.XXX<br>(X.XX, X.XXX) | X.XXX<br>(X.XXX, X.XXX) | X.XXX<br>(X.XX, X.XXX) | x.xxx<br>(x.xx, x.xxx) |
| AS MDI 90 µg (n=xxx) | | Not Applicable | x.xxx<br>(x.xxx, x.xxx) | x.xxx<br>(x.xxx, x.xxx) | X.xxx<br>(X.xxx, X.xxx) |
| AS MDI 180 µg (n=xxx) | | | Not Applicable | x.xxx<br>(x.xxx, x.xxx) | X.xxx<br>(X.xxx, X.xxx) |
| Proventil 90 µg (n=xxx) | | | | Not Applicable | X.XXX<br>(X.XX, X.XXX) |

Time to Peak FEV1 (mins) = (time of Peak FEV1 - treatment administration time). Time to peak is calculated only for subjects with a post-dose FEV $_1$ . 95% CI's of the median differences were calculated with Hodges-Lehmann CI's for paired observations.

Report generated by program: <study>/sasdir/programs/statout/t020302.sas <VERSION TYPE> YYYY-MM-DD xx:xx

 $\widehat{\mathbb{Z}}$ 

(Page n of

Notes to Programmer: Use data up to the last assessment for each visit.


Percentage of Subjects Achieving a 12% or 15% Improvement in FEV<sub>1</sub> from Baseline Within 30 Minutes Post-Dose Analysis Set: mITT Analysis Set

Table 2.3.3

| | Placebo<br>(N=xxx) | AS MDI<br>90 µg<br>(N=xxx) | AS MDI<br>180 µg<br>(N=xxx) | Proventil<br>90 µg<br>(N=xxx) | Proventil<br>180 µg<br>(N=xxx) |
|---|---|---|---|---|---|
| Reason for | n (%) | n (%) | n (%) | n (%) | n (%) |
| Subjects Achieving 12% Improvement in FEV, from Baseline Within 30 Minutes of Dose | (xx.x) | (xx) xx | xx (xx.x) | (xx) xx | (xx.x) |
| Odds Ratio (95% CI) | | | | | |
| Placebo (n=xxx) | Not Applicable | X.XXX<br>(X.XX, X.XXX) | x.xxx<br>(x.xx, x.xxx) | x.xxx<br>(x.xx, x.xxx) | X.XXX<br>(X.XX, X.XXX) |
| AS MDI 90 µg (n=xxx) | | Not Applicable | x.xxx<br>(x.xx, x.xxx) | x.xxx<br>(x.xx, x.xxx) | x.xxx<br>(x.xx, x.xxx) |
| AS MDI 180 µg (n=xxx) | | | Not Applicable | x.xxx<br>(x.xxx, x.xxx) | x.xxx<br>(x.xxx, x.xxx) |
| Proventil 90 µg (n=xxx) | | | | Not Applicable | X.XXX<br>(X.XX, X.XXX) |
| Subjects Achieving 15% Improvement in FEV1 from Baseline Within 30 Minutes of Dose | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Odds Ratio (95% CI) | | | | | |
| Placebo (n=xxx) | Not Applicable | X.XXX<br>(X.XX, X.XXX) | X.XXX<br>(X.XX, X.XXX) | x.xxx<br>(x.xx, x.xxx) | xxxx (x.xxx, x.xxx) |
| AS MDI 90 µg (n=xxx) | | Not Applicable | x.xxx<br>(x.xx, x.xxx) | x.xxx<br>(x.xx, x.xxx) | x.xxx<br>(x.xx, x.xxx) |
| AS MDI 180 µg (n=xxx) | | | Not Applicable | x.xxx<br>(x.xx, x.xxx) | x.xxx<br>(x.xx, x.xxx) |
| Proventil 90 µg (n=xxx) | | | | Not Applicable | x.xxx<br>(x.xx, x.xxx) |


N is the number of subjects with at least one post-dose  $FEV_1$  assessment within 30 minutes of dose. n is the number of subjects who did or did not achieve 12% or 15% improvement in  $FEV_1$  from baseline within 30 minutes of dose. The odds ratios are calculated from a a generalized mixed effects model with treatment as a fixed effect and the intercept for each subject as a random effect.

(Page n of Report generated by program: PT007001/sasdir/programs/statout/t020303.sas Version YYYY-MM-DD xx:xx

â

Table 2.3.4 Time to Onset of 12% Improvement in FEV<sub>1</sub>

Analysis Set: mITT Analysis Set

Note to the Programmer: Use shell for Table 2.3.2.

Replace footnote: Time to Onset of Response (minutes) =  $(time\ of\ first\ achievement\ of\ a\ 12\%$  increase in  $FEVI\ from\ baseline,\ within\ 30\ minutes\ of\ dose$ treatment administration time).

Table 2.3.5 Time to Onset of 15% Improvement in FEV<sub>1</sub>

Analysis Set: mITT Analysis Set

Note to the Programmer: Use shell for Table 2.3.2.

Replace footnote: Time to Onset of Response (minutes) =  $(time\ of\ first\ achievement\ of\ a\ 15\%$  increase in  $FEVI\ from\ baseline,\ within\ 30$  minutes of dose treatment administration time).


Table 2.3.6 Duration of 12% Improvement in FEV<sub>1</sub>
Analysis Set: mITT Analysis Set

| | | | LS | Mean Differences | LS Mean Differences Between Treatments | ts |
|---|---|---|---|---|---|---|
| | Duration of<br>Response (mins) | Placebo<br>(N=xxx) | AS MDI<br>90 µg<br>(N=xxx) | AS MDI<br>180 µg<br>(N=xxx) | Proventil<br>90 µg<br>(N=xxx) | Proventil<br>180 µg<br>(N=xxx) |
| Subjects with a 12% increase in FEV; from baseline, within 30 minutes of dose, n(%) | | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Placebo (n=xxx) N Mean SD Median Min, Max LS Mean (SE) | xx xxx xx | Not Applicable | X X X X X X X X X X X X X X X X X X X | (XXX.X) (XXX.X) | X X X X X X X X X X X X X X X X X X X | (*** * *** * ) (*** * * * * * * ) |
| P-value | | | XXXX.X | XXXXX.X | XXXX.X | XXXX.X |
| AS MDI 90 µg (n=xxx) N Mean SD Median Min, Max LS Mean (SE) 95% CI P-value | xx<br>xxx.xx<br>xxx.xx<br>x.x<br>(x.x, x.x) | | Not Applicable | x.xxx<br>(x.xxxxx)<br>x.xxx, x.xxx) | x.xxx (x.xxxx x x x x x x x x x x x x x | x.xxx<br>(x.xxxx)<br>(x.xxxx)<br>x.xxxx |
| AS MDI 180 ug (n=xxx) N Mean SD Acdian Min, Max LS Mean (SE) 95% CI P-value | ** *** *** *** *** *** (*.*, *.*) | | | Not Applicable | (x.xxxx)<br>(x.xxxx, x.xxx)<br>x.xxxx | x.xxx<br>(x.xxxx)<br>(x.xxx, x.xxx)<br>x.xxxx |


```
( xxxx, x.xxx)
                                                                                                                                                                                                                Not Applicable
                                                                             x.xxx
                                                                                         (xxxxx)
                                                                                                                 \times \times \times
                                                                            Not Applicable
                                                                                                                                                                                                                 Shown Above
                                                                                                                                                                                                                 Shown Above
                                                                                                                                                                                                                 Shown Above
                                                                                                                                                                                                                 Shown Above
                                                                 (x.x, x.x)
                                                                                                                                                                                                      (x.x, x.x)
                                        xxx.xx
                                                                                                                                                                             xx.xx
                             xxx.x
                                                                                                                                                                 \times \times \times \times
                                                    ×
                                                                                                                                                                                           ×
                                                                                                                                                     ×
                                                                                                                                       Proventil 180 µg (n=xxx)
Proventil 90 µg (n=xxx)
                                                                            LS Mean (SE)
                                                                                                                                                                                                                LS Mean (SE)
                                                               Min, Max
                                                                                                                                                                                                     Min, Max
                                                                                                              P-value
                                                                                                                                                                                                                                          P-value
                                                                                                  95% CI
                                                                                                                                                                                                                            95% CI
                                                   Median
                                                                                                                                                                                        Median
                           Mean
                                                                                                                                                                Mean
```

Duration of response (mins) = (time of offset - time of onset) where onset is defined as a 2 12% improvement from baseline in FEV1 within the 30 minutes post dose. If a subject had a 2<sup>nd</sup> onset of response subsequent to achievement of offset, their data for that LS Means (SE), 95% CIs, and P-values are from a linear mixed effect model with a random subject effect for the correlation across periods and fixed effects for treatment, treatment sequence, and period. period was excluded from the duration of response analysis.

 $\hat{z}$ 

(Page n of

Notes to Programmer: Use data up to the last assessment for each visit.

Report generated by program: <study>/sasdir/programs/statout/t020302.sas <VERSION TYPE> YYYY-MM-DD xx:xx

The linear mixed model will be replaced with a distribution-free method (Hodges-Lehmann) as appropriate to the data.

time of the last available assessment – treatment administration time. Thus, Offset of Response: For responders only: the 1st time point after achievement of response for which the increase from baseline in FEV1 is < 15% (or 12%). If offset is not achieved according to this definition, and the last available assessment is >= 15% (or 12%), offset will be treatment administration time). If offset of FEV1 < 15% (or 12%) is not achieved and the last available assessment is  $\geq$  15% (or 12%), the time to offset will be defined as (the Time to Offset of Response: For responders only: (time of first assessment after achievement of response for which the increase from baseline in FEV1 is < 15% (or 12%) — Time to Onset of Response (minutes) = (time of first achievement of a 12% increase in FEVI from baseline, within 30 minutes of dose – treatment administration time). defined as the time of the last available assessment.

Duration of response is defined n the table footnote above.:

Duration of 12% Improvement in FEV<sub>1</sub>: Subjects who Have Assessments at the 180- and 300-Minute Post-Dose Timepoints Analysis Set: mITT Analysis Set 

Table 2.3.8 Duration of 15% Improvement in FEV<sub>1</sub> Analysis Set: mITT Analysis Set

Notes to Programmer: Replace Duration footnote with: Duration of response (mins) = (time of offset – time of onset) where onset is defined as  $a \ge 15\%$  improvement from baseline in FEV1 within the 30 minutes post dose. If a subject had a  $2^{nd}$  onset of response subsequent to achievement of offset, their data for that period was excluded from the duration of response analysis.

Duration of 15% Improvement in FEV<sub>1</sub>: Subjects who Have Assessments at the 180- and 300-Minute Post-Dose Timepoints Analysis Set: mITT Analysis Set Table 2.3.9


#### 3. Safety

### Adverse Events

Overall Summary of Treatment-Emergent Adverse Events Analysis Set: Safety Analysis Set Table 3.1.1

| | Placebo<br>(N=xxx) | AS MDI 90 µg (N=xxx) | AS MDI 180 µg (N=xxx) | Proventil 90 µg (N=xxx) | Proventil 180 µg (N=xxx) |
|---|---|---|---|---|---|
| | n (%) | (%) u | (%) u | (%) u | (%) u |
| | [Events] | [Events] | [Events] | [Events] | [Events] |
| Subjects With at Least One TEAE [a] [b] | (x.xx) xx | (x.xx) xx | (xxxx) xx | (x.xx) xx | xx (xx.x) |
| | [xxx] | [xxx] | [xxx] | [xxx] | [xxx] |
| Subjects With Serious TEAEs | XX (XX.X) | (xxxx) xx | (xx.x) | xx (xx.x) | (xx.x) |
| | [xx.x] | [xxx] | [xx.x] | [xxx] | [xx.x] |
| Subjects With TEAEs Related to Study | (xxxx) xx | (×.×.) ×× | (×.×.) ×× | (xx.x) | xx (xx.x) |
| Treatment [c] | [xxx] | [xxx] | [xxx] | [xxx] | [xxx] |
| Subjects With Serious TEAEs Related to Study | (xxxx) xx | (x.xx) xx | (x.xx) xx | xx (xx.x) | xx (xx.x) |
| Treatment [c] | [xx.x] | [xxx] | [xx.x] | [xxx] | [xx.x] |
| Subjects With TEAEs Leading to Early | (x.xx) xx | (×.*x) ×x | (×.×.) ×× | (x.x.x) | (x.xx) xx |
| Discontinuation | [xxx] | [xx.x] | [xx.x] | [xx.x] | [xx.x] |
| Deaths - All Causes | (x.xx) xx | (x.xx) xx | (xx.x) | xx (xx.x) | (x.x) xx |

Report generated by program: PT007001/sasdir/programs/statout/t030101.sas Version YYYY-MM-DD xx:xx

(Page n of N)

<sup>[</sup>a] TEAE = Treatment-Emergent Adverse Event [a] Only adverse events on a Treatment Day were included in this table. [c] Related = Yes or No.

Overall Summary of Treatment-Emergent Adverse Events Including Adverse Events on a Treatment Day or During the Washout or Follow-up Table 3.1.2

Periods Analysis Set: Safety Analysis Set

| | Placebo<br>(N=xxx) | AS MDI 90 µg (N=xxx) | AS MDI 180 µg (N=xxx) | Proventil 90 µg (N=xxx) | Proventil 180 µg (N=xxx) |
|---|---|---|---|---|---|
| | (%) u | (%) u | (%) u | n (%) | (%) u |
| | [Events] | [Events] | [Events] | [Events] | [Events] |
| Subjects With at Least One TEAE [a] | (x.xx) xx | (x.xx) xx | (xxxx) xx | (x.xx) xx | xx (xx.x) |
| | [xxx] | [xxx] | [xxx] | [xxx] | [xxx] |
| Subjects With Serious TEAEs | xx (xx.x) | XX (XX.X) | (xx.x) | XX (XX.X) | (xx.x) |
| | [xx.x] | [x.x.] | [xx.x] | [xxx] | [x.x] |
| Subjects With TEAEs Related to Study | (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment [b] | [xxx] | [xxx] | [xxx] | [xxx] | [xxx] |
| Subjects With Serious TEAEs Related to Study | (xx.xx) | (x.xx) xx | (x.xx) xx | xx (xx.x) | xx (xx.x) |
| Treatment [b] | [xx.x] | [xx.x] | [xx.x] | [xxx] | [xx.x] |
| Subjects With TEAEs Leading to Early | xx (xx.x) | (x.xx) xx | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinuation | [x.x.x] | [xx.x] | [xx.x] | [xx.x] | [xx.x] |
| Deaths - All Causes | (x.xx) xx | (x.x.) | xx (xx.x) | (xx.x) | (xx.x) |

[a] TEAE = Treatment-Emergent Adverse Event [b] Related = Yes or No.

Report generated by program: PT007001/sasdir/programs/statout/t030102.sas Version YYYY-MM-DD xx:xx

(Page n of N)


Treatment-Emergent Adverse Events by MedDRA Primary System Organ Class and Preferred Term Analysis Set: Safety Analysis Set Table 3.2.1

| | Placebo<br>(N=xxx) | AS MDI 90 µg (N=xxx) | AS MDI 180 µg<br>(N=xxx) | Proventil 90 µg (N=xxx) | Proventil 90 µg Proventil 180 µg (N=xxx) |
|---|---|---|---|---|---|
| System Organ Class | u (%) | n (%) | n (%) | n (%) | n (%) |
| Preferred Term | [Events] | [Events] | [Events] | [Events] | [Events] |
| At Least One TEAE [a] | ( xx.x) xx | ( xx.x) | ( x x x x x x x x x x x x x x x x x x x | ( xx.xx ) xx | ( xx.x) xx |
| | [xx] | [xx] | [xx] | [xx] | [xx] |
| System Organ Class 1 | ( xx x x x x x x x x x x x x x x x x x | ( x x x ) xx | ( | ( | ( x x x ) xx |
| | [xx] | [xx] | [xx] | [xx] | [xx] |
| Preferred Term 1 | ( xx x x x x x x x x x x x x x x x x x | ( x x x ) xx | xx ( xx.x) | ( | ( x x x ) xx |
| | [xx] | [xx] | [xx] | [xx] | [xx] |
| Preferred Term 2 | ( xx.x) | xx (xxxx) | xx (xxx.x) | xx (xx.x) | ( xx.x) xx |
| | [xx] | [xx] | [xx] | [xx] | [xx] |
| System Organ Class 2 | ( xx x x x x x x x x x x x x x x x x x | ( x x x ) xx | ( | ( | ( x x x ) xx |
| | [xx] | [xx] | [xx] | [xx] | [xx] |
| Preferred Term 1 | ( xx x x x x x x x x x x x x x x x x x | ( x · x x ) x × | ( | ( | ( |
| | [xx] | [xx] | [xx] | [xx] | [xx] |
| Preferred Term 2 | ( xx x x x x x x x x x x x x x x x x x | ( x · x x ) x × | ( | ( | ( |
| | [xx] | [xx] | [xx] | [xx] | [xx] |
| Etc | | | | | |
| <pre>[a] TEAE = Treatment-Emergent Adverse Event</pre> | 1t. | | | | |

Report generated by program: PT007001/sasdir/programs/statout/t030201.sas Version YYYY-MM-DD xx:xx

(Page n of N)

Treatment-Emergent Adverse Events by MedDRA Primary System Organ Class and Preferred Term Including Events Occurring During the Washout or Follow-up Periods: Sensitivity Analysis Analysis Set: Safety Analysis Set Table 3.2.2

Treatment Period. Add the following footnote: "AEs that occur during the Washout or Follow-up periods are attributed to the treatment given in the preceding Treatment Period." Notes to Programmer: Same as Table 3.2.1, however, AEs that occur during the Washout Period or Follow-up periods are attributed to the treatment given in the preceding

Treatment-Emergent Adverse Events Occurring in >=2% of Subjects in a Treatment by Descending Frequency Analysis Set: Safety Analysis Set Table 3.2.3

Notes to Programmer: Sort preferred terms by descending frequency of number of events across All Subjects. Use the format of Table 3.2.1, but delete the "At Least One" row from this Table. SOCs will not be used in this Table. Non-serious Treatment-Emergent Adverse Events Occurring in >=5% of Subjects in a Treatment by MedDRA Primary System Organ Class and Preferred Term Table 3.2.4

Analysis Set: Safety Analysis Set

Notes to Programmer: use the format of Table 3.2.1.


Treatment-Related Treatment-Emergent Adverse Events by MedDRA Primary System Organ Class and Preferred Term Analysis Set: Safety Analysis Set Table 3.3

[a] Related = Yes or No.

(Page n of N) Version YYYY-MM-DD xx:xx Report generated by program: PT007001/sasdir/programs/statout/t0304.sas

Notes to Programmer: use the format of Table 3.2.1.

Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by MedDRA Primary System Organ Class and Preferred Term Analysis Set: Safety Analysis Set Table 3.4

[a] A TEAE leading to treatment discontinuation is an AE with 'Action Taken' = 'Drug withdrawn', or 'Outcome' = 'Fatal', or 'Death' as reason for Seriousness on Adverse Event' CRF.

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/t0305.sas Version YYYY-MM-DD xx:xx

Notes to Programmer: use the format of Table 3.2.1.


Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment Analysis Set: All Subjects Randomized Table 3.5

| Subject | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ΠD | | | | Onset | | | | | | | |
| (Age/ | | | | Date | | | | | | | |
| Gender/ | | | | (Study | Duration | | | | | | Study Day |
| Race) | Primary System | AE Verbatim | Treat. Event | Day) | of Event | | Relation | | AE | Outcome | Resolved/ |
| [a] | Organ Class | (Preferred Term) | Emerg. Serious | [p] | [c] | Severity | -ship Action | Action | Treated (Death) | (Death) | Death [b] |

Treatment: AS MDI 180 µg, AS MDI 90 µg, Placebo, Proventil 180 µg, or Proventil 90 µg

| (XXXXXXXXXX) |
|---------------|
| ### |
| Center |
| (Investigator |
| # |
| Center |

| T2 _ P3 |
|----------------------------------------------------------------------|
| Recoverin<br>g/Resolvi<br>ng (No)<br>Recovered<br>/Resolved<br>(Yes) |
| N Kes |
| Dose<br>not<br>changed<br>Drug<br>Interru<br>pted |
| Not<br>Related<br>Related |
| Moderate<br>Moderate |
| × |
| YYYY-MM-<br>DD<br>(T1_2)<br>YYYY-MM-<br>DD<br>(T2_P1) |
| No Yes |
| Yes Yes |
| AE 1 (XXXXXXXXXX) AE 2 (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| (54/F/W) xxx xxx xxxxx xxxxxxxxxxxxxxxxxxxxxxx |

Race: A-Asian, AIAN-American Indian or Alaska Native, B-Black or African American, NHPI-Native Hawaiian or Other Pacific Islander O=Other W=White. Gender: F=Female, M=Male.

# indicates that it could not be determined whether the AE had onset during study treatment. = System Organ Class. SOC

A negative number for study day denotes the number of days prior to the start of study treatment. Otherwise, Study Day is Date Date of dose in the Period + 1. Tx = Period. Tx\_y = Period and Day within Period. Pxx = Days after dose in the last Treatment [a]

On Study Day 1, an 0 indicates that event started before study drug administration. On Study Day 1, 00 indicates that event started after study drug administration. Duration of Event = Stop Day - Onset Day + 1

<u></u>

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/t0305.sas Version YYYY-MM-DD xx:xx Notes to Programmer: Sort by Actual Treatment, Center, Subject ID, Primary System Organ Class, and Onset Day of AE. Page by Treatment and not by Treatment and Center.

Serious Adverse Events by MedDRA Primary System Organ Class and Preferred Term Analysis Set: Safety Analysis Set Table 3.6.1

Notes to Programmer: Same as Table 3.2.1.

Serious Adverse Events by MedDRA Primary System Organ Class and Preferred Term Including Events Occurring During the Washout and Follow-up Period: Sensitivity Analysis Table 3.6.2

Analysis Set: Safety Analysis Set

Notes to Programmer: Same as Table 3.2.1, however, SAEs that occur during the Washout or Follow-up periods are attributed to the treatment given in the preceding Treatment Period. Add the following footnote: "SAEs that occur during the Washout or Follow-up periods are attributed to the treatment given in the preceding Treatment Period." 

| 3.7.1 Listing of Serious Adverse Events | s) | |
|-----------------------------------------|-------------|---|
| 3.7.1 Listing of Serious Adverse E | (SAEs) | |
| 3.7.1 Listing of Serious Adve | Events | |
| 3.7.1 Listing of S | rdve | 7 |
| 3.7.1 Listing of | | |
| able $3.7.1$ Liv | $_{\rm of}$ | |
| able 3.7.1 | Ë | |
| <u>~</u> | able | • |

| Study | / Action/ Day | - (Outcome) Resolved | (AE Treated) [a] |
|-----------|---------------|-------------------------|-------------------|
| | Severity/ | Relation- | ship |
| | Duration | t of Event | (c] |
| Onset Day | [q] | (Day of Most of Event R | Recent Dose) |
| | Treat. | Emerg. | [p] |
| | | Reason for Being | Serious (Day) [a] |
| | | SAE Verbatim | (Preferred Term) |
| | Primary | System Organ | Class |
| Age | (yrs)/ | Gender/ | Race |
| | | Subject | ΠD |

90 µg Proventil 180 µg, or Proventil Treatment: AS MDI 180 µg, AS MDI 90 µg, Placebo,

# Center # (Investigator): Center ### (xxxxxxxxx)

| 8 X H | | | | | | | | | | | | | | | 7 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| / None | (Recovered/Re | solved) | (Yes) | | Drug | Interrupted, | Date Stopped: | YYYY-12-07; | AE abated: | Yes; Date | restarted: | YYYY 12 08: | AE reoccur? | Yes | 0,000 T 0.7.7.000 Y |
| Moderate / None | Not | Related | | | | | | | | | | | | | of +0 vo neite |
| 5 | (T2_P1) | | | | | | | | | | | | | | MeH exiteN=THN |
| Yes | | | | | | | | | | | | | | | Zmor: |
| Hospitalization / | prolongation of | existing | Hospitalization | (T1 1-Tx y) | | | | | | | | | | | B=Black or African |
| XXX XXX XXXX XXX XXX | (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | | | | | | | | | | | | MIAN-American Indian or Alacka Native B=Rlack or African American NHDI=Native Hawaiian or Other Dacific Islander |
| XX XXX XXX | XXXX | | | | | | | | | | | | | | TAN=American |
| XXXXXX 70/F/W | | | | | | | | | | | | | | | |
| XXXXXX | | | | | | | | | | | | | | | ae:84=4 .00ed |

Race: A-Asian, AIAN-American Indian or Alaska Native, B-Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, O=Other W=White. Gender: F=Female, M=Male.

- A negative number for study day denotes the number of days prior to the start of study treatment. Otherwise, Study Day is Date Date of dose in the Period + 1. Tx = Period.  $Tx_y = Period$  and Day within Period. Pxx = Days after dose in the last Tx = Period. g
- On Study Day 1, an 0 indicates that event started before study drug administration. On Study Day 1, 00 indicates that event started after study drug administration. # indicates that it could not be determined whether the AE had onset during study treatment. [O]
  - Duration of Event = Stop Day Onset Day + 1

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/t030801.sas Version YYYY-MM-DD xx:xx Notes to Programmer:

Sort by Actual Treatment, Center, Subject ID, Primary System Organ Class Preferred Term, and Onset Day.

If Reason for Seriousness is Hospitalization or Prolongation of Existing Hospitalization, also present in parentheses the days subject admitted into and discharged from Hospital "(Day xx - Day xx)".

If the Reason for Seriousness is death, also present the day of death.


Table 3.7.2 Listing of SAE-Specific Report Information Analysis Set: Screened

| .p/<br>SAE<br>)) Treated | Yes/No |
|---|---|
| Severity/<br>Relationship/<br>(Outcome)<br>(YYYY-MM-DD) | Moderate / Related / (Recovered/Resolved) (2015-07-27) |
| Action Taken With<br>Study Drug | None Drug Interrupted (Stopped: YYYY-MM-DD SAE Abated: Yes/No Treatment Restarted: YYYY-MM-DD SAE Reoccur: Yes/no) Permanently Withdrawn (YYYY-MM-DD) |
| Serious Reason<br>(YYYY-MM-DD) | Death (YYYY-MM-DD) None Autopsy: yes or no Life-threatening (Sto) SAE Hospitalization or Trearisting hospitalization or Trearisting hospitalization (YYYY-MM-DD-YYYY- Perm MM-DD) A persistent or significant disability/incapac ity Congenital A significant defect A significant medical event that medical event that requires medical or surgical intervention to prevent one of the serious outcomes |
| Date of SAE Onset (YYYY-MM-DD) And Most Last Recent Dose Treatment and of Treatment Date Prior to (YYYY-MM-DD) Onset of SAE | 15-07-28 2015-07-24 YYYY-MM-DD |
| Diagnosis, Details and<br>Relevant Diagnostic Tests | Treatment: AS MDI 180 µg, AS MDI 90 µg, Placek Center # / (Investigator): ### / (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| Subject ID | Treatment: |

Notes to Programmer: Sort by Center, Subject ID, and Onset Day of SAE. Move 'Center' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header. In order for the SAE-Specific Report Information to be listed, it will need to be included in the SDTM data sets.

13 Mar 2018 

Table 3.8 Treatment Related Serious Adverse Events by MedDRA Primary System Organ Class and Preferred Term Analysis Set: Safety Analysis Set

[a] Related = Yes or No.

Notes to Programmer: Same as Table 3.2.1.


TEAEs by Primary System Organ Class, Preferred Term, and Highest Severity - Placebo Analysis Set: Safety Analysis Set Table 3.9.1

| | | LACADO (N-XXX) | (VVV_N) | |
|---|---|---|---|---|
| Primary System Organ Class<br>Preferred Term | Mild<br>n (%) | Moderate<br>n (%) | Severe n (%) | Any Severity n (%) |
| At Least One TEAE | (xxxx) xxx | xxx (xxx.x) | xxx (xxx.x) | xxx (xxxxxx) |
| System Organ Class 1 | xxx (xxx.x) | xxx (xxxx.x) | (xxxxx) xxx | (xxxxx) |
| Preferred Term 1 | (xxxx) xxx | xxx (xxx.x) | xxx (xxx.x) | (x.xx.x) |
| Preferred Term 2 | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | (xxxx.x) |
| System Organ Class 2 | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | (xxxx.x) |
| Preferred Term 1 | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) | xxx (xxx.x) |
| Preferred Term 2 | (x.xxx) xxx | xxx (xxxx.x) | (xxxxx) xxx | (xxxx.x) |

TEAEs by Primary System Organ Class, Preferred Term, and Highest Severity - AS MDI 90 µg Analysis Set: Safety Analysis Set Table 3.9.2

TEAEs by Primary System Organ Class, Preferred Term, and Highest Severity – AS MDI 180 µg Analysis Set: Safety Analysis Set Table 3.9.3

TEAEs by Primary System Organ Class, Preferred Term, and Highest Severity - Proventil 90 µg Analysis Set: Safety Analysis Set Table 3.9.4

TEAEs by Primary System Organ Class, Preferred Term, and Highest Severity - Proventil 180 µg Analysis Set: Safety Analysis Set Table 3.9.5


Analysis Set: All Subjects Screened Listing of Deaths Table 3.10

| Subject ID | Treatment<br>Sequence | Days<br>Study Day of Dose of Last Trea <sup>*</sup><br>Treatment Prior to Death [a] ment | Days on<br>Treat-<br>ment | Date and Time (YYYY-MM-DD) (24 h clock) of Death | Days Since<br>Dose<br>at Time of<br>Death [b] | Adverse Event Preferred<br>Term/Verbatim Term |
|---|---|---|---|---|---|---|
| Study Center | # / (Investiga | Study Center # / (Investigator): ### / (xxxxxxxxx) | | | | |
| ×××× | ×/× | TRT A<br>Day x<br>(vvvvv/mm-ma) | Н | YYYY-MM-DD<br>hh:mm | × | Preferred Term/AE verbatim |

Treatment: A = Placebo, B = AS MDI 90  $\mu$ g, C = AS MDI 180  $\mu$ g, D = Proventil 90  $\mu$ g, E = Proventil 180  $\mu$ g, - = Not Treated. This includes all subjects who died while on study and  $\mu$ g to 30 Days after final treatment dose.

Study Day of Dose for Treatment = Study Day 1. Days since Last Dose = Date of death - Date of last dose of study treatment  $\pm$  1. TRT = Treatment.
[a] Study Day of
[b] Days since Let

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/t0313.sas Version YYYY-MM-DD xx:xx

Notes to Programmer: For TRTN, N is the treatment period number of the last treatment received by the subject prior to the death.

Sort by Study Center and Subject within Study Center. Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header. 

#### Vital Signs

Vital Sign Parameters Analysis Set: Safety Analysis Set Table 3.11.1

| | | | | AS MDI | AS MDI | Proventil | Proventil |
|---|---|---|---|---|---|---|---|
| | | | Placebo | 90 pd | 180 µg | 90 pd | 180 µg |
| Parameter (unit) | Visit/Timepoint | Statistic | (N=XXX) | (N=xxx) | (N=XXX) | (N=xxx) | (N=xxx) |
| Daramotor 1 (1111;+) | (1 + i = i11) | . o Le. 1 77 Le. 1+0 € | | | | | |
| raimeret 1 (unitr) | OCTUBLITION (ATRICE T) | Accual value. | | | | | |
| | | п | XXX | XXX | XXX | XXX | XXX |
| | | Mean | x.xxx | x.xxx | x.xxx | x.xx.x | x.xx |
| | | SD | x.xxx | x.xxx | x.xxx | x.xx.x | x.xx |
| | | Median | X.XXX | XXX.X | XXXX.X | X.XX.X | X.XXX |
| | | Minimum | x.xx | x.xx | x.xx | xx.x | x.xx |
| | | Maximum | × × × | ×× | ××.× | × × × | ××.× |
| | Baseline (Visit 2 | Actual Value: | | | | | |
| | Pre-Dose) | п | XXX | XXX | XXX | XXX | XXX |
| | | Mean | X.XXX | XXXX.X | XXX.X | XXXX.X | XXXX.X |
| | | SD | X.XXX | XXXX.X | XXX.X | XXXX.X | XXXX.X |
| | | Median | ×.xxx | XXX.X | XXX.X | x.xx.x | XXXX.X |
| | | Minimum | ××.× | xx.x | ××××× | ××.× | XX.X |
| | | Maximum | ×. × | ×× | ×. ×. | × × × × | ×.×. |
| | | Change From Baseline: | | | | | |
| | | п | XXX | XXX | XXX | XXX | XXX |
| | | Mean | X.XXX | XXXX.X | × ×××× | ×.xxx | ×.xxx |
| | | SD | x.xxx | xxx.x | x.xxx | x.xx.x | x.xx |
| | | Median | x.xxx | x.xxx | x.xxx | x.xx.x | x.xx |
| | | Minimum | ××.× | ×.xx | ×.xx | ××.× | ××.× |
| | | Maximum | x.xx | x.xx | x.xx | x.xx | x.xx |
| For parameters Height, Weight, | ht, Weight, and BMI, c | and BMI, only include Screening. | For SPB, DBP, | and Heart Rate | include Scree | For SPB, DBP, and Heart Rate include Screening, Baseline (Visit 2 Pre- | (Visit 2 Pre- |
| Dose), Visit 2 (Pos | t-Dose), Visit 3 (Pre- | C) | e), Visit 4 (H | re-Dose), Visi | t 4 (Post-Dose | ), Visit 5 (Pre | -Dose), Visit |

5 (Post-Dose), Visit 6 (Pre-Dose), Visit 6 (Post-Dose), and End of Treatment.

Baseline is defined as the last pre-dose measurement taken prior to dosing on Day 1 of a treatment period.

End of Treatment is defined as the last non-missing on treatment assessment available for the timepoint.

Report generated by program: PT007001/sasdir/programs/statout/t031101.sas Version YYYY-MM-DD xx:xx

(Page n of N)

Notes to Programmer:

Repeat the parameter at the beginning of each page under column header. Repeat for all parameters.


#### 13 Mg

### 4. Subject Data Listings

# 4.1 Subject Discontinuations/Completions

Listing 1.1 Study Centers Analysis Set: All Subjects Screened

| Center | Investigator | Location |
|---|---|---|
| XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxxxxxxx City Country |
| XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxxxxxxxxxxxx City Country |
| XXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xxxxxxxxxxxxxx City Country |
| Source: xxxxxxx.sas7bdat | | |

Report generated by program: /sasdir/programs/statout/10101.sas

(Page n of N)

YYYY-MM-DD xx:xx

Version


Subject Disposition and Demographic Data Analysis Set: All Subjects Screened Listing 1.2

| | | | | 51 | Smoking History | istory | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Age<br>(vrs)[al/ | | | Number<br>of<br>Weeks | Number | Average<br>Number of | Number<br>of Pack | | Subject Study Status<br>(Date of Last Dose<br>[Study Day) } |
| Subject ID<br>(Treatment<br>Sequence) | Gender<br>(Race/Eth<br>nicity) | Height(cm)/<br>Weight (kg)/<br>BMI (kg/m²) | Smoking<br>Status<br>[b] | Since<br>Day<br>Quit | of<br>Years<br>Smoked | Cigarettes<br>Smoked Per<br>Day | Years<br>Smoked<br>[c] | Randomized?<br>(Study Day)<br>[d] | (Follow-up, Call? Date) Date of Death [e] |
| <pre>Center # (Investigator): Center ### (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx</pre> | igator): Cent | ter ### (xxxxxx | (XXXX) | | | | | | |
| XXXXXX<br>(A/B/E/C/D) | (xx/x) | xxx.x/<br>xx.x/<br>xx.x | Former<br>Smoker | x | × | × | × | Yes/No<br>(xx) | Completed Study (YYYY-MM-DD [xxx]) (Yes YYYY-DD-MM) |
| XXXXXX<br>(A/E/-/-) | M/xx<br>M/xx) | /xxx<br>/xx/<br>xx.xx | Former<br>Smoker | × | × | ×× | ×× | Yes/No (xx) | Discontinued Investigator's Decision (YYYY-MM-DD [Tx_y]) |
| Xxxxxx<br>(B/A/C/E/-) | (xx/x)<br>M/xX | xxx.x/<br>xxx.x/<br>xx.xx | Former<br>Smoker | ×<br>×<br>× | × | × | ×<br>×<br>× | Yes/No (xx) | Discontinued Subject Lost to Follow up (YYYY-MM-DD [Tx_Y]) |
| XXXXXX<br>(B/C/-/-/-) | (xx/x) | xxx.x/<br>xx.x/<br>xx.x | Non<br>Smoker | x | × | × | ×<br>×<br>× | No<br>(NA) | Discontinued Investigator's Decision (YYYY-MM-DD [Tx_Y]) |
| Xxxxxx $Xx/M$ $xxx.x/$ $(A/B/E/C/D)$ $(x/xx)$ $xx.x/$ $xx.x/$ | M/xx<br>M/xx) | | Former<br>Smoker | × × × | × | Former xx.x xx x | XX.X NO (NA) | | Discontinued Adverse Event (YYYY-MM-DD [Tx_y]) (No) Death: YYYY-MM-DD |

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated.

Race: A=Asian, AIAN=American Indian or Alaska Native, B=Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, O=Other W=White. Ethnicity: H=Hispanic, NH=Not Hispanic, UNK=Unknown, NR=Not Reported. Gender: F=Female, M=Male.

[a] Age = integer part of ((Visit 1 date - Birth date)/365.25)

[b] Former Smoker is defined as those who have stopped smoking for at least 6 months prior to first Screening Visit.


- Number of pack years smoked = (number of cigarettes per day / 20) x number of years smoked. @ g c
  - Study Day of randomization = date of randomization first dose of study treatment
- last contact for subjects lost-to-followup. For subjects not randomized, date of discontinuation Study Day is the last visit date date of Screening Visit 1; for treated subjects, Study Day is the date of discontinuation date of first dose of study The Date of Discontinuation is the later of the last visit date, the date of the last dose of study medication, or the date of treatment + 1.

Source: xxxxxxx.sas7bdat

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/10102.sas Version YYYY-MM-DD xx:xx

Notes to Programmer:

Sort by Center, and Subject ID within Center.

Last Contact Date on the End of Treatment CRF is date of last contact.

If Race = Other, concatenate the specified race after 'O' within parenthesis, e.g., "O (specified)".

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.
Listing 1.3 Randomized Treatment, Actual Treatment, and Duration of Treatment Analysis Set: All Subjects Randomized

| | | Period 1<br>Treatment | Period 2<br>Treatment | Period 3<br>Treatment | Period 4<br>Treatment | Period 5<br>Treatment | Study Day |
|---|---|---|---|---|---|---|---|
| zed<br>nt<br>e | (Start Stuand time - Study Day time)/ | dy Day<br>End<br>and | (Start Study Day and time - End Study Day and time)/ | Start Study Day<br>and time - End<br>Study Day and<br>time)/ | (Start Study Day and time - End Study Day and time)/ | (Start Study Day and time)/ | of First<br>and Last<br>Dose of<br>Study |
| (Actual Duration (days), Treatment Washout Length Subject ID Sequence) (days) [a] | O 1 | days)/ Dura | Duration (days)/ Washout Length (days) [a] | Duration (days)/<br>Washout Length<br>(days) [a] | Duration (days)/<br>Washout Length<br>(days) [a] | Duration (days)/<br>Washout Length<br>(days) [a] | treatment<br>in the<br>study |
| . ~ ~ ~ | . ~ ~ ~ | 00 hg / | AS MDI 90 µg (xxx hh:mm - xxx hh:mm)/ 25/ (7) | Placebo (xxx hh:mm - xxx hh:mm) / 25/ (7) | Proventil 180 µg<br>(xxx hh:mm -<br>xxx hh:mm)/<br>25/<br>(7) | Proventil 90 µg (xxx hh:mm - xxx hh:mm)/25/(7) | × |
| B/A/C/E/- Proventil 180 µg (B/A/C/E/-) (xxx hh:mm - xxx hh:mm)/ 29/ (7) | Proventil 18<br>(xxx hh:mm -<br>xxx hh:mm)/<br>29/<br>(7) | бп<br>0 | AS MDI 180 µg<br>(xxx hh:mm -<br>xxx hh:mm)/<br>25/<br>(7) | Proventil 90 µg<br>(xxx hh:mm -<br>xxx hh:mm)/<br>25/<br>(7) | Placebo<br>(xxx hh:mm -<br>xxx hh:mm)/<br>25/<br>(7) | | ×××<br>-<br>××× |
| A/B/E/C/D AS MDI 90 µg (A/E/-/-) (xxx hh:mm - xxx hh:mm)/ 25/ | | pu | Placebo (xxx hh:mm - xxx hh:mm)/25/ | | | | XXX - XXX |

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. Study Day of First Dose of Drug in the study is defined as the study day of the first dose of study medication in the study (Study Day 1) which is the study day of Treatment 1 Day 1 from the Study Drug Administration CRF. Study Dose of Study Drug in the study is defined as the Study Day of the Last Dose of Study Drug in the study is defined as the Study Day of the last dose of study medication in the study Study Day of first dose of study medication in the study + 1. NA = not applicable

Time is 24 hour clock time.

[a] Washout length (days) for the subject's last period is the number of days between the follow-up telephone call and the dose date in the last period. The duration of a washout (or follow-up) period = (start date of subsequent treatment (or follow-up telephone call) - stop date of previous study treatment.

Source: xxxxxxx.sas7bdat

Report generated by program: PT007001/sasdir/programs/statout/10103.sas Version YYYY-MM-DD xx:

Notes to Programmer: Sort by Center and Subject within Center. Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


Listing 1.4 Reasons Subjects Were Not Randomized
Analysis Set: All Subjects Not Randomized

| | | | | | | | : Islander, | | |
|---|---|---|---|---|---|---|---|---|---|
| | | hn) | (1 | (1 | (1 | (1 | ther Pacifi | | ſ |
| 7 | | xxxxxxxxxxxxx (Inclusion Criterion #n) | xxxxxxxxxxx (Inclusion Criterion #n) | xxxxxxxxxxx (Inclusion Criterion #n) | xxxxxxxxxxxx (Inclusion Criterion #n) | xxxxxxxxxxxx (Inclusion Criterion #n) | Race: A=Asian, AIAN=American Indian or Alaska Native, B=Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, O=Other W=White. | | |
| Randomizec | | :xxxx (Inc] | xxx (Inclu | xxx (Inclu | xxx (Inclu | xxx (Inclu | , NHPI=Nat. | | |
| Reason Not Randomized | | XXXXXXXXX | ××××××××× | XXXXXXXX | XXXXXXXX | XXXXXXXXX | American, | | |
| | | × | × | × | × | × | or African | | ( |
| Race | | M | W | M | M | M | B=Black o | | |
| Gender | (xxx) | Male | Female | Male | Male | Female | a Native, | | |
| Age<br>(yrs) | xxxxxxx) | × | × | ×× | ×× | ×× | or Alask | | 7 |
| Date of Screening | Center # (Investigator): Center ### (xxxxxxxxxxx | YYYY-MM-DD | YYYY-MM-DD | XXXX-MM-DD | XXXX-MM-DD | XXXX-MM-DD | =American Indian<br>:e. | 7bdat | |
| | Investigat | ХX | XX | XX | XX | XX | A=Asian, AIAN=Am<br>O=Other W=White. | xxxxx | |
| Subject ID | Center # ( | XXXXXX | ×××××× | XXXXXX | XXXXXX | XXXXXX | Race: A=As. | Source: xxxxxxx.sas7bdat | |

Notes to Programmer:

Sort by Center and Subject ID within Center.

If Race = Other ("O"), concatenate the specified race after 'O' within parenthesis, e.g., "e.g., "O: xxxxxx".

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header. If country is shown, move country to the next page if there is not enough room.


### 4.2 Protocol Deviations

Violation of Inclusion/Exclusion Criteria Analysis Set: All Subjects Randomized Listing 2

| | | | | | Eli | Eligibility | |
|---|---|---|---|---|---|---|---|
| | Age (yrs)/ | | Informed | | | Inclusion/ | |
| | Gender | Informed | Consent | | | Exclusion | Type of |
| Treatment | (Race) | Consent | Study Day | | Study Day | Criteria | Failed |
| Subject ID Sequence | [a] | Signed | [a] | Visit | [a] | Satisfied | Criteria |
| <pre>Center # (Investigator): Center ### (xxxxxxxxxx)</pre> | Center ### (xxx | (XXXXXXX) | | | | | |
| XXXXXX A/B/E/C/D | $M \times M$ | Yes | ××- | Visit 1 | XX- | No | Inclusion |
| | (BA) | | | | | | |
| Treatment: A = Placebo, B = AS MDI 90 µg, C = Dade: Alasian Alamanican Indian or Alaska | $B = AS MDI 90 \mu_0$ | ı | -80 µg, D = Pro | ventil 90 µg, E | AS MDI 180 ug, D = Proventil 90 ug, E = Proventil 180 ug, - = Not Treated. | <pre>ug, - = Not Treated.</pre> | eated. |
| Nace: A-Astan, Athar-American indian of Atasha na<br>O=Other W=White. Gender: F=Female, M=Male. | ender: F=Female, | _ | D-Drack Or Dri | TOUR DIRECTIONIL | WIII I-MACIVE MAME | Tail Of Ocher Fa | TOTETO TRIBUCE, |
| [a] A negative number for study day denotes | for study day de | the | er of days pri | or to the start | number of days prior to the start of study treatment. | nt. | |
| Source:xxxxxxx.sas7bdat | | | | | | | |
| Report generated by program: PT007001/sasdir/programs/statout/102.sas Version YYYY-MM-DD xx:xx | ram: PT007001/sa | sdir/programs/ | statout/102.sa/ | s Version YYYY- | MM-DD xx:xx | (Page n of N) | |

Notes to Programmer:

If Race = Other ("O"), concatenate the specified race after 'O' within parenthesis, e.g., "O (specified)".

Sort by Center, and Subject ID within Center.

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


# 4.3 Screening Lung Function and Reversibility

Listing 3 Screening Lung Function and Ventolin HFA Reversibility Analysis Set: All Subjects Randomized

| | Age Arrestme (1775) | 0 2 | | Time of | | Pre-Dose | še. | | | Post-Dose | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | subject Sequenc (Race) | (grs/<br>/Gender<br>(Race) | | HFA Dose<br>(24 h | | FVC | PEFR | | FVC | PEFR | Reversi- |
| OH OH | [a] | | Visit Effort Date | clock) | FEV1 (L) | (I) (I) | (L/min) | FEV1 (L) | (L) (L) | (L/min) | bility % |
| Center | # (Investig | ator): C | <pre>Center # (Investigator): Center ### (xxxxxxxxxx)</pre> | (XXXX) | | | | | | | |
| | A/B/E/C xx/x | ×/ | | ×× : ×× | xxx.x | ×××××××××××××××××××××××××××××××××××××× | xxx.xxx | x.xx | x.xx | XXX.XXX | |
| XXXXX | /D (x; | (xxx) 1 | YYYY-MM-DD | | | | | | | | |
| | | 1a | AYYY-MM-DD | ××:×× | ×××××× | ×.xxx | xxx.xxx | ×××××××××××××××××××××××××××××××××××××× | ×.xxx | xxx.xxx | ×.× |
| | | 1b | YYYY-MM-DD | | ×××××××××××××××××××××××××××××××××××××× | ×.xxx | XXX.XXX | ×.xxx | ×.xxx | XXX.XXX | ××. |
| | B/A/C/E xx/x | ×/ | | ××:×× | ×××××× | ×.xxx | xxx.xxx | ×××××××××××××××××××××××××××××××××××××× | ×.xxx | xxx.xxx | ×.× |
| XXXXX | (xxx) -/ | xx) 1 | AYYY-MM-DD | | | | | | | | |
| | A/B/E/C xx/x | ×/ | | | ×××××× | xxxxx | xxx.xxx | ×××××× | ×××××× | xxx.xxx | (V) XXX |
| XXXXX | /D (xxx) 1 | xx) 1 | XXXX-MM-DD | | | | | | | | |
| Treatme | nt: A = Pla | cebo, B | Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, | : = AS MDI 1 | 80 µg, D = | = Proventil 90 µg, | | E = Proventil 180 µg, | = - 'bd 081 | Not Treated. | |
| Race: A | =Asian, AIA | N=Americ. | Race: A-Asian, AIAN-American Indian or Alaska Native, B-Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, | ska Native, | B=Black or | : African Am | erican, NHPI= | Native Ha | awaiian or ( | Other Pacific | Islander, |
| 0 | =Other W=Wh. | ite. Gen | O=Other W=White. Gender: F=Female, M=Male. | -Male. | | | | | | | |
| NA = no | NA = not applicable. | . (1) | | | | | | | | | |
| Source: | Source: xxxxxxx.sas7bdat | s7bdat | | | | | | | | | |
| Report | generated b | y progra | Report generated by program: PT007001/sasdir/programs/statout/103.sas | .r/programs/ | statout/10 | | Version YYYY-MM-DD xx:xx | XX:XX Q | (Page n of N) | (N) | |

Notes to Programmer: Sort by Center, and Subject ID within Center. Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


### 4.4 Baseline Characteristics

Analysis Set: All Subjects Randomized Asthma Diagnosis Listing 4.1

| Subject ID Treatment Sequence Age (yrs)/Gender/Race [a] Date [s] Years Pri Center # (Investigator): Center ## (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | |
|---|---|---|---|---|---|
| (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | (yrs)/Gender/Race [a] | Date [s] | Years Prior to First Dose [b] |
| xx / Male/ xxxx | ** | | | | |
| A/B/E/C/D xx / Male/ xxxx | Jenicer # (Investigator). Center #: | | | | |
| | | XX / Mõ | ale/ xxxx | MM-XXXX | ×.× |
| xx / Female / xxxx YYYY-06* | | XX / Fe | _ | *90-XXX | ×. ×× |

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. Race: A-Asian, AIAN-American Indian or Alaska Native, B=Black or African American, NHPI=Native Hawaiian or Other Pacific Islander,

- O=Other W=White. Gender: F=Female, M=Male. [۵]
- Months Prior to First Dose When Asthma was First Diagnosed = (Date of First Dose of Study treatment in the study Date Asthma First Diagnosed)/30.4375. Day of Diagnosis was imputed for all subjects as the 1st of the month. Missing month of Date Asthma First Diagnosed was imputed as June, or the month in which  $1^{st}$  was the latest before informed consent date; '\*' indicates the month displayed was imputed. [9]

Source: xxxxxxx.sas7bdat

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/10401.sas Version YYYY-MM-DD xx:xx Notes to Programmer: Sort by Center and Subject ID within Center. Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header. 

Listing 4.2 Medical and Surgical History Analysis Set: All Subjects Randomized

| Age (yrs)/ Gender Subject Treatment (Race) Sequence [a] Category Center # (Investigator): Center ## (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
|---|
| <pre>CNS/Neurological xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx</pre> |
| Eyes/Ear/Nose/Thr xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. Race: A-Asian, AIAN=American Indian or Alaska Native, B=Black or African American, NHPI=Native Hawaiian or Other Pacific Islander,

(xxxx) /xxxxx

XXXXXXXXX

(xxxx)

 $\times \times \times$ 

xxxxxx B/A/C/E/-

XXX

XXXX-MM

οN

- Onset Day=Onset date of condition date of the first dose of study treatment. Day was imputed as  $^{1st}$  of the month. Missing month was imputed as June, or the month in which  $1^{st}$  was the latest before informed consent date; '\*' indicates the month O=Other W=White. Gender: F=Female, M=Male. displayed was imputed. [d
  - End Day=End date of condition date of the first dose of study treatment. Day was imputed as  $1^{st}$  of the month. Missing month was imputed as June, or the month in which  $1^{st}$  was the latest before informed consent date; '\*' indicates the month displayed was imputed. [0

Source: xxxxxxx.sas7bdat

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/10402.sas Version YYYY-MM-DD xx:xx

Notes to Programmer: Sort by Center, Subject ID, and Onset Day. Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header. 

Screening Reproductive Status and Pregnancy Test Results Analysis Set: All Subjects Randomized Listing 4.3

| a WOCBP, Was Pregnancy Test Test Visit Date Pregnancy Test Test [b] Visit 1 YYYY-MM-DD Not Done Visit 2 YYYY-MM-DD Serum Pregnancy xxx Posit | | | | | If Subject is | | | Pregnancy Test | Test | |
|---|---|---|---|---|---|---|---|---|---|---|
| Reproductive Test Visit Date Pregnancy Test [b] ## (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | (271) | Screening | a WOCBP, Was | | | | | |
| Performed? [a] Visit Date Pregnancy Test [b] Visit 1 YYYY-MM-DD Not Done NA NA Yes Visit 2 YYYY-MM-DD Serum Pregnancy xxx Posii | Subject | | /Gender | Reproductive | reginancy<br>Test | Visit | | Type of | Study Day of | |
| Visit 1 YYYY-MM-DD Not Done NA Yes Visit 2 YYYY-MM-DD Serum Pregnancy xxx Test | ID | Sequence | (Race) | Status | Performed? | [a] | Visit Date | Pregnancy Test | Test [b] | Result |
| A/B/E/C/D xx/F/(xxx Woman of Non- visit 1 YYYY-MM-DD Not Done NA Childbearing Potential (Non-WOCBP) B/A/C/E/- xx/F/(xxx Woman of x) Childbearing Serum Pregnancy xxx Childbearing Potential (WOCBP) | Center # | (Investigat | or): Center | ×××××××××××××××××××××××××××××××××××××× | | | | | | |
| B/A/C/E/- xx/F/(xxx Woman of Yes Visit 2 YYYY-MM-DD Serum Pregnancy xxx Childbearing Test Potential (WOCBP) | XXXXXX | A/B/E/C/D | xx/F/(xxx<br>x) | | | Visit 1 | YYYY-MM-DD | Not Done | NA | NA |
| | ×××××× | B/A/C/E/- | | | Yes | Visit 2 | YYYY-MM-DD | Serum Pregnancy<br>Test | ×<br>× | Positive |

A=Asian, AlAN=American indian or Alaska Native, B=Black or African American, NHPI= O=Other W=White. Gender: F=Female, M=Male. Pregnancy testing at Visit 2 was done prior to randomization. Study Day is defined as date of test - date of the first dose of study treatment. آ م

Source: xxxxxxx.sas7bdat

Report generated by program: PT007001/sasdir/programs/statout/10403.sas Version YYYY-MM-DD xx:xx

(Page n of N)

### Notes to Programmer:

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header. Sort by Center, Investigator, Subject ID within Center, Visit, and Study Day of Pregnancy Test. List female subjects only.


Listing 4.4 Prior, Concomitant, and Post-Treatment Asthma Medications Analysis Set: All Subjects Randomized

| | :/Post- | | | |
|---|---|---|---|---|
| | Frior/<br>Concomitant/Post-<br>Treatment | | Yes/Yes/No | Yes/Yes/No |
| . Day | stop<br>Day<br>[a] | | | |
| Study Day | begin<br>Day<br>[a] | | - 22 | -22 |
| | Duration<br>(Days) | | | |
| | Ongoi<br>ng | | Yes | Yes |
| | Stop Date (YYYY-MM-DD) | | | |
| | Begin Date<br>(YYYY-MM-DD) | (XX) | 2008-XX-XX | 2008-XX-XX |
| ť | Keason<br>for<br>Use | ××××××××) | Asthma<br>Exacer<br>bation<br># xxx | Other, |
| Dose/ | Unit/<br>Route/<br>Frequency | Center ### | 90/ MCG/<br>IH/ PRN | |
| | (Freierred<br>Term)<br>(ATC Term) | <pre>Center # (Investigator): Center ### (xxxxxxxxxx)</pre> | (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | |
| Subject<br>ID<br>(Treatm | ent<br>Sequenc<br>e) | Center # | 1001<br>(A/B/E/<br>C/D) | |

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated.

<speci

All Asthma-related medications taken within 30 days of Screening and while on study are listed.

All subjects were allowed sponsor provided Ventolin HFA, and Pulmicort if previously using regularly scheduled ICS or ICS/LABA, during the Screening period, and Atrovent and/or Pulmicort during the treatment period which were reported on the Concomitant Medications concomitant if they were reported as being taken at any point from the start of randomized study treatment to the last date of study treatment. Medications with an onset date on or after the last dose of study treatment were considered post-treatment medications. Medications were considered to be prior medications if taken prior to the start of study treatment. Medications were considered

XX = Unknown month or day.

A negative number for study day denotes the number of days prior to the start of study treatment. Pxx = Days after dose in last Treatment Period.

Sources: xxxxxxx.sas7bdat

YYYY-MM-DD xx:xx (Page n of Version Report generated by program: PT007001/sasdir/programs/statout/10404.sas

ê

### Notes to Programmer:

Sort by Center, Subject ID, Preferred Term, and Begin Date of Asthma medication. Show Anatomic and chemical portion of ATC code. Only medications with Reason for Use of Asthma on eCRF will be listed here. Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.

# Listing 4.5 Prior, Concomitant, and Post-Treatment Non-Asthma-Related Medications Analysis Set: All Subjects Randomized

Add the following footnote: All non-Asthma-related medications taken within 30 days of Screening and while on study are listed.


9.4.6 Suspect Drug Assessment for SAEs Analysis Set: All Subjects Randomized Listing 4.6

| | | | | Started | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Treatment/ | | | | | |
| | | | | Date of | | | | | |
| | | | | Most | | | | | |
| | | | | Recent | | | | | |
| | | | | Study | | | | | SAE Causally |
| | | | | Treatment/ | | | | | Related to This |
| | | | | Blinded or | | | | | Product/Does |
| | | | | Open/ | | | | | Principal |
| | | | | Treatment | | | | | Investigator |
| | | Additional | | at Onset | | | | | feel that SAE |
| | | Non-Study | Dose/ | of AE/Non- | | | | | may be related |
| Subject ID | SAE Verbatim Term/ | Medication | Unit/ | study drug | Begin Date/ | Con- | | Begin Day/ | to other |
| (Treatment | Preferred Term/ | at Onset of | Route/ | at onset | Stop Date | tin- | Duration | Stop Day | factor? |
| Sequence) | Onset Date | SAE | Frequency | of SAE | (XXXX-MM-DD) | uing | (Days) | [a] | (Specify) |

| (xxxxxxxxxx) |
|--------------|
| ### |
| Center |
| r): |
| restigato |
| estigat |

| Yes / Yes (Pre-existing /Underlying disease or Prior or Concomitant Medication | No |
|---|---|
| -22 | T1_P1/<br>T1_P5 |
| | Ŋ |
| K<br>⊕<br>S | ON |
| 2008-xx-xx | 2008-XX-XX/<br>2008-XX-XX |
| Yes/<br>YYYY-MM-<br>DD/Blinded<br>or Open-<br>Label/<br>Yes/Yes | No |
| 90/µg/<br>IH/PRN | 34/µg/<br>IH/QID |
| Ventolin<br>HFA | Atrovent<br>HFA |
| XXXXXXXXXXXXX/XXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXX/<br>XXXXXXXXX/<br>YYYY-MM-DD |
| xxxx<br>(A/B/E/C/D) | XXXX<br>(B/A/C/E/-) |

Treatment: A = Placebo, B = AS MDI 90  $\mu g$ , C = AS MDI 180  $\mu g$ , D = Proventil 90  $\mu g$ , E = Proventil 180  $\mu g$ , - = Not Treated.

XX = Unknown month or day.

[a] A negative number for study day denotes the number of days prior to the start of study treatment. Otherwise, Study Day is Date - Date of dose in the Period + 1.  $Tx_y$  = Treatment Period and Day within Treatment Pxx = Days after dose in last Treatment Period.

(Page x of y) YYYY-MM-DD xx:xx Sources: xxxxx.sas7bdat
Report generated by program: PT007001/sasdir/programs/statout/10407.sas Version Notes to Programmer: for last column, 2nd question, "Does Principal Investigator feel that SAE may be related to other factor? (Specify)") is only listed on first line for each subject. 

#### 4.5 Dosing

Listing 5.1.1 Study Drug Administration Analysis Set: All Subjects Randomized

| Subject ID | Treatment Sequence | Study Visit Admini (Study Day [a]) Visit | Study Drug<br>Administered at<br>Visit | Date and Time of<br>On-Site Study Dose<br>(Study Day [a]) | Study Medication Component ID |
|---|---|---|---|---|---|
| Study Center # / | Study Center # / (Investigator): ### (xxxxx | (XXXXX) | | | |
| ××××× | A/E/-/- | Visit x $(Tx_y)$ | Yes | YYYY-MM-DD (hh:mm) | Bxxxxx |
| | | Visit $x$ ( $Tx_y$ ) | Yes | $YYYY-MM-DD$ (hh:mm) (Tx_Y) | BXXXXX |

Treatment: A = Placebo, B = AS MDI 90  $\mu g$ , C = AS MDI 180  $\mu g$ , D = Proventil 90  $\mu g$ , E = Proventil 180  $\mu g$ , - = Not Treated. [a] Study Day is Date - Date of dose in the Period + 1. Tx = Period. Tx\_y = Period and Day within Period. Pxx=Days after last dose in the last Treatment Period.

Source: xxxxxxx.sas7bdat

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/1050101.sas Version YYYY-MM-DD xx:xx

### Notes to Programmer:

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header. Sort by Center, Subject within Center, Date Dispensed, and Component ID.


Ventolin HFA and Pulmicort Flexhaler Dispensing Analysis Set: All Subjects Randomized Listing 5.1.2

| Subject ID | Treatment Sequence Drug | Drug | Dispensed | Date Dispensed | Study Day [a]<br>of Dispensing | Study Medication Component ID |
|---|---|---|---|---|---|---|
| Study Center # | Study Center # / (Investigator): ### (xxxxxxxxxx | (************************************* | | | | |
| ××××× | A/E/-/- | Ventolin HFA | Yes | YYYY-MM-DD | TXY | Axxxxx |
| | | Pulmicort<br>Flexhaler | Yes | YYYY-MM-DD | $\mathbb{T}^{\times}$ _Y | Axxxxx |
| | | Ventolin HFA | Yes | YYYY-MM-DD | TXY | Axxxxx |
| Treatment: A = [a] Study De last dos | <pre>Treatment: A = Placebo, B = AS MDI 90 ug, [a] Study Day is Date - Date of dose in last dose in Period.</pre> | · . | 180 µg, D =<br>+ 1. Tx = Pe | C = AS MDI 180 $\mu g$ , D = Proventil 90 $\mu g$ , E = Proventil 180 $\mu g$ , - = Not Treated the Period + 1. Tx = Period. Tx_y = Period and Day within Period. Pxx = Days $\epsilon$ | = Proventil 180 µg,<br>and Day within Per | C = AS MDI 180 $\mu g$ , D = Proventil 90 $\mu g$ , E = Proventil 180 $\mu g$ , - = Not Treated. the Period + 1. Tx = Period. Tx_y = Period and Day within Period. Pxx = Days after |
| Source: xxxxxxx.sas7bdat | <pre>«x.sas7bdat</pre> | ; | | | | |

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/1050102.sas Version YYYY-MM-DD xx:xx

### Notes to Programmer:

Sort by Center, Subject within Center, Date Dispensed, and Component ID.

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


Listing 5.2 Exposure to Study Treatment Analysis Set: Safety Analysis Set

| Number of Puffs | Expected | Taken [a] | | × × × × × | ; 2 11 22 11<br>; 2 12 12 12 |
|---|---|---|---|---|---|
| | Treatment | Period | | H 0 W 4 D | H 0/ W 4/ I |
| Age (yrs)/ | Gender | (Race) | (************************************* | xx/x (xxxx)<br>xx/x (xxxx)<br>xx/x (xxxx)<br>xx/x (xxxx)<br>xx/x (xxxx) | xxxx (xxxx) x/xx<br>xxxx (xxxx) x/xx<br>xxxx (xxxx) x/xx |
| | Subject ID | (Treatment Sequence) | <pre>Center # / (Investigator):</pre> | 1001 x<br>(A/B/E/C/D) x<br>x x | 1002 × (A/B/E/C/D) × |

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated.

Race: A-Asian, AIAN-American Indian or Alaska Native, B-Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, O=Other W=White. Gender: F=Female, M=Male.

[a] The expected number of puffs for each treatment day were as follows:

- AS MDI 90 µg (2 actuations of 45 µg/actuation)
- AS MDI 180 µg (2 actuations of 90 µg/actuation)
  - Placebo MDI (2 actuations)
- Proventil 90 µg (1 actuation of 90 µg/actuation)
- Proventil 180 µg (2 actuations of 90 µg/actuation)

Source: xxxxxxx.sas7bdat

Version YYYY-MM-DD xx:xx Report generated by program: PT007001/sasdir/programs/statout/10502.sas (Page n of N)

#### Notes to Programmer:

Sort by Center, Subject within Center, and Treatment Period. Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header. Treatment is actual treatment. 

### 4.6 Individual Efficacy Data

#### 4.6.1 Efficacy

Subjects Who Failed Restrictions Prior to Spirometry Assessment Analysis Set: All Subjects Randomized Listing 6.1

| | | | | | | Prior to Study V | Prior to Study Visit, Subject has |
|---|---|---|---|---|---|---|---|
| | | | | | | Not Had Xanthine | Withheld Asthma<br>Medications Including |
| Subject<br>ID | Treatment<br>Seguence | Visit | Study Time Window of<br>Assessment | Effort<br>Date | Effort Time<br>(24 h clock) | Containing Products<br>for at Least 6 Hours | Corticosteroids for at Least 6 Hours |
| Center # | (Investigator | ): Center ## | Center # (Investigator): Center ### (xxxxxxxxx) | | | | |
| XXXXXX | A/B/E/C/D Day 1 | Day 1 | Pre-Dose<br>60 Min | YYYY-MM-DD | 8:14:57 | No | |
| Treatment<br>Note that | Treatment: A = Placebo, B = AS MDI 90 $\mu g$ , C = Note that subjects with missing data for either | , B = AS MDI<br>h missing da | Treatment: A = Placebo, B = AS MDI 90 $\mu g$ , C = AS MDI 180 $\mu g$ , D = Proventil 90 $\mu g$ , E = Note that subjects with missing data for either of the 2 restrictions are also listed. | , D = Proventil<br>strictions are | l 90 µg, E = Pr<br>also listed. | AS MDI 180 $\mu g$ , D = Proventil 90 $\mu g$ , E = Proventil 180 $\mu g$ , - = Not Treated: r of the 2 restrictions are also listed. | Ireated. |
| Source: x | Source: xxxxxxx.sas7bdat | lat | | | | | |
| Report ge | Report generated by program: PT007001/sasdir/ | ogram: PT007 | '001/sasdir/programs/statout/10601.sas | ut/10601.sas | Version YYYY | YYYY-MM-DD xx:xx | (Page n of N |

Notes to Programmer: Sort by Center, Subject ID, and Effort Date.

Only subjects with 'No' or missing responses should be listed. Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


Failure of Stability Criteria Analysis Set: All Subjects Randomized Listing 6.2

| Subject ID<br>(Treatment Sequence) | Treatment | Visit | (Date of Spirometry Assessment) | try Assessment) |
|---|---|---|---|---|
| Study Center # / (Invest | Study Center # / (Investigator): ### (xxxxxxxxx) | | | |
| XXXXXX (A/B/E/C/D) | AS MDI 90 µg | Visit xx | XXXX-MM-DD | |
| | | Visit xx | TYYYY-DD | |
| XXXXXX (B/C/-/-) | Proventil 180 µg | Visit xx | YYYY-MM-DD | |
| Treatment: A = Placebo, B = AS MDI 90 µg, C | П | AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. | = Proventil 180 µg, - = | : Not Treated. |
| Source: xxxxxxx.sas7bdat | | | | |
| Report generated by proc | Report generated by program: PT007001/sasdir/programs/statout/10602.sas Version YYYY-MM-DD xx:xx | atout/10602.sas Version Y | YYY-MM-DD xx:xx | (Page n of N) |

Notes to Programmer: Sort by Center,Subject ID within Center, and Visit. Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


Listing 6.3 Reason for Missed Visit Analysis Set: All Subjects Randomized

| Subject ID<br>(Treatment Sequence) | Treatment | Visit Missed | Missed Due to | Missed Due to Asthma Related Issues | |
|---|---|---|---|---|---|
| Study Center # / (Inves | Study Center # / (Investigator): ### (xxxxxxxxx | (X) | | | |
| XXXXXX (A/B/E/C/D) | AS MDI 90 µg | Visit xx | Yes | | |
| Xxxxxx (B/C/-/-) | Proventil 180 µg | Visit xx | No | | |
| | | Visit xx | Unknown | | |
| Treatment: A = Placebo, B = AS MDI 90 µg, | | MDI 180 µg, D = P | roventil 90 µg, | C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. | Not Treated. |
| Source: xxxxxxx.sas7bdat | T | | | | |
| Report generated by pro | Report generated by program: PT007001/sasdir/programs/statout/10603.sas Version YYYY-MM-DD xx:xx | grams/statout/1060 | 3.sas Version | YYYY-MM-DD xx:xx | (Page n of N) |

Notes to Programmer: Sort by Center, Subject ID within Center, and Visit.

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


Spirometry Measurements Analysis Set: All Subjects Randomized Listing 6.4

| | | | | | | H | _ |
|---|---|---|---|---|---|---|---|
| | | | | | | PEFT | (ms) |
| | | [ور | ( é | | | PEFR | (L/Min) |
| Spirometry Assessments | (1) | [Predicted Value at Screening] | Percent of Predicted Value) | 0] | FEF | 25-75 | (T/sec) |
| ry Asse | Raw Value | alue at | Predic | (grade) [b] | | $FEV_1/$ | FVC (%) |
| iromet | R | cted V | ent of | (g) | | | /C (I) |
| Š | | [Predi | (Perc | | | FEV6 | L) F |
| | | | | | | 된 | ( |
| | | | | | | | FEV1 (L |
| | Nominal Time | )f | Assessment | (Actual Time | Jo | Assessment | 24 h clock) $FEV_1$ (L) (L) $FVC$ (L) $FVC$ (%) (L/sec) |
| | Z | 0 | I | Rescue | Ventolin ( | HFA used? A | (Time) |
| | | | | | | | ۵] |
| | | | | | Assessment | Date (Study | Day) [a] |
| | | | | Treatment/ | Treatment | Date/Time | (24 h clock) |
| | | | | | | | Visit |
| | | Age | (Yrs)/ | reatme Gender/ | Race/ | equence Height | (cm) |
| | | Subject Age | ID | (Treatm | nt | Sequenc | _ |

## Center # (Investigator): Center ### (xxxxxxxxx)

| Xxxxxx 53/F/W/xx Visit 1 | visit 1 | XXXY-MM-DD | NA | 60 Min Pre- | ×××××× | ××××× | ×××××××××××××××××××××××××××××××××××××× | ××× | ×××××× | xxx.xxx | ×× |
|---|---|---|---|---|---|---|---|---|---|---|---|
| (A/B/E/Cx | | (××-) | XX:XX) | Dose (xx:xx) | [x.xxx] | | [x.xxx] | | [x.xxx] | [xxx.xxx] | |
| /D) | | | AM/PM) | | (XX.X%) | | (XX.XX) | | (xx.x%) | (××·××) | |
| | | | | | (×) | | (x) | | | (x, x) | |
| | Repeat for A/ | YYYY-MM-DD | Yes | 15 Min Post- | ×××××× | ×××××××××××××××××××××××××××××××××××××× | ×××××× | ××.× | ×××××× | XXX.XXX | XXX |
| | Visit 1a, YYYY-MM-DD/ | $(\mathbb{T} \times \mathbb{Y})$ | (XXXXXX) | | (××·×%) | | (××.×%) | | (××.×%) | (××.×%) | |
| | 1b, 2, 3, hh:mm | I | | | (×) | | (× | | | (× ,×) | |
| | 4, and 5 | | | | | | | | | | |
| | and any | | | | | | | | | | |
| | other | | | | | | | | | | |
| | 11,01,40 | | | | | | | | | | |

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. Race: A=Asian, AIAN=American Indian or Alaska Native, B=Black or African American, NHPI=Native Hawaiian or Other Pacific Islander,

O=Other W=White. Gender: F=Female, M=Male.

- Study Day is Date Date of dose in the Period + 1. Tx = Period.  $Tx_y = Period$  and Day within Period. Pxx = Days after dose in last Treatment Period. Grade is coded: 1=Acceptable 2=Borderline Acceptable 3=Unacceptable. NA = Not applicable.
  - [9]

Version YYYY-MM-DD xx:xx Report generated by program: PT007001/sasdir/programs/statout/10604.sas Source: xxxxxxx.sas7bdat

(Page n of N)

Notes to Programmer:

Sort by Center, Subject ID, Assessment Date, and Nominal Time of Assessment.

Show Predicted Value only for Screening Visits.

Nominal time of assessment is the SAP-specified derived time window.

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


Listing 6.5 Spirometry Derived Endpoints Analysis Set: All Subjects Randomized

| | | | | | | Spirometr | Spirometry Derived Endpoints | Indpoints | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Achieved<br>Improvement<br>in FEV <sub>1</sub> from<br>Baseline | | Time to | | |
| Subject Age<br>ID (yrs)/<br>(Treatme Gender/ | Assessment | Ť. | Change<br>from | Change<br>from | Peak<br>change<br>from | Change<br>from | ' | Within 30<br>Minutes of<br>Dose | | Onset of<br>Response<br>(minutes) | Duration of<br>Response<br>(minutes) | se se ss) |
| nt Race/<br>Sequence Height<br>) (cm) Visit | Date<br>(Study<br>Visit Day) [a] | Timepoint | Baseline<br>in FEV <sub>1</sub><br>AUC <sub>0-6</sub> | Baseline<br>in FEV <sub>1</sub><br>AUC <sub>0-4</sub> | baseline<br>in FEV <sub>1</sub><br>(L) | baseline<br>in FEV <sub>1</sub><br>(L) | Time to<br>Peak FEV <sub>1</sub><br>(hours) | 12% 1.9 | 15% 12% | 15% | 12% | 15% |
| Center # (Investigator): Center ### (xxxxxxx | Center ### | (xxxxxxxxxx) | | | | | | | | | | |
| Xxxxxx 53/F/W/xx Visit 2 YYYY-MM-DD 60 Min (A/B/E/C x (Tx_Y) Pre-Do: | c 2 YYYY-MM-D<br>(Tx_Y) | D 60 Min<br>Pre-Dose | | | | ××× × | | | | | | |
| | Repeat YYYY-MM-DD 30 Min | D 30 Min | ×.xxx | ×.xxx | ×. xxx | ×.xxx | ××.× | Yes | No x.x | × × × | x.x x.x x.xx x.xx | ×× |

×××× ×××× ×××× Š N U ××× ××××× XXXXX ××××× ××××× 1a, 1b, 2, 3, 4, and 5 timepoin all pre-Repeat for and any include visits, postother Visit dose and and ts.

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. Race: A-Asian, AIAN-American Indian or Alaska Native, B-Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, O=Other W=White. Gender: F=Female, M=Male.

NA = Not applicable.

Study Day is Date - Date of dose in the Period + 1. Tx = Period.  $Tx_y = Period$  and Day within Period. Pxx = Days after dose in last Treatment Period.

Source: xxxxxxx.sas7bdat


(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/10605.sas Version YYYY-MM-DD xx:xx

Notes to Programmer:

Report FEV AUC<sub>0-6</sub> FEV AUC<sub>0-4</sub>, Peak change from baseline in FEV, and Time to Peak FEV, only at the last timepoint for each treatment period. Report Achieved 12% Improvement in FEVI from Baseline Within 30 Minutes of Dose, Achieved 15% Improvement in FEVI from Baseline Within 30 Minutes of Dose, Time to Onset of Response, and Duration of Response only at 30 minute post-dose timepoint.

Sort by Center, Subject ID, Assessment Date, and Timepoint.
Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


### 4.7 Adverse Event Listings

Adverse Events by Primary System Organ Class, Preferred Term, Treatment, Country, Center, Subject ID, and Onset Day Analysis Set: All Subjects Randomized Listing 7.1

Primary System Organ Class: xxxxxxxxxxxxxxxx

| Preferred Term | Treatmen | Center #<br>Treatment (Investigator) | Subject ID<br>(Treatment,<br>Sequence) | Age<br>(yrs)<br>/Gender<br>(Race) | Treatment Emergent / Serious | Onset Date (Day) [b] / Occur before or after start of a treatment On Day 1 | Duration<br>of<br>Event<br>[c] | Severity /<br>Relationship | Action<br>(Outcome)<br>(AE Treated) | Study Day Resolved /Death [b] |
|---|---|---|---|---|---|---|---|---|---|---|
| ××××××××××××××××××××××××××××××××××××××× | ******* | ### XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXX XX/F (A/B/E/C/D) (XXXX) | XX/F<br>(XXXX) | Yes / No | Yes / No YYYY-MM-DD (T1_P1) | × | Moderate /<br>Related | Not<br>Applicable (Re<br>covered/Resol<br>ved) (Yes) | T1_P5 |
| | | | | XX/F<br>(XXXX) | Yes / NO | Yes / No YYYY-MM-DD<br>(T2_P2) | × | Moderate/<br>Not Related | Drug<br>Interrupted(R<br>ecovering/Res<br>olving)g<br>(Yes) | |
| | ****** | (×××××××××) ### *********************** | XXXXXX<br>(A/B/E/C/D) | Xx/F<br>(xxxx) | Yes / | YYYY-MM-DD<br>(T1_P1) | ×× | /************************************* | Dose not<br>changed<br>(Recovered/Re<br>solved with<br>sequelae) (No) | T1_P7 |
| : | | (xxxxxxxx)<br>### | XXXXXX<br>(A/B/E/C/D) | XX/F<br>(XXXX) | Yes / No | Yes / No YYYY-MMDD (T2_P2) | × | / xxxxxxxx | Dose not<br>changed<br>(Recovered/Re<br>solved with<br>sequelae) (No) | |
| ************************************** | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | (×××××××)<br>### | XXXXXX<br>(A/B/E/C/D) | XX/F<br>(XXXX) | ON/ # | YYYY-MM-DD<br>(T1_P1) | ×× | / xxxxxxxx xx | Dose not<br>changed<br>(Recovered/Re<br>solved with<br>sequelae) (Yes<br>) | |
| | | | XXXXXX<br>(A/B/E/C/D) | Xx/F<br>(xxxx) | Yes / | YYYY-MM-DD<br>(T2_P2) | ×× | / xxxxxxxx<br>/ xxxxxxxxxxxxxxxxxxxxxxxxxx | Drug<br>withdrawn<br>(Recovering/R<br>esolving) | |


Race: A-Asian, AIAN-American Indian or Alaska Native, B-Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. O=Other W=White. Gender: F=Female, M=Male.

- # indicates that it could not be determined whether the AE had onset during study treatment. [a]
- Date of dose in the Period + 1. Tx = Period. Tx y = Period and Day within Period. Pxx = Days after dose in last Treatment Period. On Study Day 1, an @ indicates that event started before study drug administration. On Study Day 1, @@ indicates that event started after study drug administration. A negative number for study day denotes the number of days prior to the start of study treatment. Otherwise, Study Day is
  - Duration of Event = Stop Day Onset Day + 1. ပြ

Source: xxxx.sas7bdat

Report generated by program: PT007001/sasdir/programs/statout/10701.sas Version YYYY-MM-DD xx:xx

(Page n of N)

Notes to Programmer:

Put a blank line after each Center. Present the preferred term, treatment, center (investigator name). Subject ID (Actual Treatment and Age/gender/Race only if start a new value Sort by Primary System Organ Class, Preferred Term, Actual Treatment, Center, Subject ID within Center, and Onset Day. or at the first line of each page.

When a date of onset or date resolved is only partial, put full date in parenthesis under Study Day.

Move 'Study CentersInv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


Glossary of Adverse Event Preferred Terms vs. Investigator's Verbatim Listing 7.2

| MedDRA Advers | MedDRA Adverse Event Coding Dictionary | |
|---|---|---|
| Primary System Organ Class | Preferred Term | Investigator's AE Verbatim |
| ××××××××××××××××××××××××××××××××××××××× | ************************************** | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| ×××××× | ××××××××××××××××××××××××××××××××××××××× | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| MedDra Version xx.x was used for coding. | or coding. | |
| Source: xxxxxxx.sas7bdat | | |
| Report generated by program: PT | Report generated by program: PT007001/sasdir/programs/statout/10702.sas Version YYYY-MM-DD xx:xx | Version YYYY-MM-DD xx:xx (Page n of N) |

Notes to Programmer: Sort by Primary System Organ Class, Preferred Term, and Verbatim Term. List all unique investigators' AE verbatim.


Adverse Events by Treatment, Center, Subject ID, and Onset Day Analysis Set: All Subjects Randomized Listing 7.3

| | Day<br>Resolved/<br>Death [a] |
|---|---|
| | AE Day Relation Treated Outcome Resolved/ Severity -ship Action ? (Death?) Death [a] |
| | AE<br>Treate |
| | Action |
| | Relation<br>-ship |
| | Severity |
| | Event<br>Seriou<br>s |
| | Treat.<br>Emerg.<br>[b] |
| | AE Verbatim Treat. Event Duration<br>tem (Preferred Emerg. Seriou of Event<br>Term) [b] s [c] |
| | of a<br>treatment Primary System<br>On Day 1 Organ Class |
| Onset Date (Day) [a]/Occur before or after start | of a<br>treatment Primary Sys<br>On Day 1 Organ Class |
| Уде | (yrs)/<br>Gender<br>(Race) |
| | Subject ID<br>(Treatment<br>Sequence) |

Treatment: AS MDI

Center # (Investigator): Center ### (xxxxxxxxx)

| | | T1 P3 | | | | |
|---|---|---|---|---|---|---|
| Recoveri<br>ng/Resol | ving | Not | Recovere | d/Not | Resolved | 1 21/ |
| o<br>N | | Yes | | | | |
| Not Dose not<br>related changed | | Drug | Interrup | ted | | |
| Moderate Not<br>related | | Moderate Related | | | | |
| | | × | | | | |
| 0<br>N | | No | | | | |
| K<br>G<br>S | | No | | | | |
| AE 1<br>(xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | AE 2 | (XXXXXXXXXX) | | | |
| ×××× ××× ××× | | XXX XXX XXX | | | | |
| YYYY-MM-DD<br>(T1 P1) | I | YYYY-MM-DD | (T1 P1) | | | |
| XXXXX $XX/F$ $(A/B/E/C/D)$ $(XXXX)$ | | | | | | |
| XXX. | | | | | | |

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. Race: A-Asian, AIAN-American Indian or Alaska Native, B=Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, O=Other W=White. Gender: F=Female, M=Male.

- A negative number for study day denotes the number of days prior to the start of study treatment. Otherwise, Study Day is Date Date of dose in the Period + 1. Tx = Period. Tx\_y = Period and Day within Period. Pxx = Days after dose in the last Treatment [g
- On Study Day 1, an 0 indicates that event started before study drug administration. On Study Day 1, 00 indicates that event started after study drug administration.
- # indicates that it could not be determined whether the AE had onset during study treatment.
  - Duration of Event = Stop Day Onset Day + 1. [] []

Sources: adae.sas7bdat

Report generated by program: PT007001/sasdir/programs/statout/10703.sas Version YYYY-MM-DD xx:xx

(Page n of N)

Notes to Programmer:

Present the preferred term, latest treatment, center (investigator name), Subject ID, and Age/gender/Race when value changes start a new value or at the first line of each page Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header Sort by Actual Treatment, Center, Subject ID, Primary System Organ Class, Preferred Term, and Onset Day. Put a blank line after each subject. If Ongoing is ticked on CRF, show 'Ongoing' under Study Day Resolved.


### 4.8 Laboratory Values

Laboratory Test Results (Hematology Panel) Analysis Set: All Subjects Randomized Listing 8.1

| Flag<br>[b] | п/н | п/н |
|---|---|---|
| Reference<br>Range<br>Low-High | xxx-xxx | ××× |
| Assay<br>Value | ××× | ××× |
| Lab<br>Parameter<br>(Unit) | ××××××× | ××××××××××××××××××××××××××××××××××××××× |
| Lab Name | ×××××× | ×××××× |
| Nominal<br>Time of<br>Collection<br>(24 hr clock) | NA (hh:mm) | Post-<br>Treamtent Day<br>(hh:mm) |
| Collection Date (Study Day) [a] | XXXXXX) YYYY-MM-DD (-xx) | YYYY-MM-DD<br>(Tx_Py) |
| Visit<br>(Study Day [a]) | <pre>Center # (Investigator): Center ### (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx</pre> | Visit 6<br>(Tx_Py) |
| Age<br>(yrs)/<br>Gender<br>(Race) | <pre>Investigator):</pre> | |
| Subject ID<br>(Treatment<br>Sequence) | Center # (Ir<br>xxxxxx<br>(A/B/E/C/D | |

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. Race: A-Asian, AIAN-American Indian or Alaska Native, B-Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, O=Other W=White. Gender: F=Female, M=Male.

NA = Not Applicable.

- A negative number for study day denotes the number of days prior to the start of study treatment. Otherwise, Study Day is Date Date of dose in the Period + 1. Tx = Period.  $Tx_y = Period$  and Day within Period. Pxx = Days after dose in last Treatment Period. Pxx = Days after dose in last Treatment Period. Pxx = Days after dose in last Treatment Period. Pxx = Days after dose in last Treatment Period. [g
  - [p]

Source: adlb.sas7bdat

(Page n of Report generated by program: PT007001/sasdir/programs/statout/10801.sas Version YYYY-MM-DD xx:xx

2

Notes to Programmer:

Sort by Actual Treatment, Center, Subject ID, Date of Visit, Nominal Time of Collection, and Lab Parameter. Thus, show Screening Visit I before Visit I will not have a treatment time.

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.

Laboratory Test Results (Chemistry Panel and Kidney Function) Analysis Set: All Subjects Randomized Listing 8.2


Laboratory Test Comments Analysis Set: All Subjects Randomized Listing 8.3

| | | | Nom: nol | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Collection | Time of | | | | | | | |
| Subject ID | | Date | Collection | | | Lab | | Reference | | |
| (Treatment | Visit | (Study Day | (24 h | Lab | | Parameter | Assay | Range | Flag | Result |
| Sequence) | (Study Day [a]) | [a]) | clock) | Name | Lab Group | (Unit) | Value | Low-High | [q] | [b] Comments |
| | ı | | | | | | | | | |
| Center # (1 | Center # (Investigator): Center ### | XXXXXXX) | (xxx) | | | | | | | |

| XXXXXX | | | |
|-------------|--------------------|-----|---------|
| Ы | | | |
| 19-34 | | | |
| 18.000 | | | |
| Bicarbonate | (mmol/L) | | |
| Chemistry | | | |
| LabCorp | | | |
| Post- | Treatment | Day | (hh:mm) |
| YYYY-MM-DD | $(\mathbb{T}_{X})$ | | |
| Visit 6 | $(Tx_Py)$ | | |
| ίV | | | |

Race: A-Asian, AIAN-American Indian or Alaska Native, B-Black or African American, NHPI-Native Hawaiian or Other Pacific Islander, Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated.

O=Other W=White. Gender: F=Female, M=Male.

- A negative number for study day denotes the number of days prior to the start of study treatment. Otherwise, Study Day is Date Date of dose in the Period + 1. Tx = Period. Tx = Period and Day within Period. Pxx = Days after dose in last Treatment Period. N = Normal; L = Low; H = High; Abn. = Abnormal; L = Indeterminate. NA = Not Applicable. [a]

Source: adlb.sas7bdat

Report generated by program: PT007001/sasdir/programs/statout/10803.sas Version YYYY-MM-DD xx:xx

(Page n of N)

### Notes to Programmer:

Sort by Actual Treatment, Center, Subject ID, Date of Visit, Nominal Time of Collection, and Lab Parameter.

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.

Protocol D6930C00001 (PT007001)

# 4.9 Other Clinical Observations and Measurements

Vital Signs, Weight, and Height Analysis Set: All Subjects Randomized Listing 9.1

| BMI<br>(kg/m^2) | | ×. ×× | | xxx.x | | ; | ٧٠٧٧ | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Weight<br>(kg) | | ×××× | | x.xx | | ; | ٧٠٧٧ | | | | | | | |
| Height<br>(cm) | | ××× | | ××× | | | × × × | | | | | | | |
| Heart<br>Rate<br>(BPM) | | ××× | | ××× | | | V V V | | ××× | | | (xx) xxx | | |
| Diastolic BP (Change from baseline) [b] (mmHg) | | ××× | | ××× | | | V V V | | ××× | | | (xx) $xxx$ $(xx)$ $xxx$ $(xx)$ $xxx$ | | |
| Systolic Diastolic BP BP (Change from from baseline) baseline) [b] (mmHg) (mmHg) | | ××× | | ××× | | | × × × | | ××× | | | (XX) XXX | | |
| Nominal Time of<br>Assessment | <u>(x)</u> | NA | | NA | | r. | 47.7 | | Pre-Dose | | | | | |
| Time of treatment (24 h clock) | ×××××××××) | | | | | - 1<br>- 1 | 1111 - 11011 | | hh:mm | | | hh:mm | | |
| Visit<br>Visit Date<br>(Study Day) | ): Center ### | Screening<br>Visit 1 | $XXX = MM = DD$ $(T \times X Y)$ | Screening | Visit Z<br>YYYY-MM-DD | $(T \times Y)$ | YYYY-MM-DD | $(\mathbb{T} \times_{\underline{\hspace{1em}}} Y)$ | Visit x | YYYY-MM-DD | $(\mathbb{T}x_{\underline{\hspace{1ex}}}Y)$ | Unsch. | XXXX-MM-DD | $(T \times Y)$ |
| Subject ID Age (yrs)/<br>(Treatment Gender<br>Sequence) (Race) | <pre>Center # (Investigator): Center ### (xxxxxxxxxx)</pre> | Xxxxxx $Xx/F$ $(A/B/E/C/D$ $(xxxx)$ | | XX/E | (xxxx) | E) *** | (XXXX) | | Xx/F | (xxxx) | | | | |

Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. Race: A=Asian, AIAN=American Indian or Alaska Native, B=Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, O=Other W=White. Gender: F=Female, M=Male.

NA = Not Applicable.

A negative number for study day denotes the number of days prior to the start of study treatment. Otherwise, Study Day is Date – Date of dose in the Period + 1. Tx = Period.  $Tx_y = Period$  and Day within Period. Pxx = Days after dose in last Treatment Period. For change from baseline, baseline is defined as the last pre-dose measurement taken prior to dosing on Day 1 of a treatment [p [0]

period.

Notes to Programmer: Sort by Actual Treatment, Center, Subject ID, Date of Visit, and Nominal Time of Assessment. Nominal time of assessment of Pre-Dose should be provided for all assessments prior to the study drug dose on a day; Post-Dose values are those after the study drug dose was given on a day. If an assessment is not Pre-Dose or Post-Dose, then show 'NA' instead.

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


Listing 9.2 12-Lead Electrocardiogram (ECG) Analysis Set: All Subjects Randomized

| | | | | | | | ı i | Interval Raw Value | w Valu | Φ | | Any<br>Clinically |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age<br>Subject ID (yrs)/ | Age<br>yrs)/ | Visit | Treatment<br>Time | 11 | Heart | | | | | | | Significant<br>Abnormalities |
| (Treatment Ger | Gender | Visit Date | (24 h | | Rate | RR | PR | QRS Axis | QRS | ΔŢ | QTCF | on a Study |
| Sequence) (Ra | (ace) | (Race) (Study Day) [a] | clock) | Nominal Time of Assessment | (BPM) | (ms) | (ns) | (degrees) | (ms) | (ms) | (ms) | Day? [b] |
| Center # (Inve | stigat | Center # (Investigator): Center ### (xxxxxx | (xxxxxxxxx) | (XX) | | | | | | | | |
| xxxxx $Xx/F$ $(A/B/E/C/D)$ $(xxxx)$ | XX/F<br>(XXXX) | Visit 1<br>YYYY-MM-DD | NA | NA | × | ×× | ×× | × | × | × | × | NO |
| | | (××-) | | | | | | | | | | |
| | | Visit 6<br>YYYY-MM-DD<br>(Tx 1) | | Post-Dose | ×<br>×<br>× | x . x x x x x x x x x x x x x x x x x x | ×<br>×<br>× | × | ×.<br>× | ×<br>×<br>× | ×××× | Yes |
| | | Unscheduled<br>YYYY-MM-DD<br>(Tx Pv) | NA | NA | × | ×<br>×<br>× | ×<br>×<br>× | × | ×.<br>× | ×<br>×<br>× | ×<br>×<br>× | No |
| | | , | | | | | | | | | | |

Race: A-Asian, AIAN-American Indian or Alaska Native, B-Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, Treatment: A = Placebo, B = AS MDI 90 µg, C = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated.

- Date of dose in the Period + 1. Tx = Period. Tx\_y = Period and Day within Period. Pxx = Days after dose in last Treatment Period. O=Other W=White. Gender: F=Female, M=Male. A negative number of days prior to the start of study treatment. Otherwise, Study Day is Date ٦
  - Abnormalities at Screening Visits and Pre-Dose on Day 1 of Treatment Period 1 were noted on the Medical History CRF; Abnormalities Post-Dose on Day 1 of Treatment Period 1 or afterward were noted on the Adverse Events CRF. [2]

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/10902.sas Version YYYY-MM-DD xx:xx Source: eg.sas7bdat

Notes to Programmer: Sort by Actual Treatment, Center, Subject ID, Date of Visit, and Nominal Time of Assessment. Nominal time of assessment of Pre-Dose should be provided for all assessments prior to the study drug dose on a day; Post-Dose values are those after the study drug dose was given on a day. If an assessment is not Pre-Dose or Post-Dose, then show 'NA' instead.

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header.


Listing 9.3 Comments Analysis Set: All Subjects Randomized

| +2 d - Cd - Cd | Treatment | Age (yrs)/<br>Gender | | | |
|---|---|---|---|---|---|
| ID | Sequence | (Race) | Visit | Comment Applies To: | Comments |
| | ı | | | | |
| Study Ce | enter # / (Inves | Study Center # / (Investigator): ### (xxxxxxxxxx) | (XXXXXXXX) | | |
| ×××× | A/B/E/C/D | XX/M (XXXX) | Screening Visit 1 | | × |
| | | | Screening Visit la | Subject Eligibility | XXXXXXXXXX |
| | | | Screening Visit 1b | Study Medication | |
| | | | Visit 2 Visit 3 | Adverse Event | |
| | | | | Vital Signs | |
| | | | Premature | 12-Lead ECG | |
| | | | Discontinuation | Laboratory Results | |
| | | | Telephone Follow-up | Spirometry | |
| | | | Unscheduled | Visit Scheduling | |
| | | | | Other: xxxxxxxxxxxxx | |
| Treatmer | nt: A = Placebo, | Treatment: A = Placebo, B = AS MDI 90 µg, C | C = AS MDI 180 µg, D = | = AS MDI 180 µg, D = Proventil 90 µg, E = Proventil 180 µg, - = Not Treated. | 1 180 µg, - = Not Treated. |
| Race: A= | =Asian, AIAN=Ame | rican Indian or Al | aska Native, B=Black or | African American, NHPI=Native | Race: A-Asian, AIAN-American Indian or Alaska Native, B-Black or African American, NHPI=Native Hawaiian or Other Pacific Islander, |
| ( | | | | | |

O=Other W=White. Gender: F=Female, M=Male.

Source: xxxxxxx.sas7bdat

(Page n of N) Report generated by program: PT007001/sasdir/programs/statout/10904.sas Version YYYY-MM-DD xx:xx

#### Notes to Programmer:

Move 'Study Center/Inv' row header to the next page whenever there is not enough room on current page to fit at least one row of data underneath this header. Column and text in YELLOW is optional for studies where one or more 'Visits' are not associated with a Study Day. Sort by Center, Investigator, Subject ID, Visit, Study Day, and category that comment applies to (Subject Eligibility, Study Medication, etc...).